CLINICAL TRIAL: NCT02429791
Title: A Phase III, Randomized, Multicenter, Parallel-group, Non-inferiority Study Evaluating the Efficacy, Safety, and Tolerability of Switching to Dolutegravir Plus Rilpivirine From Current INI-, NNRTI-, or PI-based Antiretroviral Regimen in HIV-1-Infected Adults Who Are Virologically Suppressed
Brief Title: Regimen Switch to Dolutegravir + Rilpivirine From Current Antiretroviral Regimen in Human Immunodeficiency Virus Type 1 Infected and Virologically Suppressed Adults (SWORD-1)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Janssen Pharmaceuticals (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201636; 2014-005147-40 (EudraCT Number)
Record Dates: First submitted 2015-04-09; First posted 2015-04-29 (Estimated); Results first posted 2017-12-02 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: HIV Infections
Keywords: two-drug regimen; virologically-suppressed; dolutegravir plus rilpivirine; integrase inhibitor; protease inhibitor; NNRTI-sparing; non-nucleoside reverse transcriptase inhibitor; HIV; nucleoside reverse transcriptase inhibitors
MeSH Terms: conditions — HIV Infections | interventions — dolutegravir; Automobiles

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (2):
- Current antiretroviral regimen (CAR) (Active Comparator): Participants continued to receive their CAR (two nucleoside reverse transcriptase inhibitors [NRTIs] + a third agent). A third agent included either an: integrase strand transfer inhibitor (INSTI), a non-nucleoside reverse transcriptase inhibitor (NNRTI) or a protease inhibitor (PI). CAR was administered according to the approved labeling in an open-label fashion up to Week 52 during the Early Switch Phase. At Week 52, participants with human immunodeficiency virus-1 (HIV-1) ribonucleic acid (RNA) less than (<) 50 copies (c)/mL, switched to DTG 50 mg + RPV 25 mg once daily and were followed-up through the Late Switch Phase, at Week 148 and through the Continuation Phase, after Week 148.
  Interventions: Drug: CAR
- DTG + RPV (Experimental): Participants received DTG 50 mg + RPV 25 mg together, once daily, at approximately the same time, with a meal, in an open-label fashion up to Week 52, during the Early Switch Phase. Participants continued to receive DTG 50 mg + RPV 25 mg up to Week 148 during the Late Switch Phase. Participants who successfully completed 148 weeks of treatment were given the opportunity to continue to receive DTG + RPV once daily in the Continuation Phase (after Week 148).
  Interventions: Drug: DTG 50 mg; Drug: RPV 25 mg

INTERVENTIONS:
Drug: DTG 50 mg — Participants received one oral tablet of 50 mg DTG daily administered concomitantly with RPV. Each DTG tablet contained 52.62 mg dolutegravir sodium salt, which was equivalent to 50 mg dolutegravir free acid.
  Arms: DTG + RPV
Drug: RPV 25 mg — Participants received one oral tablet of 25 mg RPV daily administered concomitantly with DTG along with a meal. Each RPV tablet contained 27.5 mg of rilpivirine hydrochloride, which was equivalent to 25 mg of RPV.
  Arms: DTG + RPV
Drug: CAR — CAR included the following combinations: 2 NRTIs + 1 INI, 2 NRTIs + 1 NNRTI, or 2 NRTIs + 1 PI
  Arms: Current antiretroviral regimen (CAR)

SUMMARY:
The aim of this study was to determine if virologically suppressed human immunodeficiency virus type 1 (HIV-1) infected adults on an antiretroviral regimen (including 2 nucleoside reverse transcriptase inhibitors [NRTIs] plus a third agent) remain suppressed upon switching to a two-drug regimen with dolutegravir (DTG) + rilpivirine (RPV). The study primarily assessed the non-inferiority antiviral activity of switching to DTG + RPV once daily compared to continuation of current antiretroviral regimen (CAR) up to Week 48 with a switch visit for eligible subjects in the CAR group to initiate DTG + RPV therapy at Week 52. CAR included 2 NRTIs plus 1 HIV-1 integrase inhibitor (INI), or 1 non-nucleoside reverse transcriptase inhibitor (NNRTI), or 1 protease inhibitor (PI). The study included a 148-week open-label treatment phase, comprising of an Early Switch Phase (Day 1 to Week 52) and a Late Switch Phase (Week 52 to Week 148). The participants fulfilling the study eligibility criteria participated in the Early Switch Phase where they either switched from their CAR to DTG + RPV, or continued taking their CAR, until Week 52. At the end of Early Switch Phase, eligible participants proceeded to the Late Switch Phase where all participants in both DTG + RPV and CAR treatment groups received DTG + RPV therapy until Week 148. After Week 148, eligible subjects were given the opportunity to continue receiving DTG +RPV, in the Continuation Phase.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have been able to understand and comply with protocol requirements, instructions, and restrictions.
* Participants must have been likely to complete the study as planned.
* Participants must have been considered appropriate candidates for participation in an investigative clinical trial with oral medication (e.g., no active substance abuse, acute major organ disease, or planned long-term work assignments out of the country, etc.).
* HIV-1 infected men or women of greater than or equal to (>=)18 years of age.
* Must have been on uninterrupted current regimen (either the initial or second combination antiretroviral therapy [cART] regimen) for at least 6 months prior to screening; Any prior switch, defined as a change of a single drug or multiple drugs simultaneously, must have occurred due to tolerability and/or safety concerns or access to medications, or convenience/simplification. Acceptable stable cART regimens prior to screening include 2 NRTIs plus INI (either the initial or second cART regimen), or an NNRTI (either the initial or second cART regimen), or a Boosted PI (or atazanavir unboosted) (either the initial or second PI-based cART regimen).
* Documented evidence of at least two plasma HIV-1 RNA measurements <50 c/mL in the 12 months prior to Screening: one within the 6 to 12 month window, and one within 6 months prior to Screening;
* Plasma HIV-1 RNA <50 c/mL at Screening;
* A female may have been eligible to enter and participate in the study if she was of : Non-child-bearing potential either defined as post-menopausal (12 months of spontaneous amenorrhea and >=45 years of age) or physically incapable of becoming pregnant with documented tubal ligation, hysterectomy or bilateral oophorectomy or, Child-bearing potential with a negative pregnancy test at both Screening and Day 1 and agrees to use one of the following methods of contraception to avoid pregnancy: Complete abstinence from intercourse from 2 weeks prior to administration of study drug, throughout the study, and for at least 2 weeks after discontinuation of all study medications and completion of the Follow-up visit; Any intrauterine device (IUD) with published data showing that the expected failure rate is <1% per year (not all IUDs meet this criterion); Male partner sterilization with documentation of azoospermia prior to the female participant's entry into the study and this male is the sole partner for that participant; The documentation on male sterility could come from the site personnel's review of participant's medical records, medical examination, and/or semen analysis, or medical history interview provided by her or her partner; Approved hormonal contraception for participants randomly assigned to DTG + RPV arm (and for participants randomly assigned to CAR following switch to DTG + RPV at Week 52) or approved hormonal contraception plus a barrier method for participants assigned to CAR through Week 52; Approved hormonal contraception included: Combined estrogen and progestogen oral contraceptive, Contraceptive subdermal implant, Injectable progestogen, Contraceptive vaginal ring, Percutaneous contraceptive patches. Any other method with published data showing that the expected failure rate is <1% per year. Any contraception method must have been used consistently, in accordance with the approved product label during treatment with study drug and for at least 2 weeks after discontinuation of study drug and completion of the Follow-Up Visit. The investigator was responsible for ensuring that participants understand how to properly use these methods of contraception. Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal were not acceptable methods of contraception.
* Participants who were willing and able to understand requirements of study participation and provided signed and dated written informed consent prior to screening.
* For participants enrolled in France: participants were eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security category.

Exclusion Criteria:

Exclusionary Criteria prior to screening or Day 1:

* Within 6 months prior to Screening and after confirmed suppression to <50 c/mL on current ART regimen, any plasma HIV-1 RNA measurement >=50 c/mL.
* Within the 6 to 12 month window prior to screening and after confirmed suppression to <50 c/mL, any plasma HIV-1 RNA measurement >200 c/mL.
* Within the 6 to 12 month window prior to screening and after confirmed suppression to <50 c/mL, 2 or more plasma HIV-1 RNA measurements >=50 c/mL.
* Any drug holiday during the window between initiating first HIV ART and 6 months prior to screening, except for brief periods (less than 1 month) where all ART was stopped due to tolerability and/or safety concerns.
* Any switch to a second line regimen, defined as change of a single drug or multiple drugs simultaneously, due to virologic failure to therapy (defined as a confirmed plasma HIV 1 RNA measurement >=400 c/mL after initial suppression to <50 c/mL while on first line HIV therapy regimen).

Exclusionary medical conditions:

* Women who were pregnant, breastfeeding or planned to become pregnant or breastfeed during the study.
* Any evidence of an active Centers for Disease Control and Prevention Category C disease. Exceptions included cutaneous Kaposi's sarcoma not requiring systemic therapy and historic CD4+ lymphocyte counts of <200 cells per cubic millimeter (cells/mm^3).
* Participants with severe hepatic impairment (Class C) as determined by Child-Pugh Classification.
* Unstable liver disease (as defined by the presence of any of the following: ascites, encephalopathy, coagulopathy, hypoalbuminemia, oesophageal or gastric varices, or persistent jaundice), cirrhosis, known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Evidence of Hepatitis B virus (HBV) infection based on the results of testing at Screening for Hepatitis B surface antigen (HBsAg), Hepatitis B core antibody (anti-HBc), and Hepatitis B surface antibody (HBsAb) as follows: Participants positive for HBsAg were excluded; Participants positive for anti-HBc (negative HBsAg status) and negative for HBsAb were excluded.
* Participants with an anticipated need for any Hepatitis C virus (HCV) therapy during the Early Switch Phase and for interferon-based therapy for HCV throughout the entire study period.
* History or presence of allergy to the study drugs or their components or drugs of their class;
* Ongoing malignancy other than cutaneous Kaposi's sarcoma, basal cell carcinoma, or resected, non-invasive cutaneous squamous cell carcinoma, or cervical intraepithelial neoplasia; other localized malignancies require agreement between the investigator and the Study medical monitor for inclusion of the participant prior to randomization;
* Participants who in the investigator's judgment posed a significant suicidality risk. Participant's history of suicidal behavior and/or suicidal ideation should have been considered when evaluating for suicide risk;
* Any pre-existing physical or mental condition which, in the opinion of the Investigator, could have interfered with the participant's ability to comply with the dosing schedule and/or protocol evaluations or which could have compromised the safety of the participants;
* Any condition which, in the opinion of the Investigator, could have interfered with the absorption, distribution, metabolism or excretion of the study drugs or render the participant unable to take oral medication;

Exclusionary Treatments prior to Screening or Day 1:

* Use of medications which were associated with Torsades de Pointes.
* Treatment with an HIV-1 immunotherapeutic vaccine within 90 days of Screening.
* Treatment with any of the following agents within 28 days of Screening: radiation therapy; cytotoxic chemotherapeutic agents; any immunomodulators that alter immune responses.
* Exposure to an experimental drug or experimental vaccine within either 28 days, 5 half-lives of the test agent, or twice the duration of the biological effect of the test agent, whichever is longer, prior to Day 1 of this study.
* Participants who were participating or anticipated to be selected to participate in any other interventional study, with the exception of the DEXA sub-study 202094, after randomization
* A history of use of any regimen consisting of only single NNRTI therapy (even if only for peri-partum treatment), or only single or dual NRTI therapy prior to starting cART.
* Current or prior history of etravirine (ETR) use.
* Current use of tipranavir/ritonavir or fosamprenavir/ritonavir.
* Participants receiving any prohibited medication and who were unwilling or unable to switch to an alternate medication.

Exclusionary Laboratory Values or Clinical Assessments at Screening:

* Evidence of viral resistance based on the presence of any resistance associated major PI, INI, NRTI, or NNRTI mutation and integrase (IN) resistance associated substitution R263K in any available prior resistance genotype assay results.
* Any verified Grade 4 laboratory abnormality, with the exception of Grade 4 lipid abnormalities. A single repeat test was allowed during the Screening period to verify a result.
* Any acute laboratory abnormality at Screening, which, in the opinion of the investigator, would preclude the participant's participation in the study of an investigational compound.
* Alanine aminotransferase (ALT) >=5 × upper limit of normal (ULN), or ALT >=3 × ULN and bilirubin >=1.5 × ULN (with greater than [>] 35% direct bilirubin).
* Corrected QT interval (QTc [Bazett]) >450 milliseconds or QTc (Bazett) >480 milliseconds for participants with bundle branch block. The QTc was the QT interval corrected for heart rate according to Bazett's formula (QTcB).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 510 (Actual)
Dates: Start 2015-04-14 (Actual); Primary Completion 2016-09-16 (Actual); Study Completion 2023-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (53):
- United States (12):
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Ft. Pierce, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Camden, New Jersey
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Lynchburg, Virginia
- GSK Investigational Site, Ciudad Autonoma de Buenos Aire, Argentina
- Australia (2):
  - GSK Investigational Site, Darlinghurst
  - GSK Investigational Site, Prahran
- Belgium (4):
  - GSK Investigational Site, Antwerp
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Liège
- Canada (5):
  - GSK Investigational Site, Ottawa
  - GSK Investigational Site, Québec
  - GSK Investigational Site, Toronto
  - GSK Investigational Site, Vancouver
  - GSK Investigational Site, Victoria
- France (3):
  - GSK Investigational Site, Garches
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Paris
- Germany (3):
  - GSK Investigational Site, Frankfurt
  - GSK Investigational Site, Hamburg
  - GSK Investigational Site, München
- Italy (2):
  - GSK Investigational Site, Brescia
  - GSK Investigational Site, Milan
- GSK Investigational Site, Rotterdam, Netherlands
- Russia (5):
  - GSK Investigational Site, Kazan'
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Oryol
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Smolensk
- Spain (11):
  - GSK Investigational Site, Alcalá de Henares
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Elche
  - GSK Investigational Site, Granada
  - GSK Investigational Site, Huelva
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Marbella
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Palma de Mallorca
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Valencia
- Taiwan (2):
  - GSK Investigational Site, Kaohsiung City
  - GSK Investigational Site, Taipei
- United Kingdom (2):
  - GSK Investigational Site, London
  - GSK Investigational Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- [Background] Llibre JM, Hung CC, Brinson C, et al. Efficacy, safety, and tolerability of dolutegravir plus rilpivirine for the maintenance of virologic suppression in HIV-1-infected adults: the phase III, randomized, open-label, active-controlled, noninferiority SWORD-1 and SWORD-2 studies. Lancet [epublished ahead of print] 6 January 2018.
- [Derived] Aboud M, Orkin C, Podzamczer D, Bogner JR, Baker D, Khuong-Josses MA, Parks D, Angelis K, Kahl LP, Blair EA, Adkison K, Underwood M, Matthews JE, Wynne B, Vandermeulen K, Gartland M, Smith K. Efficacy and safety of dolutegravir-rilpivirine for maintenance of virological suppression in adults with HIV-1: 100-week data from the randomised, open-label, phase 3 SWORD-1 and SWORD-2 studies. Lancet HIV. 2019 Sep;6(9):e576-e587. doi: 10.1016/S2352-3018(19)30149-3. Epub 2019 Jul 12. PMID 31307948
- [Derived] Llibre JM, Hung CC, Brinson C, Castelli F, Girard PM, Kahl LP, Blair EA, Angelis K, Wynne B, Vandermeulen K, Underwood M, Smith K, Gartland M, Aboud M. Efficacy, safety, and tolerability of dolutegravir-rilpivirine for the maintenance of virological suppression in adults with HIV-1: phase 3, randomised, non-inferiority SWORD-1 and SWORD-2 studies. Lancet. 2018 Mar 3;391(10123):839-849. doi: 10.1016/S0140-6736(17)33095-7. Epub 2018 Jan 6. PMID 29310899
- [Derived] McComsey GA, Lupo S, Parks D, Poggio MC, De Wet J, Kahl LP, Angelis K, Wynne B, Vandermeulen K, Gartland M, Cupo M, Aboud M; 202094 Sub-Study Investigators. Switch from tenofovir disoproxil fumarate combination to dolutegravir with rilpivirine improves parameters of bone health. AIDS. 2018 Feb 20;32(4):477-485. doi: 10.1097/QAD.0000000000001725. PMID 29239893

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 65 centers in 13 countries.
Pre-assignment Details: 510 participants were randomized and 2 participants withdrew before being exposed to study drug. The study included an Early Switch Phase, a Late Switch Phase, and a Continuation Phase.
Period: Early Switch Phase (Up to Week 52)
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Started | 252 | 256
Completed | 239 | 238
Not Completed | 13 | 18
Not completed — Adverse Event | 6 | 2
Not completed — Physician Decision | 0 | 2
Not completed — Lack of Efficacy | 2 | 1
Not completed — Lost to Follow-up | 1 | 2
Not completed — Protocol Violation | 1 | 4
Not completed — Withdrawal by Subject | 3 | 7
Period: Late Switch Phase (Week 52 to Week 148)
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Started | 239 | 238
Completed | 214 | 210
Not Completed | 25 | 28
Not completed — Adverse Event | 11 | 12
Not completed — Physician Decision | 0 | 4
Not completed — Lack of Efficacy | 4 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Violation | 3 | 3
Not completed — Withdrawal by Subject | 7 | 5
Period: Continuation Phase(Week 148 to Week 411)
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Started | 186 | 183
Completed | 179 | 178
Not Completed | 7 | 5
Not completed — Adverse Event | 3 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Investigator discretion | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR) | Total
Number analyzed (Participants) | 252 | 256 | 508
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.6 (10.93) | 43.6 (10.76) | 43.6 (10.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 51 | 109
  Male | 194 | 205 | 399
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 6 | 9
  Japanese/East Asian (EA) Heritage (H.)/South EA H. | 25 | 34 | 59
  Black/African American | 24 | 27 | 51
  Native Hawaiian or other Pacific Islander | 1 | 0 | 1
  White | 198 | 188 | 386
  American Indian or Alaska Native and white | 0 | 1 | 1
  African American/African H. and Asian | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Plasma HIV-1 RNA <50 c/mL at Week 48 Using Snapshot Algorithm
Description: Percentage of participants with plasma HIV 1 RNA <50 c/mL at Week 48 using the Food and Drug Administration (FDA) snapshot algorithm was assessed to demonstrate the non-inferior antiviral activity of switching to DTG + RPV once daily compared to continuation of CAR over 48 weeks in HIV-1 infected antiretroviral therapy (ART)-experienced participants. Virologic success or failure was determined by the last available HIV-1 RNA assessment while the participant was on-treatment within the window of the visit of interest.
  Plasma samples were collected for quantitative analysis of HIV-1 RNA.
Time Frame: Week 48
Population: The analysis was performed on the Intent-to-Treat Exposed (ITT-E) population which consisted of all randomly assigned participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 252 | 256
Percentage of participants | 95 | 96
Statistical Analysis 1: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Non-Inferiority — Non-inferiority was concluded if the lower bound of a two-sided 95% confidence interval for the difference in response rates between the two treatment arms was greater than -10%; Risk Difference (RD) = -0.6, 95% CI 2-sided [-4.3 to 3.0] — Estimates based on Cochran-Mantel Haenszel stratified analysis adjusting for Baseline stratification factors: Age group (< or >=50 years old) and Baseline third agent (PI, NNRTI, INI)

2. Secondary Outcome: Changes From Baseline in Cluster Designation (CD)4+ Lymphocyte Count at Weeks 24 and 48
Description: Blood samples were collected and CD4+ cell count assessment by flow cytometry was carried out to evaluate the immunological activity of DTG + RPV once daily compared to continuation of CAR. Value obtained at Day 1 was considered as Baseline value. Change from Baseline was calculated as value at indicated time point minus Baseline value.
Time Frame: At Weeks 24 and 48
Population: ITT-E Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Cells per millimeter cube (mm^3)
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 252 | 256
Cells per millimeter cube (mm^3)
  Week 24: number analyzed (Participants) | 247 | 249
  Week 24 | 16.2 (150.34) | 47.4 (179.68)
  Week 48: number analyzed (Participants) | 239 | 245
  Week 48 | 32.3 (149.52) | 41.8 (185.53)

3. Secondary Outcome: Percentage of Participants With Plasma HIV 1 RNA <50 c/mL at Week 24 Using Snapshot Algorithm
Description: Percentage of participants with plasma HIV 1 RNA < 50 c/mL at Week 24 using the FDA snapshot algorithm was assessed to evaluate the antiviral activity of DTG + RPV once daily compared to continuation of CAR. Virologic success or failure was determined by the last available HIV-1 RNA assessment while the participant was on-treatment within the window of the visit of interest. Plasma samples were collected for quantitative analysis of HIV-1 RNA.
Time Frame: Week 24
Population: ITT-E Population
Measure: Number; unit: Percentage of participants
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 252 | 256
Percentage of participants | 98 | 96
Statistical Analysis 1: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Other; Risk Difference (RD) = 1.0, 95% CI 2-sided [-1.9 to 4.0] — Cochran-Mantel Haenszel stratified analysis adjusting for Baseline stratification factors: Age group (< or >=50 years old) and Baseline third agent (PI, NNRTI, INI). No formal non-inferiority margin has been pre-specified for secondary endpoints

4. Secondary Outcome: Number of Participants With Common Non-serious Adverse Event (AE), Any Serious AE (SAE), AE of Maximum Toxicity Grade 1, 2, 3 or 4 and AE Leading to Discontinuation (AELD)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect, any other situation according to medical or scientific judgment that may not be immediately life-threatening or result in death or hospitalization but may jeopardize participant or may require medical or surgical intervention were categorized as SAE. AEs were graded as per Division of Acquired Immunodeficiency Syndrome (DAIDS) grading. Grade 1=mild; grade 2=moderate; grade 3=severe; grade 4=potentially life-threatening. Common AEs were those with >5% incidence for either treatment.
Time Frame: Up to Week 411 or study discontinuation
Population: Safety Population included all randomized participants who have received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 252 | 238
Participants
  Common non-serious AE | 158 | 126
  Any SAE | 37 | 30
  Maximum toxicity Grade 1 AE | 82 | 73
  Maximum toxicity Grade 2 AE | 97 | 107
  Maximum toxicity Grade 3 AE | 37 | 17
  Maximum toxicity Grade 4 AE | 15 | 9
  AELD | 22 | 13

5. Secondary Outcome: Number of Participants With Maximum Post-baseline Emergent Chemistry Toxicities Over 48 Weeks
Description: Blood samples were collected to evaluate alanine aminotransferase (ALT), albumin, alkaline phosphatase (ALP), aspartate aminotransferase (AST), total bilirubin, chloride, creatinine, glucose, potassium, phosphate, sodium, blood urea nitrogen (BUN), total carbon dioxide, lipase, creatine phosphokinase and creatinine clearance. Value obtained at Day 1 was considered as Baseline value. Number of participants who experienced maximum grade toxicity post-Baseline in clinical chemistry over 48 weeks was summarized. Clinical chemistry toxicities were graded using DAIDS grading table for grading severity of adult and pediatric adverse events. Grade 1=mild; grade 2=moderate; grade 3=severe; grade 4=potentially life-threatening. For all laboratory parameters, one assessment out of range was sufficient to be considered a chemistry toxicity.
Time Frame: Up to 48 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 252 | 256
Participants
  Grade 1 | 95 | 78
  Grade 2 | 61 | 86
  Grade 3 | 22 | 23
  Grade 4 | 5 | 9

6. Secondary Outcome: Number of Participants With Maximum Post-Baseline Emergent Hematology Toxicities Over 48 Weeks
Description: Blood samples were collected to evaluate hemoglobin, hematocrit, basophils, eosinophils, lymphocytes, monocytes, neutrophils, mean corpuscular volume (MCV), red blood cell (RBC) count, white blood cell (WBC) count and platelet count. Value obtained at Day 1 was considered as Baseline value. Number of participants who experienced maximum grade toxicity post-Baseline in hematology over 48 weeks was summarized. Hematology toxicities were graded using DAIDS grading table for grading severity of adult and pediatric adverse events. Grade 1=mild; grade 2=moderate; grade 3=severe; grade 4=potentially life-threatening. For all laboratory parameters, one assessment out of range was sufficient to be considered a hematology toxicity.
Time Frame: Up to 48 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 252 | 256
Participants
  Grade 1 | 11 | 11
  Grade 2 | 3 | 2
  Grade 3 | 3 | 1
  Grade 4 | 0 | 1

7. Secondary Outcome: Mean Change From Baseline in High-sensitivity C-reactive Protein (Hs-CRP) at Week 48
Description: Blood biomarker samples were collected at Baseline (Day 1) and Week 48 to assess hs-CRP. Change from Baseline was calculated as value at indicated time point minus Baseline value.
Time Frame: At Week 48
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: mg/ Liter (L)
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 234 | 243
mg/ Liter (L) | 0.11 (5.379) | 0.15 (4.944)

8. Secondary Outcome: Mean Change From Baseline in Cystatin C at Week 48
Description: Blood biomarker samples were collected at Baseline (Day 1) and Week 48 to assess cystatin C. Change from Baseline was calculated as value at indicated time point minus Baseline value.
Time Frame: At Week 48
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 237 | 245
mg/L | 0.00 (0.113) | -0.01 (0.106)

9. Secondary Outcome: Mean Change From Baseline in D-Dimer at Week 48
Description: Blood biomarker samples were collected at Baseline (Day 1) and Week 48 to assess D-Dimer. Change from Baseline was calculated as value at indicated time point minus Baseline value.
Time Frame: At Week 48
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Nanomole/L fibrinogen equivalent units
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 224 | 238
Nanomole/L fibrinogen equivalent units | -0.02 (2.651) | 0.02 (2.501)

10. Secondary Outcome: Mean Change From Baseline in Fatty Acid Binding Protein 2 (FABP) and Soluble Cluster Designation (CD)14 at Week 48
Description: Blood biomarker samples were collected at Baseline (Day 1) and Week 48 to assess FABP and soluble cluster designation (CD)14. Change from Baseline was calculated as value at indicated time point minus Baseline value.
Time Frame: At Week 48
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Nanogram/milliliter
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 252 | 256
Nanogram/milliliter
  FABP: number analyzed (Participants) | 233 | 242
  FABP | -2.79 (3.007) | -1.93 (2.150)
  Soluble CD14: number analyzed (Participants) | 234 | 242
  Soluble CD14 | 379.72 (634.053) | 754.54 (656.462)

11. Secondary Outcome: Mean Change From Baseline in Soluble CD163 and Oxidized Low Density Lipoprotein (LDL) at Week 48
Description: Blood biomarker samples were collected at Baseline (Day 1) and Week 48 to assess soluble CD163 and oxidized LDL. Change from Baseline was calculated as value at indicated time point minus Baseline value.
Time Frame: At Week 48
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Microgram (µg)/Liter
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 252 | 256
Microgram (µg)/Liter
  Soluble CD163: number analyzed (Participants) | 232 | 241
  Soluble CD163 | 50.18 (188.772) | 54.26 (238.900)
  Oxidized LDL: number analyzed (Participants) | 234 | 242
  Oxidized LDL | 9.49 (745.962) | -41.30 (726.014)

12. Secondary Outcome: Mean Change From Baseline in Retinol Binding Protein (RBP), Serum Creatinine and Glucose at Week 48
Description: Blood biomarker samples were collected at Baseline (Day 1) and Week 48 to assess RBP, serum creatinine and glucose. Change from Baseline was calculated as value at indicated time point minus Baseline value.
Time Frame: At Week 48
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: mg/deciliter (dL)
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 252 | 256
mg/deciliter (dL)
  RBP: number analyzed (Participants) | 235 | 243
  RBP | -0.13 (1.023) | 0.03 (0.974)
  Serum creatinine: number analyzed (Participants) | 238 | 243
  Serum creatinine | 0.087 (0.1074) | 0.011 (0.0876)
  Glucose: number analyzed (Participants) | 227 | 227
  Glucose | 0.762 (13.6194) | 2.492 (12.1674)

13. Secondary Outcome: Mean Change From Baseline in Urine Phosphate at Week 48
Description: Urine biomarker samples were collected at Baseline (Day 1) and Week 48 to assess urine phosphate. Change from Baseline was calculated as value at indicated time point minus Baseline value.
Time Frame: At Week 48
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimoles (mmol)/ L
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 218 | 224
Millimoles (mmol)/ L | -1.079 (16.9226) | -1.511 (15.8515)

14. Secondary Outcome: Mean Change From Baseline in Beta-2-microglobulin (B2M) (Blood and Urine), Urine RBP and 25 Hydroxy-vitamin D (Blood) at Week 48
Description: Blood biomarker samples were collected at Baseline (Day 1) and Week 48 to assess B2M and 25 hydroxy-vitamin D. Urine samples were collected to assess B2M and RBP. Change from Baseline was calculated as value at indicated time point minus Baseline value. For 25 hydroxy-vitamin D, analysis of changes from Baseline was performed on log-transformed data. Results were transformed back via exponential transformation such that treatment comparisons are assessed via odds ratios.
Time Frame: At Week 48
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Nanomoles/ L
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 252 | 256
Nanomoles/ L
  Blood B2M: number analyzed (Participants) | 233 | 241
  Blood B2M | -15.1452 (44.55903) | -4.5995 (38.90474)
  Blood 25 hydroxy-vitamin D: number analyzed (Participants) | 235 | 244
  Blood 25 hydroxy-vitamin D | -13.9 (22.76) | -8.2 (24.43)
  Urine B2M: number analyzed (Participants) | 89 | 96
  Urine B2M | -128.2045 (726.38825) | 39.8394 (253.43025)
  Urine RBP: number analyzed (Participants) | 221 | 231
  Urine RBP | -8.8395 (28.83977) | -0.5851 (27.56405)
Statistical Analysis 1: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Other; p = 0.007, ANCOVA — P-value for interaction between treatment group and baseline third agent (25 hydroxy-vitamin D)
Statistical Analysis 2: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Superiority; p = 0.275, ANCOVA — P value to assess difference between treatment groups (25 hydroxy-vitamin D - NNRTI); Odds Ratio (OR) = 0.958, 95% CI 2-sided [0.888 to 1.034] — Estimates are calculated from an ANCOVA model adjusting for Baseline third agent class, age, sex, BMI category, smoking status and baseline biomarker level
Statistical Analysis 3: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Superiority; p = 0.112, ANCOVA — P value to assess difference between treatment groups (25 hydroxy-vitamin D - INI); Odds Ratio (OR) = 0.902, 95% CI 2-sided [0.793 to 1.025] — [estimate comment as in outcome 14, analysis 2]
Statistical Analysis 4: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Superiority; p = 0.002, ANCOVA — P value to assess difference between treatment groups (25 hydroxy-vitamin D - PI); Odds Ratio (OR) = 0.847, 95% CI 2-sided [0.763 to 0.942] — [estimate comment as in outcome 14, analysis 2]

15. Secondary Outcome: Mean Change From Baseline in Urine Albumin/Creatinine Ratio and Urine Protein/Creatinine Ratio at Week 48
Description: Urine biomarker samples were collected at Baseline (Day 1) and Week 48 to assess urine albumin/creatinine ratio and urine protein/creatinine ratio. Change from Baseline was calculated as value at indicated time point minus Baseline value.
Time Frame: At Week 48
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams (g)/ mol
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 252 | 256
Grams (g)/ mol
  Urine albumin/creatinine ratio: number analyzed (Participants) | 166 | 171
  Urine albumin/creatinine ratio | -1.19 (3.916) | -2.59 (28.878)
  Urine protein/creatinine ratio: number analyzed (Participants) | 176 | 182
  Urine protein/creatinine ratio | -5.63 (17.219) | -1.43 (42.832)

16. Secondary Outcome: Mean Change From Baseline in Bone-specific Alkaline Phosphatase, Procollagen 1 N-terminal Propeptide, Osteocalcin, Type I Collagen C-Telopeptides and Soluble Vascular Cell Adhesion Molecule (sVCAM) at Week 48
Description: Blood biomarker samples were collected at Baseline (Day 1) and Week 48 to assess bone-specific alkaline phosphatase, procollagen 1 N-terminal propeptide, osteocalcin, Type I Collagen C-Telopeptides and sVCAM. Change from Baseline was calculated as value at indicated time point minus Baseline value. For bone-specific alkaline phosphatase, procollagen 1-N-propeptide, osteocalcin and type 1 collagen C-telopeptide, analyses of changes from baseline were performed on log-transformed data. Results were transformed back via exponential transformation such that treatment comparisons are assessed via odds ratios.
Time Frame: At Week 48
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: µg/ L
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 252 | 256
µg/ L
  Bone-specific alkaline phosphatase: number analyzed (Participants) | 234 | 244
  Bone-specific alkaline phosphatase | -2.89 (4.024) | 0.90 (4.129)
  Procollagen type 1 N-propeptide: number analyzed (Participants) | 234 | 242
  Procollagen type 1 N-propeptide | -9.1 (20.34) | -1.4 (18.95)
  Osteocalcin: number analyzed (Participants) | 233 | 242
  Osteocalcin | -4.40 (7.605) | -0.68 (6.579)
  Type I Collagen C-Telopeptides: number analyzed (Participants) | 234 | 241
  Type I Collagen C-Telopeptides | -0.18 (0.307) | -0.04 (1.160)
  sVCAM: number analyzed (Participants) | 234 | 243
  sVCAM | -2.21 (1291.994) | 89.07 (1239.465)
Statistical Analysis 1: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Other; p = 0.001, ANCOVA — P-value for interaction between treatment group and baseline third agent (bone-specific alkaline phosphatase)
Statistical Analysis 2: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Superiority; p < .001, ANCOVA — P value to assess difference between treatment groups (bone-specific alkaline phosphatase - NNRTI); Odds Ratio (OR) = 0.724, 95% CI 2-sided [0.679 to 0.772] — [estimate comment as in outcome 14, analysis 2]
Statistical Analysis 3: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Superiority; p < .001, ANCOVA — P value to assess difference between treatment groups (bone-specific alkaline phosphatase - INI); Odds Ratio (OR) = 0.825, 95% CI 2-sided [0.742 to 0.918] — [estimate comment as in outcome 14, analysis 2]
Statistical Analysis 4: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Superiority; p < .001, ANCOVA — P value to assess difference between treatment groups (bone-specific alkaline phosphatase - PI); Odds Ratio (OR) = 0.810, 95% CI 2-sided [0.742 to 0.884] — [estimate comment as in outcome 14, analysis 2]
Statistical Analysis 5: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Other; p = 0.677, ANCOVA — P-value for interaction between treatment group and Baseline third agent (procollagen type 1-N-propeptide)
Statistical Analysis 6: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Superiority; p < .001, ANCOVA — P value to assess difference between treatment groups (procollagen type 1-N-propeptide); Odds Ratio (OR) = 0.817, 95% CI 2-sided [0.774 to 0.863] — [estimate comment as in outcome 14, analysis 2]
Statistical Analysis 7: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Other; p < .001, ANCOVA — P-value for interaction between treatment group and Baseline third agent (osteocalcin)
Statistical Analysis 8: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Superiority; p < .001, ANCOVA — P value to assess difference between treatment groups (osteocalcin - NNRTI); Odds Ratio (OR) = 0.881, 95% CI 2-sided [0.823 to 0.943] — [estimate comment as in outcome 14, analysis 2]
Statistical Analysis 9: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Superiority; p = 0.001, ANCOVA — P value to assess difference between treatment groups (osteocalcin - INI); Odds Ratio (OR) = 0.829, 95% CI 2-sided [0.740 to 0.930] — [estimate comment as in outcome 14, analysis 2]
Statistical Analysis 10: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Superiority; p < .001, ANCOVA — P value to assess difference between treatment groups (osteocalcin - PI); Odds Ratio (OR) = 0.691, 95% CI 2-sided [0.628 to 0.759] — [estimate comment as in outcome 14, analysis 2]
Statistical Analysis 11: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Other; p = 0.782, ANCOVA — P-value for interaction between treatment group and baseline third agent (type 1 collagen cross-linked C-telopeptide)
Statistical Analysis 12: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Superiority; p < .001, ANCOVA — P value to assess difference between treatment groups (type 1 collagen cross-linked C-telopeptide); Odds Ratio (OR) = 0.804, 95% CI 2-sided [0.742 to 0.872] — [estimate comment as in outcome 14, analysis 2]

17. Secondary Outcome: Mean Change From Baseline in Interleukin 6 (IL-6) at Week 48
Description: Blood biomarker samples were collected at Baseline (Day 1) and Week 48 to assess IL-6. Change from Baseline was calculated as value at indicated time point minus Baseline value.
Time Frame: At Week 48
Population: Safety Population. Only those participants with data available at the specified time point were analyzed.
Measure: Mean (Standard Deviation); unit: Nanograms (ng)/ L
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 233 | 243
Nanograms (ng)/ L | 0.17 (2.736) | -0.18 (2.944)

18. Secondary Outcome: Mean Change From Baseline in Insulin Resistance Based on Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) at Week 48
Description: Blood biomarker samples were collected at Baseline (Day 1) and Week 48 to assess insulin resistance. Change from Baseline was calculated as value at indicated time point minus Baseline value. The homeostatic model assessment (HOMA) of insulin resistance (HOMA-IR) index, the product of basal glucose and insulin levels divided by 22.5 (1,2), is regarded as a simple, inexpensive, and reliable surrogate measure of insulin resistance.
Time Frame: At Week 48
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: HOMA-IR Score
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 229 | 237
HOMA-IR Score | -0.30 (5.740) | 0.51 (3.530)

19. Secondary Outcome: Mean Change From Baseline in Fasting Lipids at Weeks 24 and 48
Description: Blood samples were collected at Baseline (Day 1), Week 24 and Week 48 to assess fasting lipids which included total cholesterol, low density lipoprotein (LDL) cholesterol, high density lipoprotein (HDL) cholesterol and triglycerides. Change from Baseline was calculated as value at indicated time point minus Baseline value.
Time Frame: At Week 24 and at Week 48
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: mmol/ L
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 252 | 256
mmol/ L
  Total cholesterol, Week 24: number analyzed (Participants) | 228 | 223
  Total cholesterol, Week 24 | 0.076 (0.8398) | 0.061 (0.7368)
  Total cholesterol, Week 48: number analyzed (Participants) | 221 | 218
  Total cholesterol, Week 48 | 0.089 (0.8488) | 0.064 (0.7197)
  LDL cholesterol calculation, Week 24: number analyzed (Participants) | 224 | 217
  LDL cholesterol calculation, Week 24 | 0.165 (0.7065) | 0.103 (0.6503)
  LDL cholesterol calculation, Week 48: number analyzed (Participants) | 215 | 211
  LDL cholesterol calculation, Week 48 | 0.108 (0.7178) | 0.029 (0.6134)
  HDL cholesterol direct, Week 24: number analyzed (Participants) | 228 | 223
  HDL cholesterol direct, Week 24 | -0.030 (0.2601) | -0.044 (0.2394)
  HDL cholesterol direct, Week 48: number analyzed (Participants) | 221 | 218
  HDL cholesterol direct, Week 48 | 0.023 (0.2757) | 0.018 (0.2722)
  Triglycerides, Week 24: number analyzed (Participants) | 228 | 223
  Triglycerides, Week 24 | -0.154 (0.7324) | -0.001 (0.7712)
  Triglycerides, Week 48: number analyzed (Participants) | 221 | 218
  Triglycerides, Week 48 | -0.093 (0.9767) | 0.046 (0.8274)

20. Secondary Outcome: Number of Participants With Genotypic Resistance- Early Switch Phase
Description: Plasma samples were collected for drug resistance testing. Genotypic Resistance data for the following drugs (Rilpivirine [RPV], Dolutegravir [DTG], Emtricitabine [FTC], Tenofovir [TDF], Darunavir/r [DRV/r]) in participants Meeting CVW Criteria has been presented.
Time Frame: Up to Week 52
Population: The analysis was performed on the Confirmed Virologic Withdrawal (CVW) resistance population which was comprised of all participants in the ITT-E Population who met confirmed CVW through the end of visit window (Week 48, Week 100 or Week 148) and had available on-treatment genotypic resistance data at the time CVW criterion was met.
Measure: Count of Participants; unit: Participants
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 1 | 1
Participants
  NNRTI, RPV, Susceptible | 1 | NA — NA indicates data was not applicable as the drugs were not received. Genotypic resistance data is only shown for drugs received for Participants Meeting Confirmed Virologic Withdrawal Criteria
  NNRTI, RPV, Potential low-level resistance | 0 | NA — NA indicates data was not applicable as the drugs were not received. Genotypic resistance data is only shown for drugs received for Participants Meeting Confirmed Virologic Withdrawal Criteria
  NNRTI, RPV, Low-level resistance | 0 | NA — NA indicates data was not applicable as the drugs were not received. Genotypic resistance data is only shown for drugs received for Participants Meeting Confirmed Virologic Withdrawal Criteria
  NNRTI, RPV, Intermediate resistance | 0 | NA — NA indicates data was not applicable as the drugs were not received. Genotypic resistance data is only shown for drugs received for Participants Meeting Confirmed Virologic Withdrawal Criteria
  NNRTI, RPV, High-level resistance | 0 | NA — NA indicates data was not applicable as the drugs were not received. Genotypic resistance data is only shown for drugs received for Participants Meeting Confirmed Virologic Withdrawal Criteria
  INI, DTG, Susceptible | 1 | NA — NA indicates data was not applicable as the drugs were not received. Genotypic resistance data is only shown for drugs received for Participants Meeting Confirmed Virologic Withdrawal Criteria
  INI, DTG, Potential low-level resistance | 0 | NA — NA indicates data was not applicable as the drugs were not received. Genotypic resistance data is only shown for drugs received for Participants Meeting Confirmed Virologic Withdrawal Criteria
  INI, DTG, Low-level resistance | 0 | NA — NA indicates data was not applicable as the drugs were not received. Genotypic resistance data is only shown for drugs received for Participants Meeting Confirmed Virologic Withdrawal Criteria
  INI, DTG, Intermediate resistance | 0 | NA — NA indicates data was not applicable as the drugs were not received. Genotypic resistance data is only shown for drugs received for Participants Meeting Confirmed Virologic Withdrawal Criteria
  INI, DTG, High-level resistance | 0 | NA — NA indicates data was not applicable as the drugs were not received. Genotypic resistance data is only shown for drugs received for Participants Meeting Confirmed Virologic Withdrawal Criteria
  NRTI, FTC, Susceptible | NA — NA indicates data was not applicable as the drugs were not received. Genotypic resistance data is only shown for drugs received for Participants Meeting Confirmed Virologic Withdrawal Criteria | 1
  NRTI, FTC, Potential low-level resistance | NA — NA indicates data was not applicable as the drugs were not received. Genotypic resistance data is only shown for drugs received for Participants Meeting Confirmed Virologic Withdrawal Criteria | 0
  NRTI, FTC, Low-level resistance | NA — NA indicates data was not applicable as the drugs were not received. Genotypic resistance data is only shown for drugs received for Participants Meeting Confirmed Virologic Withdrawal Criteria | 0
  NRTI, FTC, Intermediate resistance | NA — NA indicates data was not applicable as the drugs were not received. Genotypic resistance data is only shown for drugs received for Participants Meeting Confirmed Virologic Withdrawal Criteria | 0
  NRTI, FTC, High-level resistance | NA — NA indicates data was not applicable as the drugs were not received. Genotypic resistance data is only shown for drugs received for Participants Meeting Confirmed Virologic Withdrawal Criteria | 0
  NRTI, TDF, Susceptible | NA — NA indicates data was not applicable as the drugs were not received. Genotypic resistance data is only shown for drugs received for Participants Meeting Confirmed Virologic Withdrawal Criteria | 1
  NRTI, TDF, Potential low-level resistance | NA — NA indicates data was not applicable as the drugs were not received. Genotypic resistance data is only shown for drugs received for Participants Meeting Confirmed Virologic Withdrawal Criteria | 0
  NRTI, TDF, Low-level resistance | NA — NA indicates data was not applicable as the drugs were not received. Genotypic resistance data is only shown for drugs received for Participants Meeting Confirmed Virologic Withdrawal Criteria | 0
  NRTI, TDF, Intermediate resistance | NA — NA indicates data was not applicable as the drugs were not received. Genotypic resistance data is only shown for drugs received for Participants Meeting Confirmed Virologic Withdrawal Criteria | 0
  NRTI, TDF, High-level resistance | NA — NA indicates data was not applicable as the drugs were not received. Genotypic resistance data is only shown for drugs received for Participants Meeting Confirmed Virologic Withdrawal Criteria | 0
  PI, DRV/r, Susceptible | NA — NA indicates data was not applicable as the drugs were not received. Genotypic resistance data is only shown for drugs received for Participants Meeting Confirmed Virologic Withdrawal Criteria | 1
  PI, DRV/r, Potential low-level resistance | NA — NA indicates data was not applicable as the drugs were not received. Genotypic resistance data is only shown for drugs received for Participants Meeting Confirmed Virologic Withdrawal Criteria | 0
  PI, DRV/r, Low-level resistance | NA — NA indicates data was not applicable as the drugs were not received. Genotypic resistance data is only shown for drugs received for Participants Meeting Confirmed Virologic Withdrawal Criteria | 0
  PI, DRV/r, Intermediate resistance | NA — NA indicates data was not applicable as the drugs were not received. Genotypic resistance data is only shown for drugs received for Participants Meeting Confirmed Virologic Withdrawal Criteria | 0
  PI, DRV/r, High-level resistance | NA — NA indicates data was not applicable as the drugs were not received. Genotypic resistance data is only shown for drugs received for Participants Meeting Confirmed Virologic Withdrawal Criteria | 0

21. Secondary Outcome: Number of Participants With Genotypic Resistance-DTG+RPV Group Through Early and Late Switch Phase
Description: Plasma samples were collected for drug resistance testing. Genotypic Resistance data for the following drugs (DTG, Elvitegravir [EVG], Raltegravir [RAL], Delavirdine [DLV], Efavirenz [EFV], Etravirine [ETR], Nevirapine [NVP], RPV, Lamivudine [3TC], Abacavir [ABC], FTC, TDF, Zidovudine [ZDV], Stavudine [d4T], Didanosine [ddI], Atazanavir/r [ATV/r], DRV/r, Fosamprenavir/r [FPV/r], Indinavir/r [IDV/r], Lopinavir/r [LPV/r], Nelfinavir [NFV], Ritonavir [RTV], Saquinavir/r [SQV/r], Tipranavir/r [TPV/r]) in participants Meeting CVW Criteria has been presented.
Time Frame: Up to Week 148
Population: CVW resistance Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG + RPV
Number analyzed (Participants) | 5
Participants
  INI, DTG, Susceptible | 5
  INI, DTG, Potential low-level resistance | 0
  INI, DTG, Low-level resistance | 0
  INI, DTG, Intermediate resistance | 0
  INI, DTG, High-level resistance | 0
  INI, EVG,Susceptible | 4
  INI, EVG, Potential low-level resistance | 1
  INI, EVG,Low-level resistance | 0
  INI, EVG, Intermediate resistance | 0
  INI, EVG, High-level resistance | 0
  INI, RAL,Susceptible | 4
  INI, RAL, Potential low-level resistance | 1
  INI, RAL, Low-level resistance | 0
  INI, RAL, Intermediate resistance | 0
  INI, RAL, High-level resistance | 0
  NNRTI, DLV, Susceptible | 5
  NNRTI, DLV, Potential low-level resistance | 0
  NNRTI,DLV, Low-level resistance | 0
  NNRTI, DLV, Intermediate resistance | 0
  NNRTI, DLV, High-level resistance | 0
  NNRTI, EFV, Susceptible | 3
  NNRTI, EFV, Potential low-level resistance | 0
  NNRTI, EFV, Low-level resistance | 0
  NNRTI, EFV, Intermediate resistance | 1
  NNRTI, EFV, High-level resistance | 1
  NNRTI, ETR, Susceptible | 3
  NNRTI, ETR, Potential low-level resistance | 1
  NNRTI, ETR, Low-level resistance | 0
  NNRTI, ETR, Intermediate resistance | 1
  NNRTI, ETR, High-level resistance | 0
  NNRTI,NVP, Susceptible | 3
  NNRTI,NVP, Potential low-level resistance | 0
  NNRTI,NVP, Low-level resistance | 0
  NNRTI,NVP, Intermediate resistance | 0
  NNRTI, NVP, High-level resistance | 2
  NNRTI, RPV, Susceptible | 3
  NNRTI, RPV, Potential low-level resistance | 0
  NNRTI, RPV, Low-level resistance | 1
  NNRTI, RPV, Intermediate resistance | 0
  NNRTI, RPV, High-level resistance | 1
  NRTI, 3TC, Susceptible | 5
  NRTI, 3TC, Potential low-level resistance | 0
  NRTI, 3TC, Low-level resistance | 0
  NRTI, 3TC, Intermediate resistance | 0
  NRTI, 3TC, High-level resistance | 0
  NRTI, ABC, Susceptible | 5
  NRTI, ABC, Potential low-level resistance | 0
  NRTI, ABC, Low-level resistance | 0
  NRTI, ABC, Intermediate resistance | 0
  NRTI, ABC, High-level resistance | 0
  NRTI, FTC, Susceptible | 5
  NRTI, FTC, Potential low-level resistance | 0
  NRTI, FTC, Low-level resistance | 0
  NRTI, FTC, Intermediate resistance | 0
  NRTI, FTC, High-level resistance | 0
  NRTI, TDF, Susceptible | 5
  NRTI, TDF, Potential low-level resistance | 0
  NRTI, TDF, Low-level resistance | 0
  NRTI, TDF, Intermediate resistance | 0
  NRTI, TDF, High-level resistance | 0
  NRTI, ZDV, Susceptible | 4
  NRTI, ZDV, Potential low-level resistance | 1
  NRTI, ZDV, Low-level resistance | 0
  NRTI, ZDV, Intermediate resistance | 0
  NRTI, ZDV, High-level resistance | 0
  NRTI, d4T, Susceptible | 4
  NRTI, d4T, Potential low-level resistance | 1
  NRTI, d4T, Low-level resistance | 0
  NRTI, d4T, Intermediate resistance | 0
  NRTI, d4T, High-level resistance | 0
  NRTI, ddI, Susceptible | 5
  NRTI, ddI, Potential low-level resistance | 0
  NRTI, ddI, Low-level resistance | 0
  NRTI, ddI, Intermediate resistance | 0
  NRTI, ddI, High-level resistance | 0
  PI, ATV/r, Susceptible | 5
  PI, ATV/r, Potential low-level resistance | 0
  PI, ATV/r, Low-level resistance | 0
  PI, ATV/r, Intermediate resistance | 0
  PI, ATV/r, High-level resistance | 0
  PI, DRV/r, Susceptible | 5
  PI, DRV/r, Potential low-level resistance | 0
  PI, DRV/r, Low-level resistance | 0
  PI, DRV/r, Intermediate resistance | 0
  PI, DRV/r, High-level resistance | 0
  PI, FPV/r, Susceptible | 5
  PI, FPV/r, Potential low-level resistance | 0
  PI, FPV/r, Low-level resistance | 0
  PI, FPV/r, Intermediate resistance | 0
  PI, FPV/r, High-level resistance | 0
  PI, IDV/r, Susceptible | 5
  PI, IDV/r, Potential low-level resistance | 0
  PI, IDV/r, Low-level resistance | 0
  PI, IDV/r, Intermediate resistance | 0
  PI, IDV/r, High-level resistance | 0
  PI, LPV/r, Susceptible | 5
  PI, LPV/r, Potential low-level resistance | 0
  PI, LPV/r, Low-level resistance | 0
  PI, LPV/r, Intermediate resistance | 0
  PI, LPV/r,High-level resistance | 0
  PI, NFV, Susceptible | 5
  PI, NFV, Potential low-level resistance | 0
  PI, NFV, Low-level resistance | 0
  PI, NFV, Intermediate resistance | 0
  PI, NFV, High-level resistance | 0
  PI, RTV, Susceptible | 5
  PI, RTV, Potential low-level resistance | 0
  PI, RTV, Low-level resistance | 0
  PI, RTV, Intermediate resistance | 0
  PI, RTV, High-level resistance | 0
  PI, SQV/r, Susceptible | 5
  PI, SQV/r, Potential low-level resistance | 0
  PI, SQV/r, Low-level resistance | 0
  PI, SQV/r, Intermediate resistance | 0
  PI, SQV/r, High-level resistance | 0
  PI, TPV/r, Susceptible | 5
  PI, TPV/r, Potential low-level resistance | 0
  PI, TPV/r, Low-level resistance | 0
  PI, TPV/r, Intermediate resistance | 0
  PI, TPV/r, High-level resistance | 0

22. Secondary Outcome: Number of Participants With Genotypic Resistance-CAR Group Through Late Switch Phase
Description: Plasma samples were collected for drug resistance testing. Genotypic Resistance data for the following drugs (DTG, EVG, RAL, DLV, EFV, ETR, NVP, RPV, 3TC, ABC, FTC, TDF, ZDV, d4T, ddI, ATV/r, DRV/r, FPV/r, IDV/r, LPV/r, NFV, RTV, SQV/r, TPV/r) in participants Meeting CVW Criteria has been presented.
Time Frame: Post-Late switch (LS) Baseline (Week 52) up to Week 148
Population: The analysis was performed on the Late Switch (LS) CVW resistance Population which was comprised of all participants in the LS-ITT-E Population who met CVW through the end of visit window (Week 48, Week 100 or Week 148) and had available on-treatment genotypic resistance data at the time CVW criterion was met. Only those participants with data available at the specified time point were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 1
Participants
  INI, DTG, Susceptible | 1
  INI, DTG, Potential low-level resistance | 0
  INI, DTG, Low-level resistance | 0
  INI, DTG, Intermediate resistance | 0
  INI, DTG, High-level resistance | 0
  INI, EVG,Susceptible | 1
  INI, EVG, Potential low-level resistance | 0
  INI, EVG,Low-level resistance | 0
  INI, EVG, Intermediate resistance | 0
  INI, EVG, High-level resistance | 0
  INI, RAL,Susceptible | 1
  INI, RAL, Potential low-level resistance | 0
  INI, RAL, Low-level resistance | 0
  INI, RAL, Intermediate resistance | 0
  INI, RAL, High-level resistance | 0
  NNRTI, DLV, Susceptible | 1
  NNRTI, DLV, Potential low-level resistance | 0
  NNRTI,DLV, Low-level resistance | 0
  NNRTI, DLV, Intermediate resistance | 0
  NNRTI, DLV, High-level resistance | 0
  NNRTI, EFV, Susceptible | 0
  NNRTI, EFV, Potential low-level resistance | 1
  NNRTI, EFV, Low-level resistance | 0
  NNRTI, EFV, Intermediate resistance | 0
  NNRTI, EFV, High-level resistance | 0
  NNRTI, ETR, Susceptible | 0
  NNRTI, ETR, Potential low-level resistance | 1
  NNRTI, ETR, Low-level resistance | 0
  NNRTI, ETR, Intermediate resistance | 0
  NNRTI, ETR, High-level resistance | 0
  NNRTI,NVP, Susceptible | 0
  NNRTI,NVP, Potential low-level resistance | 1
  NNRTI,NVP, Low-level resistance | 0
  NNRTI,NVP, Intermediate resistance | 0
  NNRTI, NVP, High-level resistance | 0
  NNRTI, RPV, Susceptible | 0
  NNRTI, RPV, Potential low-level resistance | 1
  NNRTI, RPV, Low-level resistance | 0
  NNRTI, RPV, Intermediate resistance | 0
  NNRTI, RPV, High-level resistance | 0
  NRTI, 3TC, Susceptible | 1
  NRTI, 3TC, Potential low-level resistance | 0
  NRTI, 3TC, Low-level resistance | 0
  NRTI, 3TC, Intermediate resistance | 0
  NRTI, 3TC, High-level resistance | 0
  NRTI, ABC, Susceptible | 1
  NRTI, ABC, Potential low-level resistance | 0
  NRTI, ABC, Low-level resistance | 0
  NRTI, ABC, Intermediate resistance | 0
  NRTI, ABC, High-level resistance | 0
  NRTI, FTC, Susceptible | 1
  NRTI, FTC, Potential low-level resistance | 0
  NRTI, FTC, Low-level resistance | 0
  NRTI, FTC, Intermediate resistance | 0
  NRTI, FTC, High-level resistance | 0
  NRTI, TDF, Susceptible | 1
  NRTI, TDF, Potential low-level resistance | 0
  NRTI, TDF, Low-level resistance | 0
  NRTI, TDF, Intermediate resistance | 0
  NRTI, TDF, High-level resistance | 0
  NRTI, ZDV, Susceptible | 1
  NRTI, ZDV, Potential low-level resistance | 0
  NRTI, ZDV, Low-level resistance | 0
  NRTI, ZDV, Intermediate resistance | 0
  NRTI, ZDV, High-level resistance | 0
  NRTI, d4T, Susceptible | 1
  NRTI, d4T, Potential low-level resistance | 0
  NRTI, d4T, Low-level resistance | 0
  NRTI, d4T, Intermediate resistance | 0
  NRTI, d4T, High-level resistance | 0
  NRTI, ddI, Susceptible | 1
  NRTI, ddI, Potential low-level resistance | 0
  NRTI, ddI, Low-level resistance | 0
  NRTI, ddI, Intermediate resistance | 0
  NRTI, ddI, High-level resistance | 0
  PI, ATV/r, Susceptible | 1
  PI, ATV/r, Potential low-level resistance | 0
  PI, ATV/r, Low-level resistance | 0
  PI, ATV/r, Intermediate resistance | 0
  PI, ATV/r, High-level resistance | 0
  PI, DRV/r, Susceptible | 1
  PI, DRV/r, Potential low-level resistance | 0
  PI, DRV/r, Low-level resistance | 0
  PI, DRV/r, Intermediate resistance | 0
  PI, DRV/r, High-level resistance | 0
  PI, FPV/r, Susceptible | 1
  PI, FPV/r, Potential low-level resistance | 0
  PI, FPV/r, Low-level resistance | 0
  PI, FPV/r, Intermediate resistance | 0
  PI, FPV/r, High-level resistance | 0
  PI, IDV/r, Susceptible | 1
  PI, IDV/r, Potential low-level resistance | 0
  PI, IDV/r, Low-level resistance | 0
  PI, IDV/r, Intermediate resistance | 0
  PI, IDV/r, High-level resistance | 0
  PI, LPV/r, Susceptible | 1
  PI, LPV/r, Potential low-level resistance | 0
  PI, LPV/r, Low-level resistance | 0
  PI, LPV/r, Intermediate resistance | 0
  PI, LPV/r,High-level resistance | 0
  PI, NFV, Susceptible | 1
  PI, NFV, Potential low-level resistance | 0
  PI, NFV, Low-level resistance | 0
  PI, NFV, Intermediate resistance | 0
  PI, NFV, High-level resistance | 0
  PI, RTV, Susceptible | 1
  PI, RTV, Potential low-level resistance | 0
  PI, RTV, Low-level resistance | 0
  PI, RTV, Intermediate resistance | 0
  PI, RTV, High-level resistance | 0
  PI, SQV/r, Susceptible | 1
  PI, SQV/r, Potential low-level resistance | 0
  PI, SQV/r, Low-level resistance | 0
  PI, SQV/r, Intermediate resistance | 0
  PI, SQV/r, High-level resistance | 0
  PI, TPV/r, Susceptible | 1
  PI, TPV/r, Potential low-level resistance | 0
  PI, TPV/r, Low-level resistance | 0
  PI, TPV/r, Intermediate resistance | 0
  PI, TPV/r, High-level resistance | 0

23. Secondary Outcome: Number of Participants With Phenotypic Resistance-Early Switch Phase
Description: Plasma samples were collected for drug resistance testing. Phenotypic Resistance data for the following drugs (DTG, RAL, EVG, RPV, ETR, 3TC, ABC, FTC, TDF, d4T, ddI, ATV/r, DRV/r, FPV/r, IDV/r, LPV/r, SQV/r, TPV/r) in participants Meeting CVW Criteria has been presented.
Time Frame: Up to Week 52
Population: CVW resistance Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 1 | 1
Participants
  INI, DTG, Resistant | 0 | 0
  INI, DTG, Partially Sensitive | 0 | 0
  INI, DTG, Sensitive | 1 | 1
  INI, EVG, Resistant | 0 | 0
  INI, EVG, Sensitive | 1 | 1
  INI, RAL, Resistant | 0 | 0
  INI, RAL, Sensitive | 1 | 1
  NNRTI, DLV, Resistant | 0 | 0
  NNRTI, DLV, Sensitive | 1 | 1
  NNRTI, EFV, Resistant | 0 | 0
  NNRTI, EFV, Sensitive | 1 | 1
  NNRTI, ETR, Resistant | 0 | 0
  NNRTI, ETR, Partially Sensitive | 0 | 0
  NNRTI, ETR, Sensitive | 1 | 1
  NNRTI, NVP, Resistant | 0 | 0
  NNRTI, NVP, Sensitive | 1 | 1
  NNRTI, RPV, Resistant | 0 | 0
  NNRTI, RPV, Sensitive | 1 | 1
  NRTI, 3TC, Resistant | 0 | 0
  NRTI, 3TC, Sensitive | 1 | 1
  NRTI, ABC, Resistant | 0 | 0
  NRTI, ABC, Partially Sensitive | 0 | 0
  NRTI, ABC, Sensitive | 1 | 1
  NRTI,FTC, Resistant | 0 | 0
  NRTI, FTC, Sensitive | 1 | 1
  NRTI, TDF, Resistant | 0 | 0
  NRTI, TDF, Partially Sensitive | 0 | 0
  NRTI, TDF, Sensitive | 1 | 1
  NRTI, ZDV, Resistant | 0 | 0
  NRTI, ZDV, Sensitive | 1 | 1
  NRTI, d4T, Resistant | 0 | 0
  NRTI, d4T, Sensitive | 1 | 1
  NRTI, ddI, Resistant | 0 | 0
  NRTI, ddI, Partially Sensitive | 0 | 0
  NRTI, ddI, Sensitive | 1 | 1
  PI, ATV/r, Resistant | 0 | 0
  PI, ATV/r, Sensitive | 1 | 1
  PI, DRV/r, Resistant | 0 | 0
  PI, DRV/r, Partially Sensitive | 0 | 0
  PI, DRV/r, Sensitive | 1 | 1
  PI, FPV/r, Resistant | 0 | 0
  PI, FPV/r, Partially Sensitive | 0 | 0
  PI, FPV/r, Sensitive | 1 | 1
  PI, IDV/r, Resistant | 0 | 0
  PI, IDV/r, Sensitive | 1 | 1
  PI, LPV/r, Resistant | 0 | 0
  PI, LPV/r, Partially Sensitive | 0 | 0
  PI, LPV/r, Sensitive | 1 | 1
  PI, NFV, Resistant | 0 | 0
  PI, NFV, Sensitive | 1 | 1
  PI, RTV, Resistant | 0 | 0
  PI, RTV, Sensitive | 1 | 1
  PI, SQV/r, Resistant | 0 | 0
  PI, SQV/r, Partially Sensitive | 0 | 0
  PI, SQV/r, Sensitive | 1 | 1
  PI, TPV/r, Resistant | 0 | 0
  PI, TPV/r, Partially Sensitive | 0 | 0
  PI, TPV/r, Sensitive | 1 | 1

24. Secondary Outcome: Number of Participants With Phenotypic Resistance-DTG+RPV Group Through Early and Late Switch Phase
Description: Plasma samples were collected for drug resistance testing. Phenotypic Resistance data for the following drugs (DTG, EVG, RAL, DLV, EFV, ETR, NVP, RPV, 3TC, ABC, FTC, TDF, ZDV, d4T, ddI, ATV/r, DRV/r, FPV/r, IDV/r, LPV/r, NFV, RTV, SQV/r, TPV/r) in participants Meeting CVW Criteria has been presented.
Time Frame: Up to Week 148
Population: CVW resistance Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG + RPV
Number analyzed (Participants) | 5
Participants
  INI, DTG, Resistant | 0
  INI, DTG, Partially Sensitive | 0
  INI, DTG, Sensitive | 5
  INI, EVG, Resistant | 0
  INI, EVG, Partially Sensitive | 0
  INI, EVG, Sensitive | 5
  INI, RAL, Resistant | 0
  INI, RAL, Partially Sensitive | 0
  INI, RAL, Sensitive | 5
  NNRTI, DLV, Resistant | 1
  NNRTI, DLV, Partially Sensitive | 0
  NNRTI, DLV, Sensitive | 4
  NNRTI, EFV, Resistant | 1
  NNRTI, EFV, Partially Sensitive | 0
  NNRTI, EFV, Sensitive | 4
  NNRTI, ETR, Resistant | 0
  NNRTI, ETR, Partially Sensitive | 1
  NNRTI, ETR, Sensitive | 4
  NNRTI, NVP, Resistant | 1
  NNRTI, NVP, Partially Sensitive | 0
  NNRTI, NVP, Sensitive | 4
  NNRTI, RPV, Resistant | 1
  NNRTI, RPV, Partially Sensitive | 0
  NNRTI, RPV, Sensitive | 4
  NRTI, 3TC, Resistant | 0
  NRTI, 3TC, Partially Sensitive | 0
  NRTI, 3TC, Sensitive | 5
  NRTI, ABC, Resistant | 0
  NRTI, ABC, Partially Sensitive | 0
  NRTI, ABC, Sensitive | 5
  NRTI, FTC, Resistant | 0
  NRTI, FTC, Partially Sensitive | 0
  NRTI, FTC, Sensitive | 5
  NRTI, TDF, Resistant | 0
  NRTI, TDF, Partially Sensitive | 0
  NRTI, TDF, Sensitive | 5
  NRTI, ZDV, Resistant | 0
  NRTI, ZDV, Partially Sensitive | 0
  NRTI, ZDV, Sensitive | 5
  NRTI, d4T, Resistant | 0
  NRTI, d4T, Partially Sensitive | 0
  NRTI, d4T, Sensitive | 5
  NRTI, ddI, Resistant | 0
  NRTI, ddI, Partially Sensitive | 0
  NRTI, ddI, Sensitive | 5
  PI, ATV/r, Resistant | 0
  PI, ATV/r, Partially Sensitive | 0
  PI, ATV/r, Sensitive | 5
  PI, DRV/r, Resistant | 0
  PI, DRV/r, Partially Sensitive | 0
  PI, DRV/r, Sensitive | 5
  PI, FPV/r, Resistant | 0
  PI, FPV/r, Partially Sensitive | 0
  PI, FPV/r, Sensitive | 5
  PI, IDV/r, Resistant | 0
  PI, IDV/r, Partially Sensitive | 0
  PI, IDV/r, Sensitive | 5
  PI, LPV/r, Resistant | 0
  PI, LPV/r, Partially Sensitive | 0
  PI, LPV/r, Sensitive | 5
  PI, NFV, Resistant | 0
  PI, NFV, Partially Sensitive | 0
  PI, NFV, Sensitive | 5
  PI, RTV, Resistant | 0
  PI, RTV, Partially Sensitive | 0
  PI, RTV, Sensitive | 5
  PI, SQV/r, Resistant | 0
  PI, SQV/r, Partially Sensitive | 0
  PI, SQV/r, Sensitive | 5
  PI, TPV/r, Resistant | 0
  PI, TPV/r, Partially Sensitive | 0
  PI, TPV/r, Sensitive | 5

25. Secondary Outcome: Number of Participants With Phenotypic Resistance-CAR Group Through Late Switch Phase
Description: Plasma samples were collected for drug resistance testing. Phenotypic Resistance data for the following drugs (DLV, EFV, ETR, NVP, RPV, 3TC, ABC, FTC, TDF, ZDV, d4T, ddI, ATV/r, DRV/r, FPV/r, IDV/r, LPV/r, NFV, RTV, SQV/r, TPV/r) in participants Meeting CVW Criteria has been presented.
Time Frame: Post-LS Baseline (Week 52) up to Week 148
Population: LS CVW resistance Population. Only those participants with data available at the specified time point were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 1
Participants
  NNRTI, DLV, Resistant | 1
  NNRTI, DLV, Partially Sensitive | 0
  NNRTI, DLV, Sensitive | 0
  NNRTI, EFV, Resistant | 1
  NNRTI, EFV, Partially Sensitive | 0
  NNRTI, EFV, Sensitive | 0
  NNRTI, ETR, Resistant | 0
  NNRTI, ETR, Partially Sensitive | 0
  NNRTI, ETR, Sensitive | 1
  NNRTI, NVP, Resistant | 1
  NNRTI, NVP, Partially Sensitive | 0
  NNRTI, NVP, Sensitive | 0
  NNRTI, RPV, Resistant | 0
  NNRTI, RPV, Partially Sensitive | 0
  NNRTI, RPV, Sensitive | 1
  NRTI, 3TC, Resistant | 0
  NRTI, 3TC, Partially Sensitive | 0
  NRTI, 3TC, Sensitive | 1
  NRTI, ABC, Resistant | 0
  NRTI, ABC, Partially Sensitive | 0
  NRTI, ABC, Sensitive | 1
  NRTI, FTC, Resistant | 0
  NRTI, FTC, Partially Sensitive | 0
  NRTI, FTC, Sensitive | 1
  NRTI, TDF, Resistant | 0
  NRTI, TDF, Partially Sensitive | 0
  NRTI, TDF, Sensitive | 1
  NRTI, ZDV, Resistant | 0
  NRTI, ZDV, Partially Sensitive | 0
  NRTI, ZDV, Sensitive | 1
  NRTI, d4T, Resistant | 0
  NRTI, d4T, Partially Sensitive | 0
  NRTI, d4T, Sensitive | 1
  NRTI, ddI, Resistant | 0
  NRTI, ddI, Partially Sensitive | 0
  NRTI, ddI, Sensitive | 1
  PI, ATV/r, Resistant | 0
  PI, ATV/r, Partially Sensitive | 0
  PI, ATV/r, Sensitive | 1
  PI, DRV/r, Resistant | 0
  PI, DRV/r, Partially Sensitive | 0
  PI, DRV/r, Sensitive | 1
  PI, FPV/r, Resistant | 0
  PI, FPV/r, Partially Sensitive | 0
  PI, FPV/r, Sensitive | 1
  PI, IDV/r, Resistant | 0
  PI, IDV/r, Partially Sensitive | 0
  PI, IDV/r, Sensitive | 1
  PI, LPV/r, Resistant | 0
  PI, LPV/r, Partially Sensitive | 0
  PI, LPV/r, Sensitive | 1
  PI, NFV, Resistant | 0
  PI, NFV, Partially Sensitive | 0
  PI, NFV, Sensitive | 1
  PI, RTV, Resistant | 0
  PI, RTV, Partially Sensitive | 0
  PI, RTV, Sensitive | 1
  PI, SQV/r, Resistant | 0
  PI, SQV/r, Partially Sensitive | 0
  PI, SQV/r, Sensitive | 1
  PI, TPV/r, Resistant | 0
  PI, TPV/r, Partially Sensitive | 0
  PI, TPV/r, Sensitive | 1

26. Secondary Outcome: Pre-dose Concentrations of DTG and RPV at Weeks 4, 24, 48, 56, 76 and 100 in Participants Switching to DTG + RPV-DTG+RPV Group Through Early and Late Switch Phase
Description: Two separate blood samples for DTG and RPV were collected pre-dose at Weeks 4, 24, 48, 56, 76, and 100. Pre-dose concentrations of DTG and RPV at Weeks 4, 24, 48, 56, 76 and 100 is summarized for the participants switching to DTG + RPV in the early + late switch phase.
Time Frame: Pre-dose at Week 4, 24, 48, 56, 76 and 100
Population: The analysis was performed on the Pharmacokinetic (PK) Parameter Population which consisted of all participants who received DTG +RPV and provided at least one evaluable estimate of predose concentration (C0). Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: µg/L
Groups:
- DTG 50 mg; RPV 25 mg: Participants received DTG 50 mg + RPV 25 mg together once daily, with a meal, in an open-label fashion up to Week 52 during early switch phase.
Arm/Group | DTG 50 mg | RPV 25 mg
Number analyzed (Participants) | 243 | 243
µg/L
  Week 4: number analyzed (Participants) | 130 | 130
  Week 4 | 1581.06 (1146.860) | 92.05 (138.288)
  Week 24: number analyzed (Participants) | 210 | 210
  Week 24 | 1835.68 (1120.539) | 87.88 (39.141)
  Week 48: number analyzed (Participants) | 215 | 211
  Week 48 | 1915.11 (1304.238) | 95.18 (48.228)
  Week 56: number analyzed (Participants) | 204 | 204
  Week 56 | 1872.65 (1173.815) | 95.38 (53.602)
  Week 76: number analyzed (Participants) | 194 | 194
  Week 76 | 1711.83 (1092.143) | 88.10 (42.250)
  Week 100: number analyzed (Participants) | 203 | 203
  Week 100 | 1854.17 (1197.958) | 92.38 (44.604)

27. Secondary Outcome: Pre-dose Concentrations of DTG and RPV at Weeks 56, 76 and 100 in Participants Switching to DTG+RPV-CAR Group Through Late Switch Phase
Description: Two separate blood samples for DTG and RPV were collected pre-dose at Weeks 56, 76, and 100. Pre-dose concentrations of DTG and RPV at Weeks 56, 76 and 100 is summarized for the participants switching to DTG + RPV in the late switch phase.
Time Frame: Pre-dose at Weeks 56, 76 and 100
Population: The analysis was performed on the LS PK Parameter Population which was comprised of all participants who were randomized to CAR and received DTG + RPV in the Late Switch Phase and provided at least one evaluable estimate of Pre-dose concentration. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: µg/L
Groups:
- CAR-DTG 50 mg: Participants from CAR arm received DTG 50 mg + RPV 25 mg together once daily, with a meal, in an open-label fashion from Week 52 to Week 148 during late switch phase.
- CAR-RPV 25 mg: Participants from CAR arm received DTG 50 mg +RPV 25 mg together once daily, with a meal, in an open-label fashion from Week 52 to Week 148 during late switch phase.
Arm/Group | CAR-DTG 50 mg | CAR-RPV 25 mg
Number analyzed (Participants) | 225 | 225
µg/L
  Week 56: number analyzed (Participants) | 198 | 198
  Week 56 | 1738.55 (1329.931) | 84.14 (47.290)
  Week 76: number analyzed (Participants) | 192 | 192
  Week 76 | 1800.39 (1162.370) | 97.79 (52.532)
  Week 100: number analyzed (Participants) | 192 | 191
  Week 100 | 1907.20 (1235.676) | 101.93 (63.296)

28. Secondary Outcome: Pre-dose Concentrations of DTG and RPV at Weeks 2, 4 and 8 in the First 20 Participants Who Switch From Efavirenz (EFV) or Nevirapine (NVP) to DTG + RPV
Description: Two blood samples were collected pre-dose for DTG and RPV at Weeks 2,4 and 8 only for the first 20 participants who switch from EFV or NVP to DTG + RPV. One blood sample was collected pre-dose for EFV or NVP at Week 2 for the first 20 participants who switch from EFV or NVP to DTG + RPV.
Time Frame: Pre-dose at Week 2, 4 and 8
Population: The analysis was performed on the PK Parameter NNRTI Subset Extra Sampling Population which consisted of the first approximately 20 participants in the PK Parameter NNRTI Subset population who have extra PK samples at weeks 2,4 and 8. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: µg/L
Arm/Group | DTG 50 mg | RPV 25 mg
Number analyzed (Participants) | 26 | 26
µg/L
  Week 2: number analyzed (Participants) | 16 | 15
  Week 2 | 821.25 (574.607) | 65.360 (31.2965)
  Week 4: number analyzed (Participants) | 19 | 19
  Week 4 | 994.00 (581.201) | 67.374 (27.5663)
  Week 8: number analyzed (Participants) | 19 | 19
  Week 8 | 1561.34 (1096.381) | 77.416 (37.7129)

29. Secondary Outcome: Percentage of Participants With Plasma HIV 1 RNA <50 c/mL at Week 48 Using Snapshot Algorithm by Baseline Third Agent Treatment Class
Description: Percentage of participants with plasma HIV 1 RNA < 50 c/mL at Week 48 using the FDA snapshot algorithm was assessed by Baseline third agent class to assess the impact of Baseline third agent class (INI, NNRTI, or PI) on efficacy of DTG +RPV compared to continuation of CAR. Plasma samples were collected for quantitative analysis of HIV-1 RNA. The analysis was done using Cochran-Mantel Haenszel test stratified by current antiretroviral third-agent class and age group.
Time Frame: Week 48
Population: ITT-E Population. Only those participants with data available at the specified time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 252 | 256
Percentage of participants
  NNRTI: number analyzed (Participants) | 131 | 134
  NNRTI | 95 | 98
  INI: number analyzed (Participants) | 46 | 48
  INI | 98 | 96
  PI: number analyzed (Participants) | 75 | 74
  PI | 95 | 92
Statistical Analysis 1: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Other; p = 0.317, Chi-squared, Corrected — One-sided p-value from weighted least squares chi-squared statistic. A p-value <=0.10 was used to indicate statistically significant evidence of heterogeneity in the difference in proportions across levels of each analysis strata
Statistical Analysis 2: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Other; Risk Difference (RD) = -3.1, 95% CI 2-sided [-7.7 to 1.5] — NNRTI: No formal non-inferiority margin has been pre-specified for secondary endpoints
Statistical Analysis 3: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Other; Risk Difference (RD) = 2.0, 95% CI 2-sided [-5.1 to 9.0] — INI: No formal non-inferiority margin has been pre-specified for secondary endpoints
Statistical Analysis 4: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Other; Risk Difference (RD) = 2.8, 95% CI 2-sided [-5.3 to 10.8] — PI: No formal non-inferiority margin has been pre-specified for secondary endpoints

30. Secondary Outcome: Changes From Baseline in Cluster Designation (CD)4+ Lymphocyte Count at Week 48 by Baseline Third Agent Treatment Class
Description: Blood samples were collected for CD4 cell count assessment by flow cytometry was carried out to assess the impact of Baseline third agent class (INI, NNRTI, or PI) on efficacy, safety and tolerability of DTG +RPV compared to continuation of CAR. Value at Day 1 was considered as Baseline. Change from Baseline was calculated as value at indicated time point minus Baseline value.
Time Frame: At Week 48
Population: ITT-E Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Cells per mm^3
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 252 | 256
Cells per mm^3
  NNRTI: number analyzed (Participants) | 124 | 130
  NNRTI | 47.9 (142.90) | 25.0 (151.27)
  INI: number analyzed (Participants) | 45 | 46
  INI | 19.9 (148.63) | 39.9 (200.38)
  PI: number analyzed (Participants) | 70 | 69
  PI | 12.5 (160.27) | 74.7 (227.78)

31. Secondary Outcome: Number of Participants With Any AE, AELD or AE With Grade 1, 2, 3 or 4 Toxicity Over 48 Weeks by Baseline Third Agent Treatment Class
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Number of participants with any AE, AELD or AE with maximum grade toxicity experienced by any one participant over 48 weeks by Baseline third agent class (INI, NNRTI, or PI) was summarized. AEs were graded as per DAIDS grading. Grade 1=mild; grade 2=moderate; grade 3=severe; grade 4=potentially life-threatening.
Time Frame: Up to 48 weeks
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 252 | 256
Participants
  Any AE, NNRTI: number analyzed (Participants) | 131 | 134
  Any AE, NNRTI | 102 | 98
  Any AE, INI: number analyzed (Participants) | 46 | 48
  Any AE, INI | 38 | 34
  Any AE, PI: number analyzed (Participants) | 75 | 74
  Any AE, PI | 60 | 58
  NNRTI, Maximum toxicity Grade 1 AE: number analyzed (Participants) | 131 | 134
  NNRTI, Maximum toxicity Grade 1 AE | 69 | 72
  NNRTI, Maximum toxicity Grade 2 AE: number analyzed (Participants) | 131 | 134
  NNRTI, Maximum toxicity Grade 2 AE | 27 | 23
  NNRTI, Maximum toxicity Grade 3 AE: number analyzed (Participants) | 131 | 134
  NNRTI, Maximum toxicity Grade 3 AE | 5 | 2
  NNRTI, Maximum toxicity Grade 4 AE: number analyzed (Participants) | 131 | 134
  NNRTI, Maximum toxicity Grade 4 AE | 1 | 1
  INI, Maximum toxicity Grade 1 AE: number analyzed (Participants) | 46 | 48
  INI, Maximum toxicity Grade 1 AE | 28 | 20
  INI, Maximum toxicity Grade 2 AE: number analyzed (Participants) | 46 | 48
  INI, Maximum toxicity Grade 2 AE | 7 | 12
  INI, Maximum toxicity Grade 3 AE: number analyzed (Participants) | 46 | 48
  INI, Maximum toxicity Grade 3 AE | 2 | 2
  INI, Maximum toxicity Grade 4 AE: number analyzed (Participants) | 46 | 48
  INI, Maximum toxicity Grade 4 AE | 1 | 0
  PI, Maximum toxicity Grade 1 AE: number analyzed (Participants) | 75 | 74
  PI, Maximum toxicity Grade 1 AE | 31 | 30
  PI, Maximum toxicity Grade 2 AE: number analyzed (Participants) | 75 | 74
  PI, Maximum toxicity Grade 2 AE | 23 | 18
  PI, Maximum toxicity Grade 3 AE: number analyzed (Participants) | 75 | 74
  PI, Maximum toxicity Grade 3 AE | 4 | 9
  PI, Maximum toxicity Grade 4 AE: number analyzed (Participants) | 75 | 74
  PI, Maximum toxicity Grade 4 AE | 2 | 1
  AELD, NNRTI: number analyzed (Participants) | 131 | 134
  AELD, NNRTI | 3 | 0
  AELD, INI: number analyzed (Participants) | 46 | 48
  AELD, INI | 2 | 0
  AELD, PI: number analyzed (Participants) | 75 | 74
  AELD, PI | 4 | 2

32. Secondary Outcome: Number of Participants With Maximum Post-baseline Emergent Chemistry Toxicities Over 48 Weeks by Baseline Third Agent Treatment Class
Description: Blood samples were collected to evaluate ALT, albumin, ALP, AST, total bilirubin, chloride, creatinine, glucose, potassium, phosphate, sodium, BUN, total carbon dioxide, lipase, creatine phosphokinase and creatinine clearance. Value at Day 1 was considered as Baseline. Number of participants who experienced maximum toxicity grade post-Baseline in chemistry parameters over 48 weeks by Baseline third agent treatment class (INI, NNRTI, PI) was summarized. Clinical chemistry toxicities were graded using DAIDS grading table for grading severity of adult and pediatric adverse events. Grade 1=mild; grade 2=moderate; grade 3=severe; grade 4=potentially life-threatening.
Time Frame: Up to 48 weeks
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 252 | 256
Participants
  NNRTI, Grade 1: number analyzed (Participants) | 131 | 134
  NNRTI, Grade 1 | 47 | 42
  NNRTI, Grade 2: number analyzed (Participants) | 131 | 134
  NNRTI, Grade 2 | 32 | 48
  NNRTI, Grade 3: number analyzed (Participants) | 131 | 134
  NNRTI, Grade 3 | 13 | 13
  NNRTI, Grade 4: number analyzed (Participants) | 131 | 134
  NNRTI, Grade 4 | 2 | 3
  INI, Grade 1: number analyzed (Participants) | 46 | 48
  INI, Grade 1 | 13 | 11
  INI, Grade 2: number analyzed (Participants) | 46 | 48
  INI, Grade 2 | 19 | 15
  INI, Grade 3: number analyzed (Participants) | 46 | 48
  INI, Grade 3 | 1 | 1
  INI, Grade 4: number analyzed (Participants) | 46 | 48
  INI, Grade 4 | 3 | 2
  PI, Grade 1: number analyzed (Participants) | 75 | 74
  PI, Grade 1 | 35 | 25
  PI, Grade 2: number analyzed (Participants) | 75 | 74
  PI, Grade 2 | 10 | 23
  PI, Grade 3: number analyzed (Participants) | 75 | 74
  PI, Grade 3 | 8 | 9
  PI, Grade 4: number analyzed (Participants) | 75 | 74
  PI, Grade 4 | 0 | 4

33. Secondary Outcome: Number of Participants With Maximum Post-Baseline Emergent Hematology Toxicities Over 48 Weeks by Baseline Third Agent Treatment Class
Description: Blood samples were collected to evaluate hemoglobin, hematocrit, basophils, eosinophils, lymphocytes, monocytes, neutrophils, MCV, RBC count, WBC count and platelet count. Value at Day 1 was considered as Baseline. Number of participants who experienced maximum toxicity grade post-Baseline in hematology parameters over 48 weeks by Baseline third agent treatment class (INSTI, NNRTI, PI) was summarized. Hematology toxicities were graded using DAIDS grading table for grading severity of adult and pediatric adverse events. Grade 1=mild; grade 2=moderate; grade 3=severe; grade 4=potentially life-threatening.
Time Frame: Up to 48 weeks
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 252 | 256
Participants
  NNRTI; Grade 1: number analyzed (Participants) | 131 | 134
  NNRTI; Grade 1 | 5 | 3
  NNRTI; Grade 2: number analyzed (Participants) | 131 | 134
  NNRTI; Grade 2 | 1 | 1
  NNRTI; Grade 3: number analyzed (Participants) | 131 | 134
  NNRTI; Grade 3 | 1 | 1
  NNRTI; Grade 4: number analyzed (Participants) | 131 | 134
  NNRTI; Grade 4 | 0 | 1
  INI; Grade 1: number analyzed (Participants) | 46 | 48
  INI; Grade 1 | 2 | 2
  INI; Grade 2: number analyzed (Participants) | 46 | 48
  INI; Grade 2 | 1 | 0
  INI; Grade 3: number analyzed (Participants) | 46 | 48
  INI; Grade 3 | 0 | 0
  INI; Grade 4: number analyzed (Participants) | 46 | 48
  INI; Grade 4 | 0 | 0
  PI; Grade 1: number analyzed (Participants) | 75 | 74
  PI; Grade 1 | 4 | 6
  PI; Grade 2: number analyzed (Participants) | 75 | 74
  PI; Grade 2 | 1 | 1
  PI; Grade 3: number analyzed (Participants) | 75 | 74
  PI; Grade 3 | 2 | 0
  PI; Grade 4: number analyzed (Participants) | 75 | 74
  PI; Grade 4 | 0 | 0

34. Secondary Outcome: Number of Participants With Observed Genotypic Resistance for Participants Meeting Virologic Withdrawal Criteria by Baseline Third Agent Treatment Class
Description: For all participants who meet virologic withdrawal criteria, plasma samples with HIV-1 RNA level >=200 c/mL were to be analyzed in an attempt to obtain genotype data on as many samples as possible. Samples for drug resistance testing (genotypic) were to be collected at Day 1. Number of participants with genotypic resistance to CAR and to DTG or RPV for those meeting virologic withdrawal criteria in subgroups stratified based on Baseline third agent treatment class (INSTI, NNRTI, PI) were to be summarized. This outcome has not been analyzed as the number of participants was low (1 CVW per arm) and summaries by Baseline third agent were not provided. Therefore, data are not available for this outcome measure due to the insufficient number of participants with events.
Time Frame: Up to Week 48
Population: CVW resistance Population
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 0 | 0

35. Secondary Outcome: Number of Participants With Observed Phenotypic Resistance for Participants Meeting Virologic Withdrawal Criteria by Baseline Third Agent Treatment Class
Description: For all participants who meet virologic withdrawal criteria, plasma samples with HIV-1 RNA level >=200 c/mL were to be analyzed in an attempt to obtain phenotype data on as many samples as possible. Samples for drug resistance testing (phenotypic) were to be collected at Day 1. Number of participants with phenotypic resistance to CAR and to DTG or RPV for those meeting virologic withdrawal criteria in subgroups stratified based on Baseline third agent treatment class (INSTI, NNRTI, PI) were to be summarized. This outcome was not analyzed as the number of participants was low (1 CVW per arm) and summaries by Baseline third agent were not provided. Therefore, data are not available for this outcome measure due to the insufficient number of participants with events.
Time Frame: Up to Week 48
Population: CVW resistance Population
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 0 | 0

36. Secondary Outcome: Change From Baseline in Fasting Lipids at Weeks 24 and 48 by Baseline Third Agent Treatment Class
Description: Blood samples were collected at Baseline (Day 1), Weeks 24 and 48 to assess fasting lipids which included total cholesterol (CHO), LDL cholesterol, HDL cholesterol and triglycerides. Change from Baseline was calculated as value at indicated time point minus Baseline value.
Time Frame: At Week 24 and at Week 48
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: mmol/mL
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 252 | 256
mmol/mL
  CHO, Week 24, overall: number analyzed (Participants) | 228 | 223
  CHO, Week 24, overall | 3.239 (18.1556) | 2.375 (14.8357)
  CHO, Week 48, overall: number analyzed (Participants) | 221 | 218
  CHO, Week 48, overall | 3.596 (18.7072) | 2.472 (14.7202)
  CHO, Week 24, NNRTI: number analyzed (Participants) | 0 | 118
  CHO, Week 24, NNRTI |  | 3.383 (13.3685)
  CHO, Week 48, NNRTI: number analyzed (Participants) | 0 | 118
  CHO, Week 48, NNRTI |  | 4.099 (13.8992)
  CHO, Week 24, INI: number analyzed (Participants) | 0 | 44
  CHO, Week 24, INI |  | 1.288 (14.8933)
  CHO, Week 48, INI: number analyzed (Participants) | 0 | 43
  CHO, Week 48, INI |  | 0.524 (15.3143)
  CHO, Week 24, PI: number analyzed (Participants) | 0 | 61
  CHO, Week 24, PI |  | 1.211 (17.3972)
  CHO, Week 48, PI: number analyzed (Participants) | 0 | 57
  CHO, Week 48, PI |  | 0.575 (15.7475)
  HDL CHO direct, Overall, Week 24: number analyzed (Participants) | 228 | 223
  HDL CHO direct, Overall, Week 24 | 0.017 (18.7575) | -2.478 (16.6754)
  HDL CHO direct, Overall, Week 48: number analyzed (Participants) | 221 | 218
  HDL CHO direct, Overall, Week 48 | 3.975 (21.1039) | 3.095 (18.8909)
  HDL CHO direct, NNRTI, Week 24: number analyzed (Participants) | 0 | 118
  HDL CHO direct, NNRTI, Week 24 |  | 0.062 (15.9300)
  HDL CHO direct, NNRTI, Week 48: number analyzed (Participants) | 0 | 118
  HDL CHO direct, NNRTI, Week 48 |  | 4.818 (16.2253)
  HDL CHO direct, INI, Week 24: number analyzed (Participants) | 0 | 44
  HDL CHO direct, INI, Week 24 |  | -4.968 (16.2973)
  HDL CHO direct, INI, Week 48: number analyzed (Participants) | 0 | 43
  HDL CHO direct, INI, Week 48 |  | 0.539 (22.6496)
  HDL CHO direct, PI, Week 24: number analyzed (Participants) | 0 | 61
  HDL CHO direct, PI, Week 24 |  | -5.594 (17.7923)
  HDL CHO direct, PI, Week 48: number analyzed (Participants) | 0 | 57
  HDL CHO direct, PI, Week 48 |  | 1.457 (20.8346)
  LDL CHO calculation, Overall, Week 24: number analyzed (Participants) | 224 | 217
  LDL CHO calculation, Overall, Week 24 | 11.504 (36.9087) | 6.196 (24.0104)
  LDL CHO calculation, Overall, Week 48: number analyzed (Participants) | 215 | 211
  LDL CHO calculation, Overall, Week 48 | 8.257 (33.0405) | 3.258 (22.3644)
  LDL CHO calculation, NNRTI, Week 24: number analyzed (Participants) | 0 | 116
  LDL CHO calculation, NNRTI, Week 24 |  | 6.816 (20.9081)
  LDL CHO calculation, NNRTI, Week 48: number analyzed (Participants) | 0 | 114
  LDL CHO calculation, NNRTI, Week 48 |  | 4.920 (20.9300)
  LDL CHO calculation, INI, Week 24: number analyzed (Participants) | 0 | 44
  LDL CHO calculation, INI, Week 24 |  | 6.355 (24.1747)
  LDL CHO calculation, INI, Week 48: number analyzed (Participants) | 0 | 43
  LDL CHO calculation, INI, Week 48 |  | 3.490 (23.3198)
  LDL CHO calculation, PI, Week 24: number analyzed (Participants) | 0 | 57
  LDL CHO calculation, PI, Week 24 |  | 4.813 (29.5705)
  LDL CHO calculation, PI, Week 48: number analyzed (Participants) | 0 | 54
  LDL CHO calculation, PI, Week 48 |  | -0.434 (24.4332)
  Triglycerides, Overall, Week 24: number analyzed (Participants) | 228 | 223
  Triglycerides, Overall, Week 24 | 0.096 (55.6357) | 8.649 (48.8249)
  Triglycerides, Overall, Week 48: number analyzed (Participants) | 221 | 218
  Triglycerides, Overall, Week 48 | 3.605 (54.4914) | 11.068 (54.6321)
  Triglycerides, NNRTI, Week 24: number analyzed (Participants) | 0 | 118
  Triglycerides, NNRTI, Week 24 |  | 6.867 (44.8605)
  Triglycerides, NNRTI, Week 48: number analyzed (Participants) | 0 | 118
  Triglycerides, NNRTI, Week 48 |  | 10.215 (58.4055)
  Triglycerides, INI, Week 24: number analyzed (Participants) | 0 | 44
  Triglycerides, INI, Week 24 |  | 8.386 (54.1265)
  Triglycerides, INI, Week 48: number analyzed (Participants) | 0 | 43
  Triglycerides, INI, Week 48 |  | 4.644 (48.8708)
  Triglycerides, PI, Week 24: number analyzed (Participants) | 0 | 61
  Triglycerides, PI, Week 24 |  | 12.283 (52.6943)
  Triglycerides, PI, Week 48: number analyzed (Participants) | 0 | 57
  Triglycerides, PI, Week 48 |  | 17.681 (50.6912)

37. Secondary Outcome: Change From Baseline in Pre-specified Treatment Symptoms Using the Symptom Distress Module at Weeks 4, 24 and 48-Early Switch Phase
Description: Symptom Distress Module, also called the HIV Symptom Index or Symptoms Impact Questionnaire, is a 20-item self-reported measure that addresses presence and perceived distress linked to symptoms commonly associated with HIV or its treatment. Symptom count is based on which of the 20 symptoms were present in participant. Symptom count is the sum of number of symptoms present and ranges from 0 (none) to 20 (all). Symptom bother score is based on score for each symptom present ranging from 1 (it doesn't bother me) to 4 (it bothers me a lot). Symptom bother score is unweighted sum of the bother item scores for each symptom. Symptom bother score ranges from 0 (minimum bother score) to 80 (maximum bother score). Last observation carried forward (LOCF) was used as primary method of analysis. Change from Baseline was calculated as value at indicated time point minus Baseline value. Day 1 was considered as Baseline value.
Time Frame: At Week 4, Week 24 and Week 48
Population: ITT-E Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 252 | 256
Scores on a scale
  Symptom count, Week 4: number analyzed (Participants) | 212 | 197
  Symptom count, Week 4 | -1.6 (4.19) | 0.2 (4.26)
  Symptom count, Week 24: number analyzed (Participants) | 214 | 201
  Symptom count, Week 24 | -0.8 (5.19) | -0.2 (4.06)
  Symptom count, Week 48: number analyzed (Participants) | 214 | 201
  Symptom count, Week 48 | -0.4 (5.52) | 0.0 (4.49)
  Symptom Bother Score, Week 4: number analyzed (Participants) | 212 | 197
  Symptom Bother Score, Week 4 | -3.0 (7.25) | -0.8 (7.82)
  Symptom Bother Score, Week 24: number analyzed (Participants) | 214 | 201
  Symptom Bother Score, Week 24 | -1.7 (8.47) | -1.3 (8.53)
  Symptom Bother Score, Week 48: number analyzed (Participants) | 214 | 201
  Symptom Bother Score, Week 48 | -1.4 (8.32) | -0.7 (9.03)
Statistical Analysis 1: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Other; p = 0.940, ANCOVA — P-value for interaction between treatment group and Baseline symptom bother score (Week 4)
Statistical Analysis 2: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Superiority; p < .001, ANCOVA — P value to assess difference between treatment groups (Week 4); Mean Difference (Final Values) = -2.924, 95% CI 2-sided [-4.260 to -1.588] — Estimates are calculated from an ANCOVA model adjusting for age, Baseline third agent, gender, race and Baseline score
Statistical Analysis 3: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Other; p = 0.001, ANCOVA — P-value for interaction between treatment group and Baseline symptom bother score (Week 24)
Statistical Analysis 4: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Superiority; p = 0.110, ANCOVA — P value to assess difference between treatment groups (Week 24); Mean Difference (Final Values) = -1.192, 95% CI 2-sided [-2.656 to 0.271] — Estimates are calculated from an ANCOVA model adjusting for age, Baseline third agent, gender, race and Baseline score
Statistical Analysis 5: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Other; p = 0.048, ANCOVA — P-value for interaction between treatment group and Baseline symptom bother score (Week 48)
Statistical Analysis 6: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Superiority; p = 0.038, ANCOVA — P value to assess difference between treatment groups (Week 48); Mean Difference (Final Values) = -1.569, 95% CI 2-sided [-3.048 to -0.090] — Estimates are calculated from an ANCOVA model adjusting for age, Baseline third agent, gender, race and Baseline score

38. Secondary Outcome: Change From Baseline in Pre-specified Treatment Symptoms Using the Symptom Distress Module at Weeks 56, 76, 100 and 148-DTG+RPV Group Through Early and Late Switch Phase
Description: Symptom Distress Module, also called the HIV Symptom Index or Symptoms Impact Questionnaire, is a 20-item self-reported measure that addresses presence and perceived distress linked to symptoms commonly associated with HIV or its treatment. Symptom count is based on which of the 20 symptoms were present in participant. Symptom count is the sum of number of symptoms present and ranges from 0 (none) to 20 (all). Symptom bother score is based on score for each symptom present ranging from 1 (it doesn't bother me) to 4 (it bothers me a lot). Symptom bother score is unweighted sum of the bother item scores for each symptom. Symptom bother score ranges from 0 (minimum bother score) to 80 (maximum bother score).
  LOCF was used as primary method of analysis. Change from Baseline was calculated as value at indicated time point minus Baseline value. Day 1 was considered as Baseline value.
Time Frame: At Week 56, Week 76, Week 100 and Week 148
Population: ITT-E Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | DTG + RPV
Number analyzed (Participants) | 214
Scores on a scale
  Symptom count, Week 56 | -0.9 (4.99)
  Symptom count, Week 76 | -0.2 (5.42)
  Symptom count, Week 100 | -0.4 (5.08)
  Symptom count, Week 148 | -0.6 (5.24)
  Symptom Bother Score, Week 56 | -1.6 (8.52)
  Symptom Bother Score, Week 76 | -0.9 (8.84)
  Symptom Bother Score, Week 100 | -0.8 (8.71)
  Symptom Bother Score, Week 148 | -0.8 (9.15)

39. Secondary Outcome: Change From LS Baseline in Pre-specified Treatment Symptoms Using the Symptom Distress Module at Weeks 56, 76, 100 and 148-CAR Group Through Late Switch Phase
Description: Symptom Distress Module, also called the HIV Symptom Index or Symptoms Impact Questionnaire, is a 20-item self-reported measure that addresses presence and perceived distress linked to symptoms commonly associated with HIV or its treatment. Symptom count is based on which of the 20 symptoms were present in participant. Symptom count is the sum of number of symptoms present and ranges from 0 (none) to 20 (all). Symptom bother score is based on score for each symptom present ranging from 1 (it doesn't bother me) to 4 (it bothers me a lot). Symptom bother score is unweighted sum of the bother item scores for each symptom. Symptom bother score ranges from 0 (minimum bother score) to 80 (maximum bother score). LOCF was used as primary method of analysis. Change from LS Baseline was calculated as value at indicated time point minus LS Baseline value. Value at Week 48 was considered as LS Baseline value.
Time Frame: At Week 56, Week 76, Week 100 and Week 148
Population: LS ITT-E Population comprised of all participants randomized to CAR who received at least one dose of study treatment at or after the Week 52 Switch visit. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 238
Scores on a scale
  Symptom count, Week 56: number analyzed (Participants) | 186
  Symptom count, Week 56 | -0.7 (4.38)
  Symptom count, Week 76: number analyzed (Participants) | 188
  Symptom count, Week 76 | 0.1 (4.19)
  Symptom count, Week 100: number analyzed (Participants) | 188
  Symptom count, Week 100 | 0.0 (4.35)
  Symptom count, Week 148: number analyzed (Participants) | 188
  Symptom count, Week 148 | 0.4 (4.92)
  Symptom Bother Score, Week 56: number analyzed (Participants) | 186
  Symptom Bother Score, Week 56 | -2.0 (8.11)
  Symptom Bother Score, Week 76: number analyzed (Participants) | 188
  Symptom Bother Score, Week 76 | -0.4 (8.33)
  Symptom Bother Score, Week 100: number analyzed (Participants) | 188
  Symptom Bother Score, Week 100 | -0.4 (9.17)
  Symptom Bother Score, Week 148: number analyzed (Participants) | 188
  Symptom Bother Score, Week 148 | 0.7 (9.57)

40. Secondary Outcome: Change From Baseline Treatment Satisfaction Using the HIV Treatment Satisfaction Questionnaire (HIV TSQ) at Weeks 4, 24 and 48-Early Switch Phase
Description: HIV TSQ is a 10-item self-reported scale that measures overall satisfaction with treatment and by specific domains e.g., convenience, flexibility. Each item is scored 0 (very dissatisfied, inconvenient) to 6 (very satisfied, convenient). The items are summed up to produce a treatment satisfaction total score (0 to 60) and 2 subscale scores: general satisfaction/clinical and lifestyle/ease subscales (0 to 30). Higher scores indicated greater treatment satisfaction as compared to the past few weeks. The HIV TSQ was administered as a paper questionnaire. Total score, lifestyle/ease score and General satisfaction/CS have been summarized. LOCF was used as primary method of analysis. Value obtained at Day 1 was considered as Baseline value. Change from Baseline was calculated as value at indicated time point minus Baseline value.
Time Frame: At Week 4, Week 24 and Week 48
Population: ITT-E Population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | DTG + RPV | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 252 | 256
Scores on a scale
  Total score, Week 4: number analyzed (Participants) | 250 | 249
  Total score, Week 4 | 0.0 [-16 to 33] | 0.0 [-25 to 21]
  Total score, Week 24: number analyzed (Participants) | 252 | 254
  Total score, Week 24 | 1.0 [-18 to 33] | 0.0 [-28 to 28]
  Total score, Week 48: number analyzed (Participants) | 252 | 254
  Total score, Week 48 | 0.5 [-24 to 33] | 0.0 [-28 to 20]
  lifestyle/ease Sub-score, Week 4: number analyzed (Participants) | 248 | 249
  lifestyle/ease Sub-score, Week 4 | 0.0 [-7 to 15] | 0.0 [-9 to 13]
  lifestyle/ease Sub-score, Week 24: number analyzed (Participants) | 252 | 254
  lifestyle/ease Sub-score, Week 24 | 0.0 [-11 to 15] | 0.0 [-14 to 12]
  lifestyle/ease Sub-score, Week 48: number analyzed (Participants) | 252 | 254
  lifestyle/ease Sub-score, Week 48 | 0.0 [-13 to 16] | 0.0 [-14 to 13]
  General Satisfaction/CS, Week 4: number analyzed (Participants) | 249 | 249
  General Satisfaction/CS, Week 4 | 0.0 [-10 to 18] | 0.0 [-16 to 13]
  General Satisfaction/CS, Week 24: number analyzed (Participants) | 252 | 254
  General Satisfaction/CS, Week 24 | 0.0 [-7 to 18] | 0.0 [-14 to 17]
  General Satisfaction/CS, Week 48: number analyzed (Participants) | 252 | 254
  General Satisfaction/CS, Week 48 | 0.0 [-14 to 18] | 0.0 [-14 to 10]
Statistical Analysis 1: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Superiority; p = 0.002, Wilcoxon rank sum test — P-value to assess HIVTSQs Total Score difference between treatment groups (Week 4)
Statistical Analysis 2: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Superiority; p < 0.001, Wilcoxon rank sum test — P-value to assess HIVTSQs Total Score difference between treatment groups (Week 24)
Statistical Analysis 3: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Superiority; p = 0.024, Wilcoxon rank sum test — P-value to assess HIVTSQs Total score difference between treatment groups (Week 48)
Statistical Analysis 4: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Superiority; p < 0.001, Wilcoxon rank sum test — P-value to assess HIVTSQs lifestyle/ease sub- score difference between treatment groups (Week 4)
Statistical Analysis 5: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Superiority; p < 0.001, Wilcoxon rank sum test — P-value to assess HIVTSQs lifestyle/ease sub- score difference between treatment groups (Week 24)
Statistical Analysis 6: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Superiority; p = 0.005, Wilcoxon rank sum test — P-value to assess HIVTSQs lifestyle/ease sub- score difference between treatment groups (Week 48)
Statistical Analysis 7: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Superiority; p = 0.063, Wilcoxon rank sum test — P-value to assess HIVTSQs General satisfaction/CS sub- score difference between treatment groups (Week 4)
Statistical Analysis 8: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Superiority; p = 0.002, Wilcoxon rank sum test — P-value to assess HIVTSQs General satisfaction/CS sub- score difference between treatment groups (Week 24)
Statistical Analysis 9: Comparison: DTG + RPV vs Current Antiretroviral Regimen (CAR); Test type: Superiority; p = 0.099, Wilcoxon rank sum test — P-value to assess HIVTSQs General satisfaction/CS sub- score difference between treatment groups (Week 48)

41. Secondary Outcome: Change From Baseline Treatment Satisfaction Using HIV TSQ at Weeks 56, 76, 100 and 148 - DTG+RPV Group Through Early and Late Switch Phase
Description: as for outcome 40
Time Frame: At Week 56, Week 76, Week 100 and Week 148
Population: ITT-E Population
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | DTG + RPV
Number analyzed (Participants) | 252
Scores on a scale
  Total score, Week 56 | 0.0 [-42 to 33]
  Total score, Week 76 | 0.5 [-35 to 33]
  Total score, Week 100 | 0.0 [-17 to 33]
  Total score, Week 148 | 1.0 [-23 to 32]
  Lifestyle/ease Sub-score, Week 56 | 0.0 [-23 to 16]
  Lifestyle/ease Sub-score, Week 76 | 0.0 [-19 to 16]
  Lifestyle/ease Sub-score, Week 100 | 0.0 [-13 to 16]
  Lifestyle/ease Sub-score, Week 148 | 0.0 [-13 to 15]
  General Satisfaction/CS, Week 56 | 0.0 [-19 to 18]
  General Satisfaction/CS, Week 76 | 0.0 [-16 to 17]
  General Satisfaction/CS, Week 100 | 0.0 [-13 to 17]
  General Satisfaction/CS, Week 148 | 0.0 [-12 to 17]

42. Secondary Outcome: Change From LS Baseline Treatment Satisfaction Using HIV TSQ at Weeks 56, 76, 100 and 148-CAR Group Through Late Switch Phase
Description: HIV TSQ is a 10-item self-reported scale that measures overall satisfaction with treatment and by specific domains e.g., convenience, flexibility. Each item is scored 0 (very dissatisfied, inconvenient) to 6 (very satisfied, convenient). The items are summed up to produce a treatment satisfaction total score (0 to 60) and 2 subscale scores: general satisfaction/clinical and lifestyle/ease subscales (0 to 30). Higher scores indicated greater treatment satisfaction as compared to the past few weeks. The HIV TSQ was administered as a paper questionnaire. Total score, lifestyle/ease score and General satisfaction/CS have been summarized. LOCF was used as primary method of analysis. Value obtained at Week 48 was considered as LS Baseline value. Change from LS Baseline was calculated as value at indicated time point minus LS Baseline value.
Time Frame: At Week 56, Week 76, Week 100 and Week 148
Population: LS ITT-E Population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 236
Scores on a scale
  Total score, Week 56 | 0.0 [-31 to 31]
  Total score, Week 76 | 0.0 [-37 to 31]
  Total score, Week 100 | 0.0 [-37 to 26]
  Total score, Week 148 | 0.0 [-37 to 26]
  Lifestyle/ease Sub-score, Week 56 | 0.0 [-14 to 16]
  Lifestyle/ease Sub-score, Week 76 | 0.0 [-21 to 16]
  Lifestyle/ease Sub-score, Week 100 | 0.0 [-21 to 18]
  Lifestyle/ease Sub-score, Week 148 | 0.0 [-21 to 16]
  General Satisfaction/CS, Week 56 | 0.0 [-17 to 16]
  General Satisfaction/CS, Week 76 | 0.0 [-17 to 16]
  General Satisfaction/CS, Week 100 | 0.0 [-17 to 14]
  General Satisfaction/CS, Week 148 | 0.0 [-17 to 13]

43. Other Pre Specified Outcome: Percentage of Participants With Plasma HIV-1 RNA <50 c/mL at Weeks 100 and 148 Using the Snapshot Algorithm-DTG+RPV Group Through Early and Late Switch Phase
Description: Plasma samples were collected for quantitative analysis of HIV-1 RNA. Percentage of participants with plasma HIV 1 RNA < 50 c/mL using the FDA snapshot algorithm was assessed. Virologic success or failure was determined by the last available HIV-1 RNA assessment while the participant was on-treatment within the window of the visit of interest.
Time Frame: At Weeks 100 and 148
Population: ITT-E Population
Measure: Number; unit: Percentage of participants
Arm/Group | DTG + RPV
Number analyzed (Participants) | 252
Percentage of participants
  Week 100 | 88
  Week 148 | 85

44. Other Pre Specified Outcome: Change From Baseline in CD4+ Lymphocyte Count at Weeks 100 and 148-DTG+RPV Group Through Early and Late Switch Phase
Description: Blood samples were collected for CD4+ cell count assessment by flow cytometry. Change from Baseline was calculated as value at indicated time point minus Baseline value.
Time Frame: At Weeks 100 and 148
Population: ITT-E Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Cells/mm^3
Arm/Group | DTG + RPV
Number analyzed (Participants) | 252
Cells/mm^3
  Week 100: number analyzed (Participants) | 224
  Week 100 | 25.1 (156.31)
  Week 148: number analyzed (Participants) | 212
  Week 148 | 39.9 (174.40)

45. Other Pre Specified Outcome: Percentage of Participants With Plasma HIV-1 RNA <50 c/mL at Weeks 100 and 148 Using the Snapshot Algorithm-CAR Group Through Late Switch Phase
Description: as for outcome 43
Time Frame: At Weeks 100 and 148
Population: LS ITT-E Population
Measure: Number; unit: Percentage of participants
Arm/Group | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 238
Percentage of participants
  Week 100 | 90
  Week 148 | 87

46. Other Pre Specified Outcome: Change From LS Baseline in CD4+ Lymphocyte Count at Weeks 100 and 148-CAR Group Through Late Switch Phase
Description: Blood samples were collected for CD4+ cell count assessment by flow cytometry. Change from LS Baseline was calculated as value at indicated time point minus LS Baseline value.
Time Frame: At Weeks 100 and 148
Population: LS ITT-E Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Cells/mm^3
Arm/Group | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 238
Cells/mm^3
  Week 100: number analyzed (Participants) | 217
  Week 100 | -3.3 (180.82)
  Week 148: number analyzed (Participants) | 207
  Week 148 | 3.7 (205.29)

47. Secondary Outcome: Number of Participants With Observed Genotypic Resistance for Participants Meeting Virologic Withdrawal Criteria by Baseline Third Agent Treatment Class-DTG+RPV Group Through Continuation Phase
Description: For all participants who met virologic withdrawal criteria, plasma samples with HIV-1 RNA level >=200 c/mL were analyzed in an attempt to obtain genotype data on as many samples as possible. Samples for drug resistance testing (genotypic) were collected at Day 1. Number of participants with genotypic resistance to DTG or RPV for those meeting virologic withdrawal criteria in subgroups, stratified based on baseline third agent treatment class (NNRTI, INI, PI) were summarized.
Time Frame: Up to Week 411
Population: The analysis was performed on the CVW Resistance population.
Measure: Count of Participants; unit: Participants
Arm/Group | DTG + RPV
Number analyzed (Participants) | 3
Participants
  NNRTI, INI, DTG, Susceptible | 3
  NNRTI, INI, DTG, Potential low-level resistance | 0
  NNRTI, INI, DTG, Low-level resistance | 0
  NNRTI, INI, DTG, Intermediate resistance | 0
  NNRTI, INI, DTG, High-level resistance | 0
  NNRTI, INI, EVG, Susceptible | 3
  NNRTI, INI, EVG, Potential low-level resistance | 0
  NNRTI, INI, EVG, Low-level resistance | 0
  NNRTI, INI, EVG, Intermediate resistance | 0
  NNRTI, INI, EVG, High-level resistance | 0
  NNRTI, INI, RAL, Susceptible | 3
  NNRTI, INI, RAL, Potential low-level resistance | 0
  NNRTI, INI, RAL, Low-level resistance | 0
  NNRTI, INI, RAL, Intermediate resistance | 0
  NNRTI, INI, RAL, High-level resistance | 0
  NNRTI, NNRTI, DLV, Susceptible | 3
  NNRTI, NNRTI, DLV, Potential low-level resistance | 0
  NNRTI, NNRTI, DLV, Low-level resistance | 0
  NNRTI, NNRTI, DLV, Intermediate resistance | 0
  NNRTI, NNRTI, DLV, High-level resistance | 0
  NNRTI, NNRTI, EFV, Susceptible | 1
  NNRTI, NNRTI, EFV, Potential low-level resistance | 0
  NNRTI, NNRTI, EFV, Low-level resistance | 1
  NNRTI, NNRTI, EFV, Intermediate resistance | 0
  NNRTI, NNRTI, EFV, High-level resistance | 1
  NNRTI, NNRTI, ETR, Susceptible | 2
  NNRTI, NNRTI, ETR, Potential low-level resistance | 0
  NNRTI, NNRTI, ETR, Low-level resistance | 1
  NNRTI, NNRTI, ETR, Intermediate resistance | 0
  NNRTI, NNRTI, ETR, High-level resistance | 0
  NNRTI, NNRTI, NVP, Susceptible | 1
  NNRTI, NNRTI, NVP, Potential low-level resistance | 0
  NNRTI, NNRTI, NVP, Low-level resistance | 0
  NNRTI, NNRTI, NVP, Intermediate resistance | 1
  NNRTI, NNRTI, NVP, High-level resistance | 1
  NNRTI, NNRTI, RPV, Susceptible | 2
  NNRTI, NNRTI, RPV, Potential low-level resistance | 0
  NNRTI, NNRTI, RPV, Low-level resistance | 0
  NNRTI, NNRTI, RPV, Intermediate resistance | 0
  NNRTI, NNRTI, RPV, High-level resistance | 1
  NNRTI, NRTI, 3TC, Susceptible | 2
  NNRTI, NRTI, 3TC, Potential low-level resistance | 0
  NNRTI, NRTI, 3TC, Low-level resistance | 0
  NNRTI, NRTI, 3TC, Intermediate resistance | 1
  NNRTI, NRTI, 3TC, High-level resistance | 0
  NNRTI, NRTI, ABC, Susceptible | 2
  NNRTI, NRTI, ABC, Potential low-level resistance | 0
  NNRTI, NRTI, ABC, Low-level resistance | 0
  NNRTI, NRTI, ABC, Intermediate resistance | 0
  NNRTI, NRTI, ABC, High-level resistance | 1
  NNRTI, NRTI, FTC, Susceptible | 2
  NNRTI, NRTI, FTC, Potential low-level resistance | 0
  NNRTI, NRTI, FTC, Low-level resistance | 0
  NNRTI, NRTI, FTC, Intermediate resistance | 1
  NNRTI, NRTI, FTC, High-level resistance | 0
  NNRTI, NRTI, TDF, Susceptible | 2
  NNRTI, NRTI, TDF, Potential low-level resistance | 0
  NNRTI, NRTI, TDF, Low-level resistance | 0
  NNRTI, NRTI, TDF, Intermediate resistance | 0
  NNRTI, NRTI, TDF, High-level resistance | 1
  NNRTI, NRTI, ZDV, Susceptible | 1
  NNRTI, NRTI, ZDV, Potential low-level resistance | 1
  NNRTI, NRTI, ZDV, Low-level resistance | 0
  NNRTI, NRTI, ZDV, Intermediate resistance | 0
  NNRTI, NRTI, ZDV, High-level resistance | 1
  NNRTI, NRTI, d4T, Susceptible | 1
  NNRTI, NRTI, d4T, Potential low-level resistance | 1
  NNRTI, NRTI, d4T, Low-level resistance | 0
  NNRTI, NRTI, d4T, Intermediate resistance | 0
  NNRTI, NRTI, d4T, High-level resistance | 1
  NNRTI, NRTI, ddI, Susceptible | 2
  NNRTI, NRTI, ddI, Potential low-level resistance | 0
  NNRTI, NRTI, ddI, Low-level resistance | 0
  NNRTI, NRTI, ddI, Intermediate resistance | 0
  NNRTI, NRTI, ddI, High-level resistance | 1
  NNRTI, PI, ATV/r, Susceptible | 3
  NNRTI, PI, ATV/r, Potential low-level resistance | 0
  NNRTI, PI, ATV/r, Low-level resistance | 0
  NNRTI, PI, ATV/r, Intermediate resistance | 0
  NNRTI, PI, ATV/r, High-level resistance | 0
  NNRTI, PI, DRV/r, Susceptible | 3
  NNRTI, PI, DRV/r, Potential low-level resistance | 0
  NNRTI, PI, DRV/r, Low-level resistance | 0
  NNRTI, PI, DRV/r, Intermediate resistance | 0
  NNRTI, PI, DRV/r, High-level resistance | 0
  NNRTI, PI, FPV/r, Susceptible | 3
  NNRTI, PI, FPV/r, Potential low-level resistance | 0
  NNRTI, PI, FPV/r, Low-level resistance | 0
  NNRTI, PI, FPV/r, Intermediate resistance | 0
  NNRTI, PI, FPV/r, High-level resistance | 0
  NNRTI, PI, IDV/r, Susceptible | 3
  NNRTI, PI, IDV/r, Potential low-level resistance | 0
  NNRTI, PI, IDV/r, Low-level resistance | 0
  NNRTI, PI, IDV/r, Intermediate resistance | 0
  NNRTI, PI, IDV/r, High-level resistance | 0
  NNRTI, PI, LPV/r, Susceptible | 3
  NNRTI, PI, LPV/r, Potential low-level resistance | 0
  NNRTI, PI, LPV/r, Low-level resistance | 0
  NNRTI, PI, LPV/r, Intermediate resistance | 0
  NNRTI, PI, LPV/r, High-level resistance | 0
  NNRTI, PI, NFV, Susceptible | 3
  NNRTI, PI, NFV, Potential low-level resistance | 0
  NNRTI, PI, NFV, Low-level resistance | 0
  NNRTI, PI, NFV, Intermediate resistance | 0
  NNRTI, PI, NFV, High-level resistance | 0
  NNRTI, PI, RTV, Susceptible | 3
  NNRTI, PI, RTV, Potential low-level resistance | 0
  NNRTI, PI, RTV, Low-level resistance | 0
  NNRTI, PI, RTV, Intermediate resistance | 0
  NNRTI, PI, RTV, High-level resistance | 0
  NNRTI, PI, SQV/r, Susceptible | 3
  NNRTI, PI, SQV/r, Potential low-level resistance | 0
  NNRTI, PI, SQV/r, Low-level resistance | 0
  NNRTI, PI, SQV/r, Intermediate resistance | 0
  NNRTI, PI, SQV/r, High-level resistance | 0
  NNRTI, PI, TPV/r, Susceptible | 3
  NNRTI, PI, TPV/r, Potential low-level resistance | 0
  NNRTI, PI, TPV/r, Low-level resistance | 0
  NNRTI, PI, TPV/r, Intermediate resistance | 0
  NNRTI, PI, TPV/r, High-level resistance | 0
  INI, INI, DTG, Susceptible: number analyzed (Participants) | 2
  INI, INI, DTG, Susceptible | 2
  INI, INI, DTG, Potential low-level resistance: number analyzed (Participants) | 2
  INI, INI, DTG, Potential low-level resistance | 0
  INI, INI, DTG, Low-level resistance: number analyzed (Participants) | 2
  INI, INI, DTG, Low-level resistance | 0
  INI, INI, DTG, Intermediate resistance: number analyzed (Participants) | 2
  INI, INI, DTG, Intermediate resistance | 0
  INI, INI, DTG, High-level resistance: number analyzed (Participants) | 2
  INI, INI, DTG, High-level resistance | 0
  INI, INI, EVG, Susceptible: number analyzed (Participants) | 2
  INI, INI, EVG, Susceptible | 1
  INI, INI, EVG, Potential low-level resistance: number analyzed (Participants) | 2
  INI, INI, EVG, Potential low-level resistance | 1
  INI, INI, EVG, Low-level resistance: number analyzed (Participants) | 2
  INI, INI, EVG, Low-level resistance | 0
  INI, INI, EVG, Intermediate resistance: number analyzed (Participants) | 2
  INI, INI, EVG, Intermediate resistance | 0
  INI, INI, EVG, High-level resistance: number analyzed (Participants) | 2
  INI, INI, EVG, High-level resistance | 0
  INI, INI, RAL, Susceptible: number analyzed (Participants) | 2
  INI, INI, RAL, Susceptible | 1
  INI, INI, RAL, Potential low-level resistance: number analyzed (Participants) | 2
  INI, INI, RAL, Potential low-level resistance | 1
  INI, INI, RAL, Low-level resistance: number analyzed (Participants) | 2
  INI, INI, RAL, Low-level resistance | 0
  INI, INI, RAL, Intermediate resistance: number analyzed (Participants) | 2
  INI, INI, RAL, Intermediate resistance | 0
  INI, INI, RAL, High-level resistance: number analyzed (Participants) | 2
  INI, INI, RAL, High-level resistance | 0
  INI, NNRTI, DLV, Susceptible: number analyzed (Participants) | 2
  INI, NNRTI, DLV, Susceptible | 2
  INI, NNRTI, DLV, Potential low-level resistance: number analyzed (Participants) | 2
  INI, NNRTI, DLV, Potential low-level resistance | 0
  INI, NNRTI, DLV, Low-level resistance: number analyzed (Participants) | 2
  INI, NNRTI, DLV, Low-level resistance | 0
  INI, NNRTI, DLV, Intermediate resistance: number analyzed (Participants) | 2
  INI, NNRTI, DLV, Intermediate resistance | 0
  INI, NNRTI, DLV, High-level resistance: number analyzed (Participants) | 2
  INI, NNRTI, DLV, High-level resistance | 0
  INI, NNRTI, EFV, Susceptible: number analyzed (Participants) | 2
  INI, NNRTI, EFV, Susceptible | 1
  INI, NNRTI, EFV, Potential low-level resistance: number analyzed (Participants) | 2
  INI, NNRTI, EFV, Potential low-level resistance | 0
  INI, NNRTI, EFV, Low-level resistance: number analyzed (Participants) | 2
  INI, NNRTI, EFV, Low-level resistance | 0
  INI, NNRTI, EFV, Intermediate resistance: number analyzed (Participants) | 2
  INI, NNRTI, EFV, Intermediate resistance | 1
  INI, NNRTI, EFV, High-level resistance: number analyzed (Participants) | 2
  INI, NNRTI, EFV, High-level resistance | 0
  INI, NNRTI, ETR, Susceptible: number analyzed (Participants) | 2
  INI, NNRTI, ETR, Susceptible | 0
  INI, NNRTI, ETR, Potential low-level resistance: number analyzed (Participants) | 2
  INI, NNRTI, ETR, Potential low-level resistance | 1
  INI, NNRTI, ETR, Low-level resistance: number analyzed (Participants) | 2
  INI, NNRTI, ETR, Low-level resistance | 0
  INI, NNRTI, ETR, Intermediate resistance: number analyzed (Participants) | 2
  INI, NNRTI, ETR, Intermediate resistance | 1
  INI, NNRTI, ETR, High-level resistance: number analyzed (Participants) | 2
  INI, NNRTI, ETR, High-level resistance | 0
  INI, NNRTI, NVP, Susceptible: number analyzed (Participants) | 2
  INI, NNRTI, NVP, Susceptible | 1
  INI, NNRTI, NVP, Potential low-level resistance: number analyzed (Participants) | 2
  INI, NNRTI, NVP, Potential low-level resistance | 0
  INI, NNRTI, NVP, Low-level resistance: number analyzed (Participants) | 2
  INI, NNRTI, NVP, Low-level resistance | 0
  INI, NNRTI, NVP, Intermediate resistance: number analyzed (Participants) | 2
  INI, NNRTI, NVP, Intermediate resistance | 0
  INI, NNRTI, NVP, High-level resistance: number analyzed (Participants) | 2
  INI, NNRTI, NVP, High-level resistance | 1
  INI, NNRTI, RPV, Susceptible: number analyzed (Participants) | 2
  INI, NNRTI, RPV, Susceptible | 0
  INI, NNRTI, RPV, Potential low-level resistance: number analyzed (Participants) | 2
  INI, NNRTI, RPV, Potential low-level resistance | 0
  INI, NNRTI, RPV, Low-level resistance: number analyzed (Participants) | 2
  INI, NNRTI, RPV, Low-level resistance | 1
  INI, NNRTI, RPV, Intermediate resistance: number analyzed (Participants) | 2
  INI, NNRTI, RPV, Intermediate resistance | 0
  INI, NNRTI, RPV, High-level resistance: number analyzed (Participants) | 2
  INI, NNRTI, RPV, High-level resistance | 1
  INI, NRTI, 3TC, Susceptible: number analyzed (Participants) | 2
  INI, NRTI, 3TC, Susceptible | 2
  INI, NRTI, 3TC, Potential low-level resistance: number analyzed (Participants) | 2
  INI, NRTI, 3TC, Potential low-level resistance | 0
  INI, NRTI, 3TC, Low-level resistance: number analyzed (Participants) | 2
  INI, NRTI, 3TC, Low-level resistance | 0
  INI, NRTI, 3TC, Intermediate resistance: number analyzed (Participants) | 2
  INI, NRTI, 3TC, Intermediate resistance | 0
  INI, NRTI, 3TC, High-level resistance: number analyzed (Participants) | 2
  INI, NRTI, 3TC, High-level resistance | 0
  INI, NRTI, ABC, Susceptible: number analyzed (Participants) | 2
  INI, NRTI, ABC, Susceptible | 2
  INI, NRTI, ABC, Potential low-level resistance: number analyzed (Participants) | 2
  INI, NRTI, ABC, Potential low-level resistance | 0
  INI, NRTI, ABC, Low-level resistance: number analyzed (Participants) | 2
  INI, NRTI, ABC, Low-level resistance | 0
  INI, NRTI, ABC, Intermediate resistance: number analyzed (Participants) | 2
  INI, NRTI, ABC, Intermediate resistance | 0
  INI, NRTI, ABC, High-level resistance: number analyzed (Participants) | 2
  INI, NRTI, ABC, High-level resistance | 0
  INI, NRTI, FTC, Susceptible: number analyzed (Participants) | 2
  INI, NRTI, FTC, Susceptible | 2
  INI, NRTI, FTC, Potential low-level resistance: number analyzed (Participants) | 2
  INI, NRTI, FTC, Potential low-level resistance | 0
  INI, NRTI, FTC, Low-level resistance: number analyzed (Participants) | 2
  INI, NRTI, FTC, Low-level resistance | 0
  INI, NRTI, FTC, Intermediate resistance: number analyzed (Participants) | 2
  INI, NRTI, FTC, Intermediate resistance | 0
  INI, NRTI, FTC, High-level resistance: number analyzed (Participants) | 2
  INI, NRTI, FTC, High-level resistance | 0
  INI, NRTI, TDF, Susceptible: number analyzed (Participants) | 2
  INI, NRTI, TDF, Susceptible | 2
  INI, NRTI, TDF, Potential low-level resistance: number analyzed (Participants) | 2
  INI, NRTI, TDF, Potential low-level resistance | 0
  INI, NRTI, TDF, Low-level resistance: number analyzed (Participants) | 2
  INI, NRTI, TDF, Low-level resistance | 0
  INI, NRTI, TDF, Intermediate resistance: number analyzed (Participants) | 2
  INI, NRTI, TDF, Intermediate resistance | 0
  INI, NRTI, TDF, High-level resistance: number analyzed (Participants) | 2
  INI, NRTI, TDF, High-level resistance | 0
  INI, NRTI, ZDV, Susceptible: number analyzed (Participants) | 2
  INI, NRTI, ZDV, Susceptible | 2
  INI, NRTI, ZDV, Potential low-level resistance: number analyzed (Participants) | 2
  INI, NRTI, ZDV, Potential low-level resistance | 0
  INI, NRTI, ZDV, Low-level resistance: number analyzed (Participants) | 2
  INI, NRTI, ZDV, Low-level resistance | 0
  INI, NRTI, ZDV, Intermediate resistance: number analyzed (Participants) | 2
  INI, NRTI, ZDV, Intermediate resistance | 0
  INI, NRTI, ZDV, High-level resistance: number analyzed (Participants) | 2
  INI, NRTI, ZDV, High-level resistance | 0
  INI, NRTI, d4T, Susceptible: number analyzed (Participants) | 2
  INI, NRTI, d4T, Susceptible | 2
  INI, NRTI, d4T, Potential low-level resistance: number analyzed (Participants) | 2
  INI, NRTI, d4T, Potential low-level resistance | 0
  INI, NRTI, d4T, Low-level resistance: number analyzed (Participants) | 2
  INI, NRTI, d4T, Low-level resistance | 0
  INI, NRTI, d4T, Intermediate resistance: number analyzed (Participants) | 2
  INI, NRTI, d4T, Intermediate resistance | 0
  INI, NRTI, d4T, High-level resistance: number analyzed (Participants) | 2
  INI, NRTI, d4T, High-level resistance | 0
  INI, NRTI, ddI, Susceptible: number analyzed (Participants) | 2
  INI, NRTI, ddI, Susceptible | 2
  INI, NRTI, ddI, Potential low-level resistance: number analyzed (Participants) | 2
  INI, NRTI, ddI, Potential low-level resistance | 0
  INI, NRTI, ddI, Low-level resistance: number analyzed (Participants) | 2
  INI, NRTI, ddI, Low-level resistance | 0
  INI, NRTI, ddI, Intermediate resistance: number analyzed (Participants) | 2
  INI, NRTI, ddI, Intermediate resistance | 0
  INI, NRTI, ddI, High-level resistance: number analyzed (Participants) | 2
  INI, NRTI, ddI, High-level resistance | 0
  INI, PI, ATV/r, Susceptible: number analyzed (Participants) | 2
  INI, PI, ATV/r, Susceptible | 2
  INI, PI, ATV/r, Potential low-level resistance: number analyzed (Participants) | 2
  INI, PI, ATV/r, Potential low-level resistance | 0
  INI, PI, ATV/r, Low-level resistance: number analyzed (Participants) | 2
  INI, PI, ATV/r, Low-level resistance | 0
  INI, PI, ATV/r, Intermediate resistance: number analyzed (Participants) | 2
  INI, PI, ATV/r, Intermediate resistance | 0
  INI, PI, ATV/r, High-level resistance: number analyzed (Participants) | 2
  INI, PI, ATV/r, High-level resistance | 0
  INI, PI, DRV/r, Susceptible: number analyzed (Participants) | 2
  INI, PI, DRV/r, Susceptible | 2
  INI, PI, DRV/r, Potential low-level resistance: number analyzed (Participants) | 2
  INI, PI, DRV/r, Potential low-level resistance | 0
  INI, PI, DRV/r, Low-level resistance: number analyzed (Participants) | 2
  INI, PI, DRV/r, Low-level resistance | 0
  INI, PI, DRV/r, Intermediate resistance: number analyzed (Participants) | 2
  INI, PI, DRV/r, Intermediate resistance | 0
  INI, PI, DRV/r, High-level resistance: number analyzed (Participants) | 2
  INI, PI, DRV/r, High-level resistance | 0
  INI, PI, FPV/r, Susceptible: number analyzed (Participants) | 2
  INI, PI, FPV/r, Susceptible | 2
  INI, PI, FPV/r, Potential low-level resistance: number analyzed (Participants) | 2
  INI, PI, FPV/r, Potential low-level resistance | 0
  INI, PI, FPV/r, Low-level resistance: number analyzed (Participants) | 2
  INI, PI, FPV/r, Low-level resistance | 0
  INI, PI, FPV/r, Intermediate resistance: number analyzed (Participants) | 2
  INI, PI, FPV/r, Intermediate resistance | 0
  INI, PI, FPV/r, High-level resistance: number analyzed (Participants) | 2
  INI, PI, FPV/r, High-level resistance | 0
  INI, PI, IDV/r, Susceptible: number analyzed (Participants) | 2
  INI, PI, IDV/r, Susceptible | 2
  INI, PI, IDV/r, Potential low-level resistance: number analyzed (Participants) | 2
  INI, PI, IDV/r, Potential low-level resistance | 0
  INI, PI, IDV/r, Low-level resistance: number analyzed (Participants) | 2
  INI, PI, IDV/r, Low-level resistance | 0
  INI, PI, IDV/r, Intermediate resistance: number analyzed (Participants) | 2
  INI, PI, IDV/r, Intermediate resistance | 0
  INI, PI, IDV/r, High-level resistance: number analyzed (Participants) | 2
  INI, PI, IDV/r, High-level resistance | 0
  INI, PI, LPV/r, Susceptible: number analyzed (Participants) | 2
  INI, PI, LPV/r, Susceptible | 2
  INI, PI, LPV/r, Potential low-level resistance: number analyzed (Participants) | 2
  INI, PI, LPV/r, Potential low-level resistance | 0
  INI, PI, LPV/r, Low-level resistance: number analyzed (Participants) | 2
  INI, PI, LPV/r, Low-level resistance | 0
  INI, PI, LPV/r, Intermediate resistance: number analyzed (Participants) | 2
  INI, PI, LPV/r, Intermediate resistance | 0
  INI, PI, LPV/r, High-level resistance: number analyzed (Participants) | 2
  INI, PI, LPV/r, High-level resistance | 0
  INI, PI, NFV, Susceptible: number analyzed (Participants) | 2
  INI, PI, NFV, Susceptible | 2
  INI, PI, NFV, Potential low-level resistance: number analyzed (Participants) | 2
  INI, PI, NFV, Potential low-level resistance | 0
  INI, PI, NFV, Low-level resistance: number analyzed (Participants) | 2
  INI, PI, NFV, Low-level resistance | 0
  INI, PI, NFV, Intermediate resistance: number analyzed (Participants) | 2
  INI, PI, NFV, Intermediate resistance | 0
  INI, PI, NFV, High-level resistance: number analyzed (Participants) | 2
  INI, PI, NFV, High-level resistance | 0
  INI, PI, RTV, Susceptible: number analyzed (Participants) | 2
  INI, PI, RTV, Susceptible | 2
  INI, PI, RTV, Potential low-level resistance: number analyzed (Participants) | 2
  INI, PI, RTV, Potential low-level resistance | 0
  INI, PI, RTV, Low-level resistance: number analyzed (Participants) | 2
  INI, PI, RTV, Low-level resistance | 0
  INI, PI, RTV, Intermediate resistance: number analyzed (Participants) | 2
  INI, PI, RTV, Intermediate resistance | 0
  INI, PI, RTV, High-level resistance: number analyzed (Participants) | 2
  INI, PI, RTV, High-level resistance | 0
  INI, PI, SQV/r, Susceptible: number analyzed (Participants) | 2
  INI, PI, SQV/r, Susceptible | 2
  INI, PI, SQV/r, Potential low-level resistance: number analyzed (Participants) | 2
  INI, PI, SQV/r, Potential low-level resistance | 0
  INI, PI, SQV/r, Low-level resistance: number analyzed (Participants) | 2
  INI, PI, SQV/r, Low-level resistance | 0
  INI, PI, SQV/r, Intermediate resistance: number analyzed (Participants) | 2
  INI, PI, SQV/r, Intermediate resistance | 0
  INI, PI, SQV/r, High-level resistance: number analyzed (Participants) | 2
  INI, PI, SQV/r, High-level resistance | 0
  INI, PI, TPV/r, Susceptible: number analyzed (Participants) | 2
  INI, PI, TPV/r, Susceptible | 2
  INI, PI, TPV/r, Potential low-level resistance: number analyzed (Participants) | 2
  INI, PI, TPV/r, Potential low-level resistance | 0
  INI, PI, TPV/r, Low-level resistance: number analyzed (Participants) | 2
  INI, PI, TPV/r, Low-level resistance | 0
  INI, PI, TPV/r, Intermediate resistance: number analyzed (Participants) | 2
  INI, PI, TPV/r, Intermediate resistance | 0
  INI, PI, TPV/r, High-level resistance: number analyzed (Participants) | 2
  INI, PI, TPV/r, High-level resistance | 0
  PI, INI, DTG, Susceptible: number analyzed (Participants) | 1
  PI, INI, DTG, Susceptible | 1
  PI, INI, DTG, Potential low-level resistance: number analyzed (Participants) | 1
  PI, INI, DTG, Potential low-level resistance | 0
  PI, INI, DTG, Low-level resistance: number analyzed (Participants) | 1
  PI, INI, DTG, Low-level resistance | 0
  PI, INI, DTG, Intermediate resistance: number analyzed (Participants) | 1
  PI, INI, DTG, Intermediate resistance | 0
  PI, INI, DTG, High-level resistance: number analyzed (Participants) | 1
  PI, INI, DTG, High-level resistance | 0
  PI, INI, EVG, Susceptible: number analyzed (Participants) | 1
  PI, INI, EVG, Susceptible | 1
  PI, INI, EVG, Potential low-level resistance: number analyzed (Participants) | 1
  PI, INI, EVG, Potential low-level resistance | 0
  PI, INI, EVG, Low-level resistance: number analyzed (Participants) | 1
  PI, INI, EVG, Low-level resistance | 0
  PI, INI, EVG, Intermediate resistance: number analyzed (Participants) | 1
  PI, INI, EVG, Intermediate resistance | 0
  PI, INI, EVG, High-level resistance: number analyzed (Participants) | 1
  PI, INI, EVG, High-level resistance | 0
  PI, INI, RAL, Susceptible: number analyzed (Participants) | 1
  PI, INI, RAL, Susceptible | 1
  PI, INI, RAL, Potential low-level resistance: number analyzed (Participants) | 1
  PI, INI, RAL, Potential low-level resistance | 0
  PI, INI, RAL, Low-level resistance: number analyzed (Participants) | 1
  PI, INI, RAL, Low-level resistance | 0
  PI, INI, RAL, Intermediate resistance: number analyzed (Participants) | 1
  PI, INI, RAL, Intermediate resistance | 0
  PI, INI, RAL, High-level resistance: number analyzed (Participants) | 1
  PI, INI, RAL, High-level resistance | 0
  PI, NNRTI, DLV, Susceptible: number analyzed (Participants) | 1
  PI, NNRTI, DLV, Susceptible | 1
  PI, NNRTI, DLV, Potential low-level resistance: number analyzed (Participants) | 1
  PI, NNRTI, DLV, Potential low-level resistance | 0
  PI, NNRTI, DLV, Low-level resistance: number analyzed (Participants) | 1
  PI, NNRTI, DLV, Low-level resistance | 0
  PI, NNRTI, DLV, Intermediate resistance: number analyzed (Participants) | 1
  PI, NNRTI, DLV, Intermediate resistance | 0
  PI, NNRTI, DLV, High-level resistance: number analyzed (Participants) | 1
  PI, NNRTI, DLV, High-level resistance | 0
  PI, NNRTI, EFV, Susceptible: number analyzed (Participants) | 1
  PI, NNRTI, EFV, Susceptible | 1
  PI, NNRTI, EFV, Potential low-level resistance: number analyzed (Participants) | 1
  PI, NNRTI, EFV, Potential low-level resistance | 0
  PI, NNRTI, EFV, Low-level resistance: number analyzed (Participants) | 1
  PI, NNRTI, EFV, Low-level resistance | 0
  PI, NNRTI, EFV, Intermediate resistance: number analyzed (Participants) | 1
  PI, NNRTI, EFV, Intermediate resistance | 0
  PI, NNRTI, EFV, High-level resistance: number analyzed (Participants) | 1
  PI, NNRTI, EFV, High-level resistance | 0
  PI, NNRTI, ETR, Susceptible: number analyzed (Participants) | 1
  PI, NNRTI, ETR, Susceptible | 1
  PI, NNRTI, ETR, Potential low-level resistance: number analyzed (Participants) | 1
  PI, NNRTI, ETR, Potential low-level resistance | 0
  PI, NNRTI, ETR, Low-level resistance: number analyzed (Participants) | 1
  PI, NNRTI, ETR, Low-level resistance | 0
  PI, NNRTI, ETR, Intermediate resistance: number analyzed (Participants) | 1
  PI, NNRTI, ETR, Intermediate resistance | 0
  PI, NNRTI, ETR, High-level resistance: number analyzed (Participants) | 1
  PI, NNRTI, ETR, High-level resistance | 0
  PI, NNRTI, NVP, Susceptible: number analyzed (Participants) | 1
  PI, NNRTI, NVP, Susceptible | 1
  PI, NNRTI, NVP, Potential low-level resistance: number analyzed (Participants) | 1
  PI, NNRTI, NVP, Potential low-level resistance | 0
  PI, NNRTI, NVP, Low-level resistance: number analyzed (Participants) | 1
  PI, NNRTI, NVP, Low-level resistance | 0
  PI, NNRTI, NVP, Intermediate resistance: number analyzed (Participants) | 1
  PI, NNRTI, NVP, Intermediate resistance | 0
  PI, NNRTI, NVP, High-level resistance: number analyzed (Participants) | 1
  PI, NNRTI, NVP, High-level resistance | 0
  PI, NNRTI, RPV, Susceptible: number analyzed (Participants) | 1
  PI, NNRTI, RPV, Susceptible | 1
  PI, NNRTI, RPV, Potential low-level resistance: number analyzed (Participants) | 1
  PI, NNRTI, RPV, Potential low-level resistance | 0
  PI, NNRTI, RPV, Low-level resistance: number analyzed (Participants) | 1
  PI, NNRTI, RPV, Low-level resistance | 0
  PI, NNRTI, RPV, Intermediate resistance: number analyzed (Participants) | 1
  PI, NNRTI, RPV, Intermediate resistance | 0
  PI, NNRTI, RPV, High-level resistance: number analyzed (Participants) | 1
  PI, NNRTI, RPV, High-level resistance | 0
  PI, NRTI, 3TC, Susceptible: number analyzed (Participants) | 1
  PI, NRTI, 3TC, Susceptible | 1
  PI, NRTI, 3TC, Potential low-level resistance: number analyzed (Participants) | 1
  PI, NRTI, 3TC, Potential low-level resistance | 0
  PI, NRTI, 3TC, Low-level resistance: number analyzed (Participants) | 1
  PI, NRTI, 3TC, Low-level resistance | 0
  PI, NRTI, 3TC, Intermediate resistance: number analyzed (Participants) | 1
  PI, NRTI, 3TC, Intermediate resistance | 0
  PI, NRTI, 3TC, High-level resistance: number analyzed (Participants) | 1
  PI, NRTI, 3TC, High-level resistance | 0
  PI, NRTI, ABC, Susceptible: number analyzed (Participants) | 1
  PI, NRTI, ABC, Susceptible | 1
  PI, NRTI, ABC, Potential low-level resistance: number analyzed (Participants) | 1
  PI, NRTI, ABC, Potential low-level resistance | 0
  PI, NRTI, ABC, Low-level resistance: number analyzed (Participants) | 1
  PI, NRTI, ABC, Low-level resistance | 0
  PI, NRTI, ABC, Intermediate resistance: number analyzed (Participants) | 1
  PI, NRTI, ABC, Intermediate resistance | 0
  PI, NRTI, ABC, High-level resistance: number analyzed (Participants) | 1
  PI, NRTI, ABC, High-level resistance | 0
  PI, NRTI, FTC, Susceptible: number analyzed (Participants) | 1
  PI, NRTI, FTC, Susceptible | 1
  PI, NRTI, FTC, Potential low-level resistance: number analyzed (Participants) | 1
  PI, NRTI, FTC, Potential low-level resistance | 0
  PI, NRTI, FTC, Low-level resistance: number analyzed (Participants) | 1
  PI, NRTI, FTC, Low-level resistance | 0
  PI, NRTI, FTC, Intermediate resistance: number analyzed (Participants) | 1
  PI, NRTI, FTC, Intermediate resistance | 0
  PI, NRTI, FTC, High-level resistance: number analyzed (Participants) | 1
  PI, NRTI, FTC, High-level resistance | 0
  PI, NRTI, TDF, Susceptible: number analyzed (Participants) | 1
  PI, NRTI, TDF, Susceptible | 1
  PI, NRTI, TDF, Potential low-level resistance: number analyzed (Participants) | 1
  PI, NRTI, TDF, Potential low-level resistance | 0
  PI, NRTI, TDF, Low-level resistance: number analyzed (Participants) | 1
  PI, NRTI, TDF, Low-level resistance | 0
  PI, NRTI, TDF, Intermediate resistance: number analyzed (Participants) | 1
  PI, NRTI, TDF, Intermediate resistance | 0
  PI, NRTI, TDF, High-level resistance: number analyzed (Participants) | 1
  PI, NRTI, TDF, High-level resistance | 0
  PI, NRTI, ZDV, Susceptible: number analyzed (Participants) | 1
  PI, NRTI, ZDV, Susceptible | 1
  PI, NRTI, ZDV, Potential low-level resistance: number analyzed (Participants) | 1
  PI, NRTI, ZDV, Potential low-level resistance | 0
  PI, NRTI, ZDV, Low-level resistance: number analyzed (Participants) | 1
  PI, NRTI, ZDV, Low-level resistance | 0
  PI, NRTI, ZDV, Intermediate resistance: number analyzed (Participants) | 1
  PI, NRTI, ZDV, Intermediate resistance | 0
  PI, NRTI, ZDV, High-level resistance: number analyzed (Participants) | 1
  PI, NRTI, ZDV, High-level resistance | 0
  PI, NRTI, d4T, Susceptible: number analyzed (Participants) | 1
  PI, NRTI, d4T, Susceptible | 1
  PI, NRTI, d4T, Potential low-level resistance: number analyzed (Participants) | 1
  PI, NRTI, d4T, Potential low-level resistance | 0
  PI, NRTI, d4T, Low-level resistance: number analyzed (Participants) | 1
  PI, NRTI, d4T, Low-level resistance | 0
  PI, NRTI, d4T, Intermediate resistance: number analyzed (Participants) | 1
  PI, NRTI, d4T, Intermediate resistance | 0
  PI, NRTI, d4T, High-level resistance: number analyzed (Participants) | 1
  PI, NRTI, d4T, High-level resistance | 0
  PI, NRTI, ddI, Susceptible: number analyzed (Participants) | 1
  PI, NRTI, ddI, Susceptible | 1
  PI, NRTI, ddI, Potential low-level resistance: number analyzed (Participants) | 1
  PI, NRTI, ddI, Potential low-level resistance | 0
  PI, NRTI, ddI, Low-level resistance: number analyzed (Participants) | 1
  PI, NRTI, ddI, Low-level resistance | 0
  PI, NRTI, ddI, Intermediate resistance: number analyzed (Participants) | 1
  PI, NRTI, ddI, Intermediate resistance | 0
  PI, NRTI, ddI, High-level resistance: number analyzed (Participants) | 1
  PI, NRTI, ddI, High-level resistance | 0
  PI, PI, ATV/r, Susceptible: number analyzed (Participants) | 1
  PI, PI, ATV/r, Susceptible | 1
  PI, PI, ATV/r, Potential low-level resistance: number analyzed (Participants) | 1
  PI, PI, ATV/r, Potential low-level resistance | 0
  PI, PI, ATV/r, Low-level resistance: number analyzed (Participants) | 1
  PI, PI, ATV/r, Low-level resistance | 0
  PI, PI, ATV/r, Intermediate resistance: number analyzed (Participants) | 1
  PI, PI, ATV/r, Intermediate resistance | 0
  PI, PI, ATV/r, High-level resistance: number analyzed (Participants) | 1
  PI, PI, ATV/r, High-level resistance | 0
  PI, PI, DRV/r, Susceptible: number analyzed (Participants) | 1
  PI, PI, DRV/r, Susceptible | 1
  PI, PI, DRV/r, Potential low-level resistance: number analyzed (Participants) | 1
  PI, PI, DRV/r, Potential low-level resistance | 0
  PI, PI, DRV/r, Low-level resistance: number analyzed (Participants) | 1
  PI, PI, DRV/r, Low-level resistance | 0
  PI, PI, DRV/r, Intermediate resistance: number analyzed (Participants) | 1
  PI, PI, DRV/r, Intermediate resistance | 0
  PI, PI, DRV/r, High-level resistance: number analyzed (Participants) | 1
  PI, PI, DRV/r, High-level resistance | 0
  PI, PI, FPV/r, Susceptible: number analyzed (Participants) | 1
  PI, PI, FPV/r, Susceptible | 1
  PI, PI, FPV/r, Potential low-level resistance: number analyzed (Participants) | 1
  PI, PI, FPV/r, Potential low-level resistance | 0
  PI, PI, FPV/r, Low-level resistance: number analyzed (Participants) | 1
  PI, PI, FPV/r, Low-level resistance | 0
  PI, PI, FPV/r, Intermediate resistance: number analyzed (Participants) | 1
  PI, PI, FPV/r, Intermediate resistance | 0
  PI, PI, FPV/r, High-level resistance: number analyzed (Participants) | 1
  PI, PI, FPV/r, High-level resistance | 0
  PI, PI, IDV/r, Susceptible: number analyzed (Participants) | 1
  PI, PI, IDV/r, Susceptible | 1
  PI, PI, IDV/r, Potential low-level resistance: number analyzed (Participants) | 1
  PI, PI, IDV/r, Potential low-level resistance | 0
  PI, PI, IDV/r, Low-level resistance: number analyzed (Participants) | 1
  PI, PI, IDV/r, Low-level resistance | 0
  PI, PI, IDV/r, Intermediate resistance: number analyzed (Participants) | 1
  PI, PI, IDV/r, Intermediate resistance | 0
  PI, PI, IDV/r, High-level resistance: number analyzed (Participants) | 1
  PI, PI, IDV/r, High-level resistance | 0
  PI, PI, LPV/r, Susceptible: number analyzed (Participants) | 1
  PI, PI, LPV/r, Susceptible | 1
  PI, PI, LPV/r, Potential low-level resistance: number analyzed (Participants) | 1
  PI, PI, LPV/r, Potential low-level resistance | 0
  PI, PI, LPV/r, Low-level resistance: number analyzed (Participants) | 1
  PI, PI, LPV/r, Low-level resistance | 0
  PI, PI, LPV/r, Intermediate resistance: number analyzed (Participants) | 1
  PI, PI, LPV/r, Intermediate resistance | 0
  PI, PI, LPV/r, High-level resistance: number analyzed (Participants) | 1
  PI, PI, LPV/r, High-level resistance | 0
  PI, PI, NFV, Susceptible: number analyzed (Participants) | 1
  PI, PI, NFV, Susceptible | 1
  PI, PI, NFV, Potential low-level resistance: number analyzed (Participants) | 1
  PI, PI, NFV, Potential low-level resistance | 0
  PI, PI, NFV, Low-level resistance: number analyzed (Participants) | 1
  PI, PI, NFV, Low-level resistance | 0
  PI, PI, NFV, Intermediate resistance: number analyzed (Participants) | 1
  PI, PI, NFV, Intermediate resistance | 0
  PI, PI, NFV, High-level resistance: number analyzed (Participants) | 1
  PI, PI, NFV, High-level resistance | 0
  PI, PI, RTV, Susceptible: number analyzed (Participants) | 1
  PI, PI, RTV, Susceptible | 1
  PI, PI, RTV, Potential low-level resistance: number analyzed (Participants) | 1
  PI, PI, RTV, Potential low-level resistance | 0
  PI, PI, RTV, Low-level resistance: number analyzed (Participants) | 1
  PI, PI, RTV, Low-level resistance | 0
  PI, PI, RTV, Intermediate resistance: number analyzed (Participants) | 1
  PI, PI, RTV, Intermediate resistance | 0
  PI, PI, RTV, High-level resistance: number analyzed (Participants) | 1
  PI, PI, RTV, High-level resistance | 0
  PI, PI, SQV/r, Susceptible: number analyzed (Participants) | 1
  PI, PI, SQV/r, Susceptible | 1
  PI, PI, SQV/r, Potential low-level resistance: number analyzed (Participants) | 1
  PI, PI, SQV/r, Potential low-level resistance | 0
  PI, PI, SQV/r, Low-level resistance: number analyzed (Participants) | 1
  PI, PI, SQV/r, Low-level resistance | 0
  PI, PI, SQV/r, Intermediate resistance: number analyzed (Participants) | 1
  PI, PI, SQV/r, Intermediate resistance | 0
  PI, PI, SQV/r, High-level resistance: number analyzed (Participants) | 1
  PI, PI, SQV/r, High-level resistance | 0
  PI, PI, TPV/r, Susceptible: number analyzed (Participants) | 1
  PI, PI, TPV/r, Susceptible | 1
  PI, PI, TPV/r, Potential low-level resistance: number analyzed (Participants) | 1
  PI, PI, TPV/r, Potential low-level resistance | 0
  PI, PI, TPV/r, Low-level resistance: number analyzed (Participants) | 1
  PI, PI, TPV/r, Low-level resistance | 0
  PI, PI, TPV/r, Intermediate resistance: number analyzed (Participants) | 1
  PI, PI, TPV/r, Intermediate resistance | 0
  PI, PI, TPV/r, High-level resistance: number analyzed (Participants) | 1
  PI, PI, TPV/r, High-level resistance | 0

48. Secondary Outcome: Number of Participants With Observed Phenotypic Resistance for Participants Meeting Virologic Withdrawal Criteria by Baseline Third Agent Treatment Class-DTG+RPV Group Through Continuation Phase
Description: For all participants who met virologic withdrawal criteria, plasma samples with HIV-1 RNA level >=200 c/mL were analyzed in an attempt to obtain phenotype data on as many samples as possible. Samples for drug resistance testing (phenotypic) were collected at Day 1. Number of participants with phenotypic resistance to DTG or RPV for those meeting virologic withdrawal criteria in subgroups, stratified based on baseline third agent treatment class (NNRTI, INI, PI) were summarized.
Time Frame: Up to Week 411
Population: The analysis was performed on the CVW Resistance population.
Measure: Count of Participants; unit: Participants
Arm/Group | DTG + RPV
Number analyzed (Participants) | 3
Participants
  NNRTI, INI, DTG, Resistant: number analyzed (Participants) | 2
  NNRTI, INI, DTG, Resistant | 0
  NNRTI, INI, DTG, Partially Sensitive: number analyzed (Participants) | 2
  NNRTI, INI, DTG, Partially Sensitive | 0
  NNRTI, INI, DTG, Sensitive: number analyzed (Participants) | 2
  NNRTI, INI, DTG, Sensitive | 2
  NNRTI, INI, EVG, Resistant: number analyzed (Participants) | 2
  NNRTI, INI, EVG, Resistant | 0
  NNRTI, INI, EVG, Partially Sensitive: number analyzed (Participants) | 2
  NNRTI, INI, EVG, Partially Sensitive | 0
  NNRTI, INI, EVG, Sensitive: number analyzed (Participants) | 2
  NNRTI, INI, EVG, Sensitive | 2
  NNRTI, INI, RAL, Resistant: number analyzed (Participants) | 2
  NNRTI, INI, RAL, Resistant | 0
  NNRTI, INI, RAL, Partially Sensitive: number analyzed (Participants) | 2
  NNRTI, INI, RAL, Partially Sensitive | 0
  NNRTI, INI, RAL, Sensitive: number analyzed (Participants) | 2
  NNRTI, INI, RAL, Sensitive | 2
  NNRTI, NNRTI, DLV, Resistant | 1
  NNRTI, NNRTI, DLV, Partially Sensitive | 0
  NNRTI, NNRTI, DLV, Sensitive | 2
  NNRTI, NNRTI, EFV, Resistant | 1
  NNRTI, NNRTI, EFV, Partially Sensitive | 0
  NNRTI, NNRTI, EFV, Sensitive | 2
  NNRTI, NNRTI, ETR, Resistant | 0
  NNRTI, NNRTI, ETR, Partially Sensitive | 1
  NNRTI, NNRTI, ETR, Sensitive | 2
  NNRTI, NNRTI, NVP, Resistant | 1
  NNRTI, NNRTI, NVP, Partially Sensitive | 0
  NNRTI, NNRTI, NVP, Sensitive | 2
  NNRTI, NNRTI, RPV, Resistant | 1
  NNRTI, NNRTI, RPV, Partially Sensitive | 0
  NNRTI, NNRTI, RPV, Sensitive | 2
  NNRTI, NRTI, 3TC, Resistant | 0
  NNRTI, NRTI, 3TC, Partially Sensitive | 0
  NNRTI, NRTI, 3TC, Sensitive | 3
  NNRTI, NRTI, ABC, Resistant | 0
  NNRTI, NRTI, ABC, Partially Sensitive | 0
  NNRTI, NRTI, ABC, Sensitive | 3
  NNRTI, NRTI, FTC, Resistant | 0
  NNRTI, NRTI, FTC, Partially Sensitive | 0
  NNRTI, NRTI, FTC, Sensitive | 3
  NNRTI, NRTI, TDF, Resistant | 0
  NNRTI, NRTI, TDF, Partially Sensitive | 0
  NNRTI, NRTI, TDF, Sensitive | 3
  NNRTI, NRTI, ZDV, Resistant | 0
  NNRTI, NRTI, ZDV, Partially Sensitive | 0
  NNRTI, NRTI, ZDV, Sensitive | 3
  NNRTI, NRTI, d4T, Resistant | 0
  NNRTI, NRTI, d4T, Partially Sensitive | 0
  NNRTI, NRTI, d4T, Sensitive | 3
  NNRTI, NRTI, ddI, Resistant | 0
  NNRTI, NRTI, ddI, Partially Sensitive | 0
  NNRTI, NRTI, ddI, Sensitive | 3
  NNRTI, PI, ATV/r, Resistant | 0
  NNRTI, PI, ATV/r, Partially Sensitive | 0
  NNRTI, PI, ATV/r, Sensitive | 3
  NNRTI, PI, DRV/r, Resistant | 0
  NNRTI, PI, DRV/r, Partially Sensitive | 0
  NNRTI, PI, DRV/r, Sensitive | 3
  NNRTI, PI, FPV/r, Resistant | 0
  NNRTI, PI, FPV/r, Partially Sensitive | 0
  NNRTI, PI, FPV/r, Sensitive | 3
  NNRTI, PI, IDV/r, Resistant | 0
  NNRTI, PI, IDV/r, Partially Sensitive | 0
  NNRTI, PI, IDV/r, Sensitive | 3
  NNRTI, PI, LPV/r, Resistant | 0
  NNRTI, PI, LPV/r, Partially Sensitive | 0
  NNRTI, PI, LPV/r, Sensitive | 3
  NNRTI, PI, NFV, Resistant | 0
  NNRTI, PI, NFV, Partially Sensitive | 0
  NNRTI, PI, NFV, Sensitive | 3
  NNRTI, PI, RTV, Resistant | 0
  NNRTI, PI, RTV, Partially Sensitive | 0
  NNRTI, PI, RTV, Sensitive | 3
  NNRTI, PI, SQV/r, Resistant | 0
  NNRTI, PI, SQV/r, Partially Sensitive | 0
  NNRTI, PI, SQV/r, Sensitive | 3
  NNRTI, PI, TPV/r, Resistant | 0
  NNRTI, PI, TPV/r, Partially Sensitive | 0
  NNRTI, PI, TPV/r, Sensitive | 3
  INI, INI, DTG, Resistant: number analyzed (Participants) | 2
  INI, INI, DTG, Resistant | 0
  INI, INI, DTG, Partially Sensitive: number analyzed (Participants) | 2
  INI, INI, DTG, Partially Sensitive | 0
  INI, INI, DTG, Sensitive: number analyzed (Participants) | 2
  INI, INI, DTG, Sensitive | 2
  INI, INI, EVG, Resistant: number analyzed (Participants) | 2
  INI, INI, EVG, Resistant | 0
  INI, INI, EVG, Partially Sensitive: number analyzed (Participants) | 2
  INI, INI, EVG, Partially Sensitive | 0
  INI, INI, EVG, Sensitive: number analyzed (Participants) | 2
  INI, INI, EVG, Sensitive | 2
  INI, INI, RAL, Resistant: number analyzed (Participants) | 2
  INI, INI, RAL, Resistant | 0
  INI, INI, RAL, Partially Sensitive: number analyzed (Participants) | 2
  INI, INI, RAL, Partially Sensitive | 0
  INI, INI, RAL, Sensitive: number analyzed (Participants) | 2
  INI, INI, RAL, Sensitive | 2
  INI, NNRTI, DLV, Resistant: number analyzed (Participants) | 2
  INI, NNRTI, DLV, Resistant | 0
  INI, NNRTI, DLV, Partially Sensitive: number analyzed (Participants) | 2
  INI, NNRTI, DLV, Partially Sensitive | 0
  INI, NNRTI, DLV, Sensitive: number analyzed (Participants) | 2
  INI, NNRTI, DLV, Sensitive | 2
  INI, NNRTI, EFV, Resistant: number analyzed (Participants) | 2
  INI, NNRTI, EFV, Resistant | 0
  INI, NNRTI, EFV, Partially Sensitive: number analyzed (Participants) | 2
  INI, NNRTI, EFV, Partially Sensitive | 0
  INI, NNRTI, EFV, Sensitive: number analyzed (Participants) | 2
  INI, NNRTI, EFV, Sensitive | 2
  INI, NNRTI, ETR, Resistant: number analyzed (Participants) | 2
  INI, NNRTI, ETR, Resistant | 0
  INI, NNRTI, ETR, Partially Sensitive: number analyzed (Participants) | 2
  INI, NNRTI, ETR, Partially Sensitive | 0
  INI, NNRTI, ETR, Sensitive: number analyzed (Participants) | 2
  INI, NNRTI, ETR, Sensitive | 2
  INI, NNRTI, NVP, Resistant: number analyzed (Participants) | 2
  INI, NNRTI, NVP, Resistant | 0
  INI, NNRTI, NVP, Partially Sensitive: number analyzed (Participants) | 2
  INI, NNRTI, NVP, Partially Sensitive | 0
  INI, NNRTI, NVP, Sensitive: number analyzed (Participants) | 2
  INI, NNRTI, NVP, Sensitive | 2
  INI, NNRTI, RPV, Resistant: number analyzed (Participants) | 2
  INI, NNRTI, RPV, Resistant | 0
  INI, NNRTI, RPV, Partially Sensitive: number analyzed (Participants) | 2
  INI, NNRTI, RPV, Partially Sensitive | 0
  INI, NNRTI, RPV, Sensitive: number analyzed (Participants) | 2
  INI, NNRTI, RPV, Sensitive | 2
  INI, NRTI, 3TC, Resistant: number analyzed (Participants) | 2
  INI, NRTI, 3TC, Resistant | 0
  INI, NRTI, 3TC, Partially Sensitive: number analyzed (Participants) | 2
  INI, NRTI, 3TC, Partially Sensitive | 0
  INI, NRTI, 3TC, Sensitive: number analyzed (Participants) | 2
  INI, NRTI, 3TC, Sensitive | 2
  INI, NRTI, ABC, Resistant: number analyzed (Participants) | 2
  INI, NRTI, ABC, Resistant | 0
  INI, NRTI, ABC, Partially Sensitive: number analyzed (Participants) | 2
  INI, NRTI, ABC, Partially Sensitive | 0
  INI, NRTI, ABC, Sensitive: number analyzed (Participants) | 2
  INI, NRTI, ABC, Sensitive | 2
  INI, NRTI, FTC, Resistant: number analyzed (Participants) | 2
  INI, NRTI, FTC, Resistant | 0
  INI, NRTI, FTC, Partially Sensitive: number analyzed (Participants) | 2
  INI, NRTI, FTC, Partially Sensitive | 0
  INI, NRTI, FTC, Sensitive: number analyzed (Participants) | 2
  INI, NRTI, FTC, Sensitive | 2
  INI, NRTI, TDF, Resistant: number analyzed (Participants) | 2
  INI, NRTI, TDF, Resistant | 0
  INI, NRTI, TDF, Partially Sensitive: number analyzed (Participants) | 2
  INI, NRTI, TDF, Partially Sensitive | 0
  INI, NRTI, TDF, Sensitive: number analyzed (Participants) | 2
  INI, NRTI, TDF, Sensitive | 2
  INI, NRTI, ZDV, Resistant: number analyzed (Participants) | 2
  INI, NRTI, ZDV, Resistant | 0
  INI, NRTI, ZDV, Partially Sensitive: number analyzed (Participants) | 2
  INI, NRTI, ZDV, Partially Sensitive | 0
  INI, NRTI, ZDV, Sensitive: number analyzed (Participants) | 2
  INI, NRTI, ZDV, Sensitive | 2
  INI, NRTI, d4T, Resistant: number analyzed (Participants) | 2
  INI, NRTI, d4T, Resistant | 0
  INI, NRTI, d4T, Partially Sensitive: number analyzed (Participants) | 2
  INI, NRTI, d4T, Partially Sensitive | 0
  INI, NRTI, d4T, Sensitive: number analyzed (Participants) | 2
  INI, NRTI, d4T, Sensitive | 2
  INI, NRTI, ddI, Resistant: number analyzed (Participants) | 2
  INI, NRTI, ddI, Resistant | 0
  INI, NRTI, ddI, Partially Sensitive: number analyzed (Participants) | 2
  INI, NRTI, ddI, Partially Sensitive | 0
  INI, NRTI, ddI, Sensitive: number analyzed (Participants) | 2
  INI, NRTI, ddI, Sensitive | 2
  INI, PI, ATV/r, Resistant: number analyzed (Participants) | 2
  INI, PI, ATV/r, Resistant | 0
  INI, PI, ATV/r, Partially Sensitive: number analyzed (Participants) | 2
  INI, PI, ATV/r, Partially Sensitive | 0
  INI, PI, ATV/r, Sensitive: number analyzed (Participants) | 2
  INI, PI, ATV/r, Sensitive | 2
  INI, PI, DRV/r, Resistant: number analyzed (Participants) | 2
  INI, PI, DRV/r, Resistant | 0
  INI, PI, DRV/r, Partially Sensitive: number analyzed (Participants) | 2
  INI, PI, DRV/r, Partially Sensitive | 0
  INI, PI, DRV/r, Sensitive: number analyzed (Participants) | 2
  INI, PI, DRV/r, Sensitive | 2
  INI, PI, FPV/r, Resistant: number analyzed (Participants) | 2
  INI, PI, FPV/r, Resistant | 0
  INI, PI, FPV/r, Partially Sensitive: number analyzed (Participants) | 2
  INI, PI, FPV/r, Partially Sensitive | 0
  INI, PI, FPV/r, Sensitive: number analyzed (Participants) | 2
  INI, PI, FPV/r, Sensitive | 2
  INI, PI, IDV/r, Resistant: number analyzed (Participants) | 2
  INI, PI, IDV/r, Resistant | 0
  INI, PI, IDV/r, Partially Sensitive: number analyzed (Participants) | 2
  INI, PI, IDV/r, Partially Sensitive | 0
  INI, PI, IDV/r, Sensitive: number analyzed (Participants) | 2
  INI, PI, IDV/r, Sensitive | 2
  INI, PI, LPV/r, Resistant: number analyzed (Participants) | 2
  INI, PI, LPV/r, Resistant | 0
  INI, PI, LPV/r, Partially Sensitive: number analyzed (Participants) | 2
  INI, PI, LPV/r, Partially Sensitive | 0
  INI, PI, LPV/r, Sensitive: number analyzed (Participants) | 2
  INI, PI, LPV/r, Sensitive | 2
  INI, PI, NFV, Resistant: number analyzed (Participants) | 2
  INI, PI, NFV, Resistant | 0
  INI, PI, NFV, Partially Sensitive: number analyzed (Participants) | 2
  INI, PI, NFV, Partially Sensitive | 0
  INI, PI, NFV, Sensitive: number analyzed (Participants) | 2
  INI, PI, NFV, Sensitive | 2
  INI, PI, RTV, Resistant: number analyzed (Participants) | 2
  INI, PI, RTV, Resistant | 0
  INI, PI, RTV, Partially Sensitive: number analyzed (Participants) | 2
  INI, PI, RTV, Partially Sensitive | 0
  INI, PI, RTV, Sensitive: number analyzed (Participants) | 2
  INI, PI, RTV, Sensitive | 2
  INI, PI, SQV/r, Resistant: number analyzed (Participants) | 2
  INI, PI, SQV/r, Resistant | 0
  INI, PI, SQV/r, Partially Sensitive: number analyzed (Participants) | 2
  INI, PI, SQV/r, Partially Sensitive | 0
  INI, PI, SQV/r, Sensitive: number analyzed (Participants) | 2
  INI, PI, SQV/r, Sensitive | 2
  INI, PI, TPV/r, Resistant: number analyzed (Participants) | 2
  INI, PI, TPV/r, Resistant | 0
  INI, PI, TPV/r, Partially Sensitive: number analyzed (Participants) | 2
  INI, PI, TPV/r, Partially Sensitive | 0
  INI, PI, TPV/r, Sensitive: number analyzed (Participants) | 2
  INI, PI, TPV/r, Sensitive | 2
  PI, INI, DTG, Resistant: number analyzed (Participants) | 1
  PI, INI, DTG, Resistant | 0
  PI, INI, DTG, Partially Sensitive: number analyzed (Participants) | 1
  PI, INI, DTG, Partially Sensitive | 0
  PI, INI, DTG, Sensitive: number analyzed (Participants) | 1
  PI, INI, DTG, Sensitive | 1
  PI, INI, EVG, Resistant: number analyzed (Participants) | 1
  PI, INI, EVG, Resistant | 0
  PI, INI, EVG, Partially Sensitive: number analyzed (Participants) | 1
  PI, INI, EVG, Partially Sensitive | 0
  PI, INI, EVG, Sensitive: number analyzed (Participants) | 1
  PI, INI, EVG, Sensitive | 1
  PI, INI, RAL, Resistant: number analyzed (Participants) | 1
  PI, INI, RAL, Resistant | 0
  PI, INI, RAL, Partially Sensitive: number analyzed (Participants) | 1
  PI, INI, RAL, Partially Sensitive | 0
  PI, INI, RAL, Sensitive: number analyzed (Participants) | 1
  PI, INI, RAL, Sensitive | 1
  PI, NNRTI, DLV, Resistant: number analyzed (Participants) | 1
  PI, NNRTI, DLV, Resistant | 0
  PI, NNRTI, DLV, Partially Sensitive: number analyzed (Participants) | 1
  PI, NNRTI, DLV, Partially Sensitive | 0
  PI, NNRTI, DLV, Sensitive: number analyzed (Participants) | 1
  PI, NNRTI, DLV, Sensitive | 1
  PI, NNRTI, EFV, Resistant: number analyzed (Participants) | 1
  PI, NNRTI, EFV, Resistant | 0
  PI, NNRTI, EFV, Partially Sensitive: number analyzed (Participants) | 1
  PI, NNRTI, EFV, Partially Sensitive | 0
  PI, NNRTI, EFV, Sensitive: number analyzed (Participants) | 1
  PI, NNRTI, EFV, Sensitive | 1
  PI, NNRTI, ETR, Resistant: number analyzed (Participants) | 1
  PI, NNRTI, ETR, Resistant | 0
  PI, NNRTI, ETR, Partially Sensitive: number analyzed (Participants) | 1
  PI, NNRTI, ETR, Partially Sensitive | 0
  PI, NNRTI, ETR, Sensitive: number analyzed (Participants) | 1
  PI, NNRTI, ETR, Sensitive | 1
  PI, NNRTI, NVP, Resistant: number analyzed (Participants) | 1
  PI, NNRTI, NVP, Resistant | 0
  PI, NNRTI, NVP, Partially Sensitive: number analyzed (Participants) | 1
  PI, NNRTI, NVP, Partially Sensitive | 0
  PI, NNRTI, NVP, Sensitive: number analyzed (Participants) | 1
  PI, NNRTI, NVP, Sensitive | 1
  PI, NNRTI, RPV, Resistant: number analyzed (Participants) | 1
  PI, NNRTI, RPV, Resistant | 0
  PI, NNRTI, RPV, Partially Sensitive: number analyzed (Participants) | 1
  PI, NNRTI, RPV, Partially Sensitive | 0
  PI, NNRTI, RPV, Sensitive: number analyzed (Participants) | 1
  PI, NNRTI, RPV, Sensitive | 1
  PI, NRTI, 3TC, Resistant: number analyzed (Participants) | 1
  PI, NRTI, 3TC, Resistant | 0
  PI, NRTI, 3TC, Partially Sensitive: number analyzed (Participants) | 1
  PI, NRTI, 3TC, Partially Sensitive | 0
  PI, NRTI, 3TC, Sensitive: number analyzed (Participants) | 1
  PI, NRTI, 3TC, Sensitive | 1
  PI, NRTI, ABC, Resistant: number analyzed (Participants) | 1
  PI, NRTI, ABC, Resistant | 0
  PI, NRTI, ABC, Partially Sensitive: number analyzed (Participants) | 1
  PI, NRTI, ABC, Partially Sensitive | 0
  PI, NRTI, ABC, Sensitive: number analyzed (Participants) | 1
  PI, NRTI, ABC, Sensitive | 1
  PI, NRTI, FTC, Resistant: number analyzed (Participants) | 1
  PI, NRTI, FTC, Resistant | 0
  PI, NRTI, FTC, Partially Sensitive: number analyzed (Participants) | 1
  PI, NRTI, FTC, Partially Sensitive | 0
  PI, NRTI, FTC, Sensitive: number analyzed (Participants) | 1
  PI, NRTI, FTC, Sensitive | 1
  PI, NRTI, TDF, Resistant: number analyzed (Participants) | 1
  PI, NRTI, TDF, Resistant | 0
  PI, NRTI, TDF, Partially Sensitive: number analyzed (Participants) | 1
  PI, NRTI, TDF, Partially Sensitive | 0
  PI, NRTI, TDF, Sensitive: number analyzed (Participants) | 1
  PI, NRTI, TDF, Sensitive | 1
  PI, NRTI, ZDV, Resistant: number analyzed (Participants) | 1
  PI, NRTI, ZDV, Resistant | 0
  PI, NRTI, ZDV, Partially Sensitive: number analyzed (Participants) | 1
  PI, NRTI, ZDV, Partially Sensitive | 0
  PI, NRTI, ZDV, Sensitive: number analyzed (Participants) | 1
  PI, NRTI, ZDV, Sensitive | 1
  PI, NRTI, d4T, Resistant: number analyzed (Participants) | 1
  PI, NRTI, d4T, Resistant | 0
  PI, NRTI, d4T, Partially Sensitive: number analyzed (Participants) | 1
  PI, NRTI, d4T, Partially Sensitive | 0
  PI, NRTI, d4T, Sensitive: number analyzed (Participants) | 1
  PI, NRTI, d4T, Sensitive | 1
  PI, NRTI, ddI, Resistant: number analyzed (Participants) | 1
  PI, NRTI, ddI, Resistant | 0
  PI, NRTI, ddI, Partially Sensitive: number analyzed (Participants) | 1
  PI, NRTI, ddI, Partially Sensitive | 0
  PI, NRTI, ddI, Sensitive: number analyzed (Participants) | 1
  PI, NRTI, ddI, Sensitive | 1
  PI, PI, ATV/r, Resistant: number analyzed (Participants) | 1
  PI, PI, ATV/r, Resistant | 0
  PI, PI, ATV/r, Partially Sensitive: number analyzed (Participants) | 1
  PI, PI, ATV/r, Partially Sensitive | 0
  PI, PI, ATV/r, Sensitive: number analyzed (Participants) | 1
  PI, PI, ATV/r, Sensitive | 1
  PI, PI, DRV/r, Resistant: number analyzed (Participants) | 1
  PI, PI, DRV/r, Resistant | 0
  PI, PI, DRV/r, Partially Sensitive: number analyzed (Participants) | 1
  PI, PI, DRV/r, Partially Sensitive | 0
  PI, PI, DRV/r, Sensitive: number analyzed (Participants) | 1
  PI, PI, DRV/r, Sensitive | 1
  PI, PI, FPV/r, Resistant: number analyzed (Participants) | 1
  PI, PI, FPV/r, Resistant | 0
  PI, PI, FPV/r, Partially Sensitive: number analyzed (Participants) | 1
  PI, PI, FPV/r, Partially Sensitive | 0
  PI, PI, FPV/r, Sensitive: number analyzed (Participants) | 1
  PI, PI, FPV/r, Sensitive | 1
  PI, PI, IDV/r, Resistant: number analyzed (Participants) | 1
  PI, PI, IDV/r, Resistant | 0
  PI, PI, IDV/r, Partially Sensitive: number analyzed (Participants) | 1
  PI, PI, IDV/r, Partially Sensitive | 0
  PI, PI, IDV/r, Sensitive: number analyzed (Participants) | 1
  PI, PI, IDV/r, Sensitive | 1
  PI, PI, LPV/r, Resistant: number analyzed (Participants) | 1
  PI, PI, LPV/r, Resistant | 0
  PI, PI, LPV/r, Partially Sensitive: number analyzed (Participants) | 1
  PI, PI, LPV/r, Partially Sensitive | 0
  PI, PI, LPV/r, Sensitive: number analyzed (Participants) | 1
  PI, PI, LPV/r, Sensitive | 1
  PI, PI, NFV, Resistant: number analyzed (Participants) | 1
  PI, PI, NFV, Resistant | 0
  PI, PI, NFV, Partially Sensitive: number analyzed (Participants) | 1
  PI, PI, NFV, Partially Sensitive | 0
  PI, PI, NFV, Sensitive: number analyzed (Participants) | 1
  PI, PI, NFV, Sensitive | 1
  PI, PI, RTV, Resistant: number analyzed (Participants) | 1
  PI, PI, RTV, Resistant | 0
  PI, PI, RTV, Partially Sensitive: number analyzed (Participants) | 1
  PI, PI, RTV, Partially Sensitive | 0
  PI, PI, RTV, Sensitive: number analyzed (Participants) | 1
  PI, PI, RTV, Sensitive | 1
  PI, PI, SQV/r, Resistant: number analyzed (Participants) | 1
  PI, PI, SQV/r, Resistant | 0
  PI, PI, SQV/r, Partially Sensitive: number analyzed (Participants) | 1
  PI, PI, SQV/r, Partially Sensitive | 0
  PI, PI, SQV/r, Sensitive: number analyzed (Participants) | 1
  PI, PI, SQV/r, Sensitive | 1
  PI, PI, TPV/r, Resistant: number analyzed (Participants) | 1
  PI, PI, TPV/r, Resistant | 0
  PI, PI, TPV/r, Partially Sensitive: number analyzed (Participants) | 1
  PI, PI, TPV/r, Partially Sensitive | 0
  PI, PI, TPV/r, Sensitive: number analyzed (Participants) | 1
  PI, PI, TPV/r, Sensitive | 1

49. Secondary Outcome: Number of Participants With Observed Genotypic Resistance for Participants Meeting Virologic Withdrawal Criteria by Baseline Third Agent Treatment Class- CAR Group Through Continuation Phase
Description: For all participants who meet virologic withdrawal criteria, plasma samples with HIV-1 RNA level >=200 c/mL were analyzed in an attempt to obtain genotype data on as many samples as possible. Number of participants with genotypic resistance to CAR for those meeting virologic withdrawal criteria in subgroups, stratified based on baseline third agent treatment class (INI) were summarized.
Time Frame: Week 52 to Week 411
Population: The analysis was to be performed on the Late Switch CVW Resistance population.
Measure: Count of Participants; unit: Participants
Arm/Group | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 1
Participants
  INI, INI, DTG, Susceptible | 1
  INI, INI, DTG, Potential low-level resistance | 0
  INI, INI, DTG, Low-level resistance | 0
  INI, INI, DTG, Intermediate resistance | 0
  INI, INI, DTG, High-level resistance | 0
  INI, INI, EVG, Susceptible | 1
  INI, INI, EVG, Potential low-level resistance | 0
  INI, INI, EVG, Low-level resistance | 0
  INI, INI, EVG, Intermediate resistance | 0
  INI, INI, EVG, High-level resistance | 0
  INI, INI, RAL, Susceptible | 1
  INI, INI, RAL, Potential low-level resistance | 0
  INI, INI, RAL, Low-level resistance | 0
  INI, INI, RAL, Intermediate resistance | 0
  INI, INI, RAL, High-level resistance | 0
  INI, NNRTI, DLV, Susceptible | 1
  INI, NNRTI, DLV, Potential low-level resistance | 0
  INI, NNRTI, DLV, Low-level resistance | 0
  INI, NNRTI, DLV, Intermediate resistance | 0
  INI, NNRTI, DLV, High-level resistance | 0
  INI, NNRTI, EFV, Susceptible | 0
  INI, NNRTI, EFV, Potential low-level resistance | 1
  INI, NNRTI, EFV, Low-level resistance | 0
  INI, NNRTI, EFV, Intermediate resistance | 0
  INI, NNRTI, EFV, High-level resistance | 0
  INI, NNRTI, ETR, Susceptible | 0
  INI, NNRTI, ETR, Potential low-level resistance | 1
  INI, NNRTI, ETR, Low-level resistance | 0
  INI, NNRTI, ETR, Intermediate resistance | 0
  INI, NNRTI, ETR, High-level resistance | 0
  INI, NNRTI, NVP, Susceptible | 0
  INI, NNRTI, NVP, Potential low-level resistance | 1
  INI, NNRTI, NVP, Low-level resistance | 0
  INI, NNRTI, NVP, Intermediate resistance | 0
  INI, NNRTI, NVP, High-level resistance | 0
  INI, NNRTI, RPV, Susceptible | 0
  INI, NNRTI, RPV, Potential low-level resistance | 1
  INI, NNRTI, RPV, Low-level resistance | 0
  INI, NNRTI, RPV, Intermediate resistance | 0
  INI, NNRTI, RPV, High-level resistance | 0
  INI, NRTI, 3TC, Susceptible | 1
  INI, NRTI, 3TC, Potential low-level resistance | 0
  INI, NRTI, 3TC, Low-level resistance | 0
  INI, NRTI, 3TC, Intermediate resistance | 0
  INI, NRTI, 3TC, High-level resistance | 0
  INI, NRTI, ABC, Susceptible | 1
  INI, NRTI, ABC, Potential low-level resistance | 0
  INI, NRTI, ABC, Low-level resistance | 0
  INI, NRTI, ABC, Intermediate resistance | 0
  INI, NRTI, ABC, High-level resistance | 0
  INI, NRTI, FTC, Susceptible | 1
  INI, NRTI, FTC, Potential low-level resistance | 0
  INI, NRTI, FTC, Low-level resistance | 0
  INI, NRTI, FTC, Intermediate resistance | 0
  INI, NRTI, FTC, High-level resistance | 0
  INI, NRTI, TDF, Susceptible | 1
  INI, NRTI, TDF, Potential low-level resistance | 0
  INI, NRTI, TDF, Low-level resistance | 0
  INI, NRTI, TDF, Intermediate resistance | 0
  INI, NRTI, TDF, High-level resistance | 0
  INI, NRTI, ZDV, Susceptible | 1
  INI, NRTI, ZDV, Potential low-level resistance | 0
  INI, NRTI, ZDV, Low-level resistance | 0
  INI, NRTI, ZDV, Intermediate resistance | 0
  INI, NRTI, ZDV, High-level resistance | 0
  INI, NRTI, d4T, Susceptible | 1
  INI, NRTI, d4T, Potential low-level resistance | 0
  INI, NRTI, d4T, Low-level resistance | 0
  INI, NRTI, d4T, Intermediate resistance | 0
  INI, NRTI, d4T, High-level resistance | 0
  INI, NRTI, ddI, Susceptible | 1
  INI, NRTI, ddI, Potential low-level resistance | 0
  INI, NRTI, ddI, Low-level resistance | 0
  INI, NRTI, ddI, Intermediate resistance | 0
  INI, NRTI, ddI, High-level resistance | 0
  INI, PI, ATV/r, Susceptible | 1
  INI, PI, ATV/r, Potential low-level resistance | 0
  INI, PI, ATV/r, Low-level resistance | 0
  INI, PI, ATV/r, Intermediate resistance | 0
  INI, PI, ATV/r, High-level resistance | 0
  INI, PI, DRV/r, Susceptible | 1
  INI, PI, DRV/r, Potential low-level resistance | 0
  INI, PI, DRV/r, Low-level resistance | 0
  INI, PI, DRV/r, Intermediate resistance | 0
  INI, PI, DRV/r, High-level resistance | 0
  INI, PI, FPV/r, Susceptible | 1
  INI, PI, FPV/r, Potential low-level resistance | 0
  INI, PI, FPV/r, Low-level resistance | 0
  INI, PI, FPV/r, Intermediate resistance | 0
  INI, PI, FPV/r, High-level resistance | 0
  INI, PI, IDV/r, Susceptible | 1
  INI, PI, IDV/r, Potential low-level resistance | 0
  INI, PI, IDV/r, Low-level resistance | 0
  INI, PI, IDV/r, Intermediate resistance | 0
  INI, PI, IDV/r, High-level resistance | 0
  INI, PI, LPV/r, Susceptible | 1
  INI, PI, LPV/r, Potential low-level resistance | 0
  INI, PI, LPV/r, Low-level resistance | 0
  INI, PI, LPV/r, Intermediate resistance | 0
  INI, PI, LPV/r, High-level resistance | 0
  INI, PI, NFV, Susceptible | 1
  INI, PI, NFV, Potential low-level resistance | 0
  INI, PI, NFV, Low-level resistance | 0
  INI, PI, NFV, Intermediate resistance | 0
  INI, PI, NFV, High-level resistance | 0
  INI, PI, RTV, Susceptible | 1
  INI, PI, RTV, Potential low-level resistance | 0
  INI, PI, RTV, Low-level resistance | 0
  INI, PI, RTV, Intermediate resistance | 0
  INI, PI, RTV, High-level resistance | 0
  INI, PI, SQV/r, Susceptible | 1
  INI, PI, SQV/r, Potential low-level resistance | 0
  INI, PI, SQV/r, Low-level resistance | 0
  INI, PI, SQV/r, Intermediate resistance | 0
  INI, PI, SQV/r, High-level resistance | 0
  INI, PI, TPV/r, Susceptible | 1
  INI, PI, TPV/r, Potential low-level resistance | 0
  INI, PI, TPV/r, Low-level resistance | 0
  INI, PI, TPV/r, Intermediate resistance | 0
  INI, PI, TPV/r, High-level resistance | 0

50. Secondary Outcome: Number of Participants With Observed Phenotypic Resistance for Participants Meeting Virologic Withdrawal Criteria by Baseline Third Agent Treatment Class- CAR Group Through Continuation Phase
Description: For all participants who meet virologic withdrawal criteria, plasma samples with HIV-1 RNA level >=200 c/mL were analyzed in an attempt to obtain phenotype data on as many samples as possible. Number of participants with phenotypic resistance to CAR for those meeting virologic withdrawal criteria in subgroups, stratified based on baseline third agent treatment class (INI) were summarized.
Time Frame: Week 52 to Week 411
Population: The analysis was performed on the Late Switch CVW resistance population.
Measure: Count of Participants; unit: Participants
Arm/Group | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 1
Participants
  INI, NNRTI, DLV, Resistant | 1
  INI, NNRTI, DLV, Partially Sensitive | 0
  INI, NNRTI, DLV, Sensitive | 0
  INI, NNRTI, EFV, Resistant | 1
  INI, NNRTI, EFV, Partially Sensitive | 0
  INI, NNRTI, EFV, Sensitive | 0
  INI, NNRTI, ETR, Resistant | 0
  INI, NNRTI, ETR, Partially Sensitive | 0
  INI, NNRTI, ETR, Sensitive | 1
  INI, NNRTI, NVP, Resistant | 1
  INI, NNRTI, NVP, Partially Sensitive | 0
  INI, NNRTI, NVP, Sensitive | 0
  INI, NNRTI, RPV, Resistant | 0
  INI, NNRTI, RPV, Partially Sensitive | 0
  INI, NNRTI, RPV, Sensitive | 1
  INI, NRTI, 3TC, Resistant | 0
  INI, NRTI, 3TC, Partially Sensitive | 0
  INI, NRTI, 3TC, Sensitive | 1
  INI, NRTI, ABC, Resistant | 0
  INI, NRTI, ABC, Partially Sensitive | 0
  INI, NRTI, ABC, Sensitive | 1
  INI, NRTI, FTC, Resistant | 0
  INI, NRTI, FTC, Partially Sensitive | 0
  INI, NRTI, FTC, Sensitive | 1
  INI, NRTI, TDF, Resistant | 0
  INI, NRTI, TDF, Partially Sensitive | 0
  INI, NRTI, TDF, Sensitive | 1
  INI, NRTI, ZDV, Resistant | 0
  INI, NRTI, ZDV, Partially Sensitive | 0
  INI, NRTI, ZDV, Sensitive | 1
  INI, NRTI, d4T, Resistant | 0
  INI, NRTI, d4T, Partially Sensitive | 0
  INI, NRTI, d4T, Sensitive | 1
  INI, NRTI, ddI, Resistant | 0
  INI, NRTI, ddI, Partially Sensitive | 0
  INI, NRTI, ddI, Sensitive | 1
  INI, PI, ATV/r, Resistant | 0
  INI, PI, ATV/r, Partially Sensitive | 0
  INI, PI, ATV/r, Sensitive | 1
  INI, PI, DRV/r, Resistant | 0
  INI, PI, DRV/r, Partially Sensitive | 0
  INI, PI, DRV/r, Sensitive | 1
  INI, PI, FPV/r, Resistant | 0
  INI, PI, FPV/r, Partially Sensitive | 0
  INI, PI, FPV/r, Sensitive | 1
  INI, PI, IDV/r, Resistant | 0
  INI, PI, IDV/r, Partially Sensitive | 0
  INI, PI, IDV/r, Sensitive | 1
  INI, PI, LPV/r, Resistant | 0
  INI, PI, LPV/r, Partially Sensitive | 0
  INI, PI, LPV/r, Sensitive | 1
  INI, PI, NFV, Resistant | 0
  INI, PI, NFV, Partially Sensitive | 0
  INI, PI, NFV, Sensitive | 1
  INI, PI, RTV, Resistant | 0
  INI, PI, RTV, Partially Sensitive | 0
  INI, PI, RTV, Sensitive | 1
  INI, PI, SQV/r, Resistant | 0
  INI, PI, SQV/r, Partially Sensitive | 0
  INI, PI, SQV/r, Sensitive | 1
  INI, PI, TPV/r, Resistant | 0
  INI, PI, TPV/r, Partially Sensitive | 0
  INI, PI, TPV/r, Sensitive | 1

51. Secondary Outcome: Number of Participants With Genotypic Resistance-DTG+RPV Group Through Continuation Phase
Description: Plasma samples were collected for participants meeting the CVW criteria (previous plasma HIV-1 RNA >=50 c/mL and current plasma HIV-1 RNA >= 200 c/mL) to evaluate any potential genotypic evolution of resistance. Genotypic resistance data for the following drugs was presented: DTG, EVG, RAL, DLV, EFV, ETR, NVP, RPV, 3TC, ABC, FTC, TDF, ZDV, d4T, ddI, ATV/r, DRV/r, FPV/r, IDV/r, LPV/r, NFV, RTV, SQV/r, TPV/r.
Time Frame: Up to Week 411
Population: The analysis was performed on the CVW Resistance population which included all participants from the Intent-to-Treat Exposed (ITT-E) population who met CVW through the end of the visit window and had available on-treatment genotypic resistance data at the time the CVW criterion was met.
Measure: Count of Participants; unit: Participants
Arm/Group | DTG + RPV
Number analyzed (Participants) | 6
Participants
  INI, DTG, Susceptible | 6
  INI, DTG, Potential low-level resistance | 0
  INI, DTG, Low-level resistance | 0
  INI, DTG, Intermediate resistance | 0
  INI, DTG, High-level resistance | 0
  INI, EVG, Susceptible | 5
  INI, EVG, Potential low-level resistance | 1
  INI, EVG, Low-level resistance | 0
  INI, EVG, Intermediate resistance | 0
  INI, EVG, High-level resistance | 0
  INI, RAL, Susceptible | 5
  INI, RAL, Potential low-level resistance | 1
  INI, RAL, Low-level resistance | 0
  INI, RAL, Intermediate resistance | 0
  INI, RAL, High-level resistance | 0
  NNRTI, DLV, Susceptible | 6
  NNRTI, DLV, Potential low-level resistance | 0
  NNRTI, DLV, Low-level resistance | 0
  NNRTI, DLV, Intermediate resistance | 0
  NNRTI, DLV, High-level resistance | 0
  NNRTI, EFV, Susceptible | 3
  NNRTI, EFV, Potential low-level resistance | 0
  NNRTI, EFV, Low-level resistance | 1
  NNRTI, EFV, Intermediate resistance | 1
  NNRTI, EFV, High-level resistance | 1
  NNRTI, ETR, Susceptible | 3
  NNRTI, ETR, Potential low-level resistance | 1
  NNRTI, ETR, Low-level resistance | 1
  NNRTI, ETR, Intermediate resistance | 1
  NNRTI, ETR, High-level resistance | 0
  NNRTI, NVP, Susceptible | 3
  NNRTI, NVP, Potential low-level resistance | 0
  NNRTI, NVP, Low-level resistance | 0
  NNRTI, NVP, Intermediate resistance | 1
  NNRTI, NVP, High-level resistance | 2
  NNRTI, RPV, Susceptible | 3
  NNRTI, RPV, Potential low-level resistance | 0
  NNRTI, RPV, Low-level resistance | 1
  NNRTI, RPV, Intermediate resistance | 0
  NNRTI, RPV, High-level resistance | 2
  NRTI, 3TC, Susceptible | 5
  NRTI, 3TC, Potential low-level resistance | 0
  NRTI, 3TC, Low-level resistance | 0
  NRTI, 3TC, Intermediate resistance | 1
  NRTI, 3TC, High-level resistance | 0
  NRTI, ABC, Susceptible | 5
  NRTI, ABC, Potential low-level resistance | 0
  NRTI, ABC, Low-level resistance | 0
  NRTI, ABC, Intermediate resistance | 0
  NRTI, ABC, High-level resistance | 1
  NRTI, FTC, Susceptible | 5
  NRTI, FTC, Potential low-level resistance | 0
  NRTI, FTC, Low-level resistance | 0
  NRTI, FTC, Intermediate resistance | 1
  NRTI, FTC, High-level resistance | 0
  NRTI, TDF, Susceptible | 5
  NRTI, TDF, Potential low-level resistance | 0
  NRTI, TDF, Low-level resistance | 0
  NRTI, TDF, Intermediate resistance | 0
  NRTI, TDF, High-level resistance | 1
  NRTI, ZDV, Susceptible | 4
  NRTI, ZDV, Potential low-level resistance | 1
  NRTI, ZDV, Low-level resistance | 0
  NRTI, ZDV, Intermediate resistance | 0
  NRTI, ZDV, High-level resistance | 1
  NRTI, d4T, Susceptible | 4
  NRTI, d4T, Potential low-level resistance | 1
  NRTI, d4T, Low-level resistance | 0
  NRTI, d4T, Intermediate resistance | 0
  NRTI, d4T, High-level resistance | 1
  NRTI, ddI, Susceptible | 5
  NRTI, ddI, Potential low-level resistance | 0
  NRTI, ddI, Low-level resistance | 0
  NRTI, ddI, Intermediate resistance | 0
  NRTI, ddI, High-level resistance | 1
  PI, ATV/r, Susceptible | 6
  PI, ATV/r, Potential low-level resistance | 0
  PI, ATV/r, Low-level resistance | 0
  PI, ATV/r, Intermediate resistance | 0
  PI, ATV/r, High-level resistance | 0
  PI, DRV/r, Susceptible | 6
  PI, DRV/r, Potential low-level resistance | 0
  PI, DRV/r, Low-level resistance | 0
  PI, DRV/r, Intermediate resistance | 0
  PI, DRV/r, High-level resistance | 0
  PI, FPV/r, Susceptible | 6
  PI, FPV/r, Potential low-level resistance | 0
  PI, FPV/r, Low-level resistance | 0
  PI, FPV/r, Intermediate resistance | 0
  PI, FPV/r, High-level resistance | 0
  PI, IDV/r, Susceptible | 6
  PI, IDV/r, Potential low-level resistance | 0
  PI, IDV/r, Low-level resistance | 0
  PI, IDV/r, Intermediate resistance | 0
  PI, IDV/r, High-level resistance | 0
  PI, LPV/r, Susceptible | 6
  PI, LPV/r, Potential low-level resistance | 0
  PI, LPV/r, Low-level resistance | 0
  PI, LPV/r, Intermediate resistance | 0
  PI, LPV/r, High-level resistance | 0
  PI, NFV, Susceptible | 6
  PI, NFV, Potential low-level resistance | 0
  PI, NFV, Low-level resistance | 00
  PI, NFV, Intermediate resistance | 0
  PI, NFV, High-level resistance | 0
  PI, RTV, Susceptible | 6
  PI, RTV, Potential low-level resistance | 0
  PI, RTV, Low-level resistance | 0
  PI, RTV, Intermediate resistance | 0
  PI, RTV, High-level resistance | 0
  PI, SQV/r, Susceptible | 6
  PI, SQV/r, Potential low-level resistance | 0
  PI, SQV/r, Low-level resistance | 0
  PI, SQV/r, Intermediate resistance | 0
  PI, SQV/r, High-level resistance | 0
  PI, TPV/r, Susceptible | 6
  PI, TPV/r, Potential low-level resistance | 0
  PI, TPV/r, Low-level resistance | 0
  PI, TPV/r, Intermediate resistance | 0
  PI, TPV/r, High-level resistance | 0

52. Secondary Outcome: Number of Participants With Phenotypic Resistance-DTG+RPV Group Through Continuation Phase
Description: Plasma samples were collected for participants meeting the CVW criteria (previous plasma HIV-1 RNA >=50 c/mL and current plasma HIV-1 RNA >= 200 c/mL) to evaluate any potential phenotypic evolution of resistance. Phenotypic resistance data for the following drugs was presented: DTG, EVG, RAL, DLV, EFV, ETR, NVP, RPV, 3TC, ABC, FTC, TDF, ZDV, d4T, ddI, ATV/r, DRV/r, FPV/r, IDV/r, LPV/r, NFV, RTV, SQV/r, TPV/r.
Time Frame: Up to Week 411
Population: The analysis was performed on the CVW Resistance population which included all participants from the ITT-E population who met CVW through the end of the visit window and had available on-treatment phenotypic resistance data at the time the CVW criterion was met.
Measure: Count of Participants; unit: Participants
Arm/Group | DTG + RPV
Number analyzed (Participants) | 6
Participants
  INI, DTG, Resistant: number analyzed (Participants) | 5
  INI, DTG, Resistant | 0
  INI, DTG, Partially Sensitive: number analyzed (Participants) | 5
  INI, DTG, Partially Sensitive | 0
  INI, DTG, Sensitive: number analyzed (Participants) | 5
  INI, DTG, Sensitive | 5
  INI, EVG, Resistant: number analyzed (Participants) | 5
  INI, EVG, Resistant | 0
  INI, EVG, Partially Sensitive: number analyzed (Participants) | 5
  INI, EVG, Partially Sensitive | 0
  INI, EVG, Sensitive: number analyzed (Participants) | 5
  INI, EVG, Sensitive | 5
  INI, RAL, Resistant: number analyzed (Participants) | 5
  INI, RAL, Resistant | 0
  INI, RAL, Partially Sensitive: number analyzed (Participants) | 5
  INI, RAL, Partially Sensitive | 0
  INI, RAL, Sensitive: number analyzed (Participants) | 5
  INI, RAL, Sensitive | 5
  NNRTI, DLV, Resistant | 1
  NNRTI, DLV, Partially Sensitive | 0
  NNRTI, DLV, Sensitive | 5
  NNRTI, EFV, Resistant | 1
  NNRTI, EFV, Partially Sensitive | 0
  NNRTI, EFV, Sensitive | 5
  NNRTI, ETR, Resistant | 0
  NNRTI, ETR, Partially Sensitive | 1
  NNRTI, ETR, Sensitive | 5
  NNRTI, NVP, Resistant | 1
  NNRTI, NVP, Partially Sensitive | 0
  NNRTI, NVP, Sensitive | 5
  NNRTI, RPV, Resistant | 1
  NNRTI, RPV, Partially Sensitive | 0
  NNRTI, RPV, Sensitive | 5
  NRTI, 3TC, Resistant | 0
  NRTI, 3TC, Partially Sensitive | 0
  NRTI, 3TC, Sensitive | 6
  NRTI, ABC, Resistant | 0
  NRTI, ABC, Partially Sensitive | 0
  NRTI, ABC, Sensitive | 6
  NRTI, FTC, Resistant | 0
  NRTI, FTC, Partially Sensitive | 0
  NRTI, FTC, Sensitive | 6
  NRTI, TDF, Resistant | 0
  NRTI, TDF, Partially Sensitive | 0
  NRTI, TDF, Sensitive | 6
  NRTI, ZDV, Resistant | 0
  NRTI, ZDV, Partially Sensitive | 0
  NRTI, ZDV, Sensitive | 6
  NRTI, d4T, Resistant | 0
  NRTI, d4T, Partially Sensitive | 0
  NRTI, d4T, Sensitive | 6
  NRTI, ddI, Resistant | 0
  NRTI, ddI, Partially Sensitive | 0
  NRTI, ddI, Sensitive | 6
  PI, ATV/r, Resistant | 0
  PI, ATV/r, Partially Sensitive | 0
  PI, ATV/r, Sensitive | 6
  PI, DRV/r, Resistant | 0
  PI, DRV/r, Partially Sensitive | 0
  PI, DRV/r, Sensitive | 6
  PI, FPV/r, Resistant | 0
  PI, FPV/r, Partially Sensitive | 0
  PI, FPV/r, Sensitive | 6
  PI, IDV/r, Resistant | 0
  PI, IDV/r, Partially Sensitive | 0
  PI, IDV/r, Sensitive | 6
  PI, LPV/r, Resistant | 0
  PI, LPV/r, Partially Sensitive | 0
  PI, LPV/r, Sensitive | 6
  PI, NFV, Resistant | 0
  PI, NFV, Partially Sensitive | 0
  PI, NFV, Sensitive | 6
  PI, RTV, Resistant | 0
  PI, RTV, Partially Sensitive | 0
  PI, RTV, Sensitive | 6
  PI, SQV/r, Resistant | 0
  PI, SQV/r, Partially Sensitive | 0
  PI, SQV/r, Sensitive | 6
  PI, TPV/r, Resistant | 0
  PI, TPV/r, Partially Sensitive | 0
  PI, TPV/r, Sensitive | 6

53. Secondary Outcome: Number of Participants With Genotypic Resistance-CAR Group Through Continuation Phase
Description: as for outcome 51
Time Frame: Week 52 to Week 411
Population: The analysis was performed on the Late Switch CVW resistance population which included all participants from the Late Switch ITT-E population who met CVW through the end of visit window and had available on-treatment genotypic resistance data at the time the CVW criterion was met.
Measure: Count of Participants; unit: Participants
Arm/Group | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 2
Participants
  INI, DTG, Susceptible: number analyzed (Participants) | 1
  INI, DTG, Susceptible | 1
  INI, DTG, Potential low-level resistance: number analyzed (Participants) | 1
  INI, DTG, Potential low-level resistance | 0
  INI, DTG, Low-level resistance: number analyzed (Participants) | 1
  INI, DTG, Low-level resistance | 0
  INI, DTG, Intermediate resistance: number analyzed (Participants) | 1
  INI, DTG, Intermediate resistance | 0
  INI, DTG, High-level resistance: number analyzed (Participants) | 1
  INI, DTG, High-level resistance | 0
  INI, EVG, Susceptible: number analyzed (Participants) | 1
  INI, EVG, Susceptible | 1
  INI, EVG, Potential low-level resistance: number analyzed (Participants) | 1
  INI, EVG, Potential low-level resistance | 0
  INI, EVG, Low-level resistance: number analyzed (Participants) | 1
  INI, EVG, Low-level resistance | 0
  INI, EVG, Intermediate resistance: number analyzed (Participants) | 1
  INI, EVG, Intermediate resistance | 0
  INI, EVG, High-level resistance: number analyzed (Participants) | 1
  INI, EVG, High-level resistance | 0
  INI, RAL, Susceptible: number analyzed (Participants) | 1
  INI, RAL, Susceptible | 1
  INI, RAL, Potential low-level resistance: number analyzed (Participants) | 1
  INI, RAL, Potential low-level resistance | 0
  INI, RAL, Low-level resistance: number analyzed (Participants) | 1
  INI, RAL, Low-level resistance | 0
  INI, RAL, Intermediate resistance: number analyzed (Participants) | 1
  INI, RAL, Intermediate resistance | 0
  INI, RAL, High-level resistance: number analyzed (Participants) | 1
  INI, RAL, High-level resistance | 0
  NNRTI, DLV, Susceptible: number analyzed (Participants) | 1
  NNRTI, DLV, Susceptible | 1
  NNRTI, DLV, Potential low-level resistance: number analyzed (Participants) | 1
  NNRTI, DLV, Potential low-level resistance | 0
  NNRTI, DLV, Low-level resistance: number analyzed (Participants) | 1
  NNRTI, DLV, Low-level resistance | 0
  NNRTI, DLV, Intermediate resistance: number analyzed (Participants) | 1
  NNRTI, DLV, Intermediate resistance | 0
  NNRTI, DLV, High-level resistance: number analyzed (Participants) | 1
  NNRTI, DLV, High-level resistance | 0
  NNRTI, EFV, Susceptible: number analyzed (Participants) | 1
  NNRTI, EFV, Susceptible | 0
  NNRTI, EFV, Potential low-level resistance: number analyzed (Participants) | 1
  NNRTI, EFV, Potential low-level resistance | 1
  NNRTI, EFV, Low-level resistance: number analyzed (Participants) | 1
  NNRTI, EFV, Low-level resistance | 0
  NNRTI, EFV, Intermediate resistance: number analyzed (Participants) | 1
  NNRTI, EFV, Intermediate resistance | 0
  NNRTI, EFV, High-level resistance: number analyzed (Participants) | 1
  NNRTI, EFV, High-level resistance | 0
  NNRTI, ETR, Susceptible: number analyzed (Participants) | 1
  NNRTI, ETR, Susceptible | 0
  NNRTI, ETR, Potential low-level resistance: number analyzed (Participants) | 1
  NNRTI, ETR, Potential low-level resistance | 1
  NNRTI, ETR, Low-level resistance: number analyzed (Participants) | 1
  NNRTI, ETR, Low-level resistance | 0
  NNRTI, ETR, Intermediate resistance: number analyzed (Participants) | 1
  NNRTI, ETR, Intermediate resistance | 0
  NNRTI, ETR, High-level resistance: number analyzed (Participants) | 1
  NNRTI, ETR, High-level resistance | 0
  NNRTI, NVP, Susceptible: number analyzed (Participants) | 1
  NNRTI, NVP, Susceptible | 0
  NNRTI, NVP, Potential low-level resistance: number analyzed (Participants) | 1
  NNRTI, NVP, Potential low-level resistance | 1
  NNRTI, NVP, Low-level resistance: number analyzed (Participants) | 1
  NNRTI, NVP, Low-level resistance | 0
  NNRTI, NVP, Intermediate resistance: number analyzed (Participants) | 1
  NNRTI, NVP, Intermediate resistance | 0
  NNRTI, NVP, High-level resistance: number analyzed (Participants) | 1
  NNRTI, NVP, High-level resistance | 0
  NNRTI, RPV, Susceptible: number analyzed (Participants) | 1
  NNRTI, RPV, Susceptible | 0
  NNRTI, RPV, Potential low-level resistance: number analyzed (Participants) | 1
  NNRTI, RPV, Potential low-level resistance | 1
  NNRTI, RPV, Low-level resistance: number analyzed (Participants) | 1
  NNRTI, RPV, Low-level resistance | 0
  NNRTI, RPV, Intermediate resistance: number analyzed (Participants) | 1
  NNRTI, RPV, Intermediate resistance | 0
  NNRTI, RPV, High-level resistance: number analyzed (Participants) | 1
  NNRTI, RPV, High-level resistance | 0
  NRTI, 3TC, Susceptible: number analyzed (Participants) | 1
  NRTI, 3TC, Susceptible | 1
  NRTI, 3TC, Potential low-level resistance: number analyzed (Participants) | 1
  NRTI, 3TC, Potential low-level resistance | 0
  NRTI, 3TC, Low-level resistance: number analyzed (Participants) | 1
  NRTI, 3TC, Low-level resistance | 0
  NRTI, 3TC, Intermediate resistance: number analyzed (Participants) | 1
  NRTI, 3TC, Intermediate resistance | 0
  NRTI, 3TC, High-level resistance: number analyzed (Participants) | 1
  NRTI, 3TC, High-level resistance | 0
  NRTI, ABC, Susceptible: number analyzed (Participants) | 1
  NRTI, ABC, Susceptible | 1
  NRTI, ABC, Potential low-level resistance: number analyzed (Participants) | 1
  NRTI, ABC, Potential low-level resistance | 0
  NRTI, ABC, Low-level resistance: number analyzed (Participants) | 1
  NRTI, ABC, Low-level resistance | 0
  NRTI, ABC, Intermediate resistance: number analyzed (Participants) | 1
  NRTI, ABC, Intermediate resistance | 0
  NRTI, ABC, High-level resistance: number analyzed (Participants) | 1
  NRTI, ABC, High-level resistance | 0
  NRTI, FTC, Susceptible: number analyzed (Participants) | 1
  NRTI, FTC, Susceptible | 1
  NRTI, FTC, Potential low-level resistance: number analyzed (Participants) | 1
  NRTI, FTC, Potential low-level resistance | 0
  NRTI, FTC, Low-level resistance: number analyzed (Participants) | 1
  NRTI, FTC, Low-level resistance | 0
  NRTI, FTC, Intermediate resistance: number analyzed (Participants) | 1
  NRTI, FTC, Intermediate resistance | 0
  NRTI, FTC, High-level resistance: number analyzed (Participants) | 1
  NRTI, FTC, High-level resistance | 0
  NRTI, TDF, Susceptible: number analyzed (Participants) | 1
  NRTI, TDF, Susceptible | 1
  NRTI, TDF, Potential low-level resistance: number analyzed (Participants) | 1
  NRTI, TDF, Potential low-level resistance | 0
  NRTI, TDF, Low-level resistance: number analyzed (Participants) | 1
  NRTI, TDF, Low-level resistance | 0
  NRTI, TDF, Intermediate resistance: number analyzed (Participants) | 1
  NRTI, TDF, Intermediate resistance | 0
  NRTI, TDF, High-level resistance: number analyzed (Participants) | 1
  NRTI, TDF, High-level resistance | 0
  NRTI, ZDV, Susceptible: number analyzed (Participants) | 1
  NRTI, ZDV, Susceptible | 1
  NRTI, ZDV, Potential low-level resistance: number analyzed (Participants) | 1
  NRTI, ZDV, Potential low-level resistance | 0
  NRTI, ZDV, Low-level resistance: number analyzed (Participants) | 1
  NRTI, ZDV, Low-level resistance | 0
  NRTI, ZDV, Intermediate resistance: number analyzed (Participants) | 1
  NRTI, ZDV, Intermediate resistance | 0
  NRTI, ZDV, High-level resistance: number analyzed (Participants) | 1
  NRTI, ZDV, High-level resistance | 0
  NRTI, d4T, Susceptible: number analyzed (Participants) | 1
  NRTI, d4T, Susceptible | 1
  NRTI, d4T, Potential low-level resistance: number analyzed (Participants) | 1
  NRTI, d4T, Potential low-level resistance | 0
  NRTI, d4T, Low-level resistance: number analyzed (Participants) | 1
  NRTI, d4T, Low-level resistance | 0
  NRTI, d4T, Intermediate resistance: number analyzed (Participants) | 1
  NRTI, d4T, Intermediate resistance | 0
  NRTI, d4T, High-level resistance: number analyzed (Participants) | 1
  NRTI, d4T, High-level resistance | 0
  NRTI, ddI, Susceptible: number analyzed (Participants) | 1
  NRTI, ddI, Susceptible | 1
  NRTI, ddI, Potential low-level resistance: number analyzed (Participants) | 1
  NRTI, ddI, Potential low-level resistance | 0
  NRTI, ddI, Low-level resistance: number analyzed (Participants) | 1
  NRTI, ddI, Low-level resistance | 0
  NRTI, ddI, Intermediate resistance: number analyzed (Participants) | 1
  NRTI, ddI, Intermediate resistance | 0
  NRTI, ddI, High-level resistance: number analyzed (Participants) | 1
  NRTI, ddI, High-level resistance | 0
  PI, ATV/r, Susceptible: number analyzed (Participants) | 1
  PI, ATV/r, Susceptible | 1
  PI, ATV/r, Potential low-level resistance: number analyzed (Participants) | 1
  PI, ATV/r, Potential low-level resistance | 0
  PI, ATV/r, Low-level resistance: number analyzed (Participants) | 1
  PI, ATV/r, Low-level resistance | 0
  PI, ATV/r, Intermediate resistance: number analyzed (Participants) | 1
  PI, ATV/r, Intermediate resistance | 0
  PI, ATV/r, High-level resistance: number analyzed (Participants) | 1
  PI, ATV/r, High-level resistance | 0
  PI, DRV/r, Susceptible: number analyzed (Participants) | 1
  PI, DRV/r, Susceptible | 1
  PI, DRV/r, Potential low-level resistance: number analyzed (Participants) | 1
  PI, DRV/r, Potential low-level resistance | 0
  PI, DRV/r, Low-level resistance: number analyzed (Participants) | 1
  PI, DRV/r, Low-level resistance | 0
  PI, DRV/r, Intermediate resistance: number analyzed (Participants) | 1
  PI, DRV/r, Intermediate resistance | 0
  PI, DRV/r, High-level resistance: number analyzed (Participants) | 1
  PI, DRV/r, High-level resistance | 0
  PI, FPV/r, Susceptible: number analyzed (Participants) | 1
  PI, FPV/r, Susceptible | 1
  PI, FPV/r, Potential low-level resistance: number analyzed (Participants) | 1
  PI, FPV/r, Potential low-level resistance | 0
  PI, FPV/r, Low-level resistance: number analyzed (Participants) | 1
  PI, FPV/r, Low-level resistance | 0
  PI, FPV/r, Intermediate resistance: number analyzed (Participants) | 1
  PI, FPV/r, Intermediate resistance | 0
  PI, FPV/r, High-level resistance: number analyzed (Participants) | 1
  PI, FPV/r, High-level resistance | 0
  PI, IDV/r, Susceptible: number analyzed (Participants) | 1
  PI, IDV/r, Susceptible | 1
  PI, IDV/r, Potential low-level resistance: number analyzed (Participants) | 1
  PI, IDV/r, Potential low-level resistance | 0
  PI, IDV/r, Low-level resistance: number analyzed (Participants) | 1
  PI, IDV/r, Low-level resistance | 0
  PI, IDV/r, Intermediate resistance: number analyzed (Participants) | 1
  PI, IDV/r, Intermediate resistance | 0
  PI, IDV/r, High-level resistance: number analyzed (Participants) | 1
  PI, IDV/r, High-level resistance | 0
  PI, LPV/r, Susceptible: number analyzed (Participants) | 1
  PI, LPV/r, Susceptible | 1
  PI, LPV/r, Potential low-level resistance: number analyzed (Participants) | 1
  PI, LPV/r, Potential low-level resistance | 0
  PI, LPV/r, Low-level resistance: number analyzed (Participants) | 1
  PI, LPV/r, Low-level resistance | 0
  PI, LPV/r, Intermediate resistance: number analyzed (Participants) | 1
  PI, LPV/r, Intermediate resistance | 0
  PI, LPV/r, High-level resistance: number analyzed (Participants) | 1
  PI, LPV/r, High-level resistance | 0
  PI, NFV, Susceptible: number analyzed (Participants) | 1
  PI, NFV, Susceptible | 1
  PI, NFV, Potential low-level resistance: number analyzed (Participants) | 1
  PI, NFV, Potential low-level resistance | 0
  PI, NFV, Low-level resistance: number analyzed (Participants) | 1
  PI, NFV, Low-level resistance | 0
  PI, NFV, Intermediate resistance: number analyzed (Participants) | 1
  PI, NFV, Intermediate resistance | 0
  PI, NFV, High-level resistance: number analyzed (Participants) | 1
  PI, NFV, High-level resistance | 0
  PI, RTV, Susceptible: number analyzed (Participants) | 1
  PI, RTV, Susceptible | 1
  PI, RTV, Potential low-level resistance: number analyzed (Participants) | 1
  PI, RTV, Potential low-level resistance | 0
  PI, RTV, Low-level resistance: number analyzed (Participants) | 1
  PI, RTV, Low-level resistance | 0
  PI, RTV, Intermediate resistance: number analyzed (Participants) | 1
  PI, RTV, Intermediate resistance | 0
  PI, RTV, High-level resistance: number analyzed (Participants) | 1
  PI, RTV, High-level resistance | 0
  PI, SQV/r, Susceptible: number analyzed (Participants) | 1
  PI, SQV/r, Susceptible | 1
  PI, SQV/r, Potential low-level resistance: number analyzed (Participants) | 1
  PI, SQV/r, Potential low-level resistance | 0
  PI, SQV/r, Low-level resistance: number analyzed (Participants) | 1
  PI, SQV/r, Low-level resistance | 0
  PI, SQV/r, Intermediate resistance: number analyzed (Participants) | 1
  PI, SQV/r, Intermediate resistance | 0
  PI, SQV/r, High-level resistance: number analyzed (Participants) | 1
  PI, SQV/r, High-level resistance | 0
  PI, TPV/r, Susceptible: number analyzed (Participants) | 1
  PI, TPV/r, Susceptible | 1
  PI, TPV/r, Potential low-level resistance: number analyzed (Participants) | 1
  PI, TPV/r, Potential low-level resistance | 0
  PI, TPV/r, Low-level resistance: number analyzed (Participants) | 1
  PI, TPV/r, Low-level resistance | 0
  PI, TPV/r, Intermediate resistance: number analyzed (Participants) | 1
  PI, TPV/r, Intermediate resistance | 0
  PI, TPV/r, High-level resistance: number analyzed (Participants) | 1
  PI, TPV/r, High-level resistance | 0

54. Secondary Outcome: Number of Participants With Phenotypic Resistance- CAR Group Through Continuation Phase
Description: as for outcome 52
Time Frame: Week 52 to Week 411
Population: The analysis was performed on the Late Switch CVW Resistance population which included all participants from the Late Switch ITT-E population who met CVW through the end of visit window and had available on-treatment phenotypic resistance data at the time the CVW criterion was met.
Measure: Count of Participants; unit: Participants
Arm/Group | Current Antiretroviral Regimen (CAR)
Number analyzed (Participants) | 2
Participants
  NNRTI, DLV, Resistant: number analyzed (Participants) | 1
  NNRTI, DLV, Resistant | 1
  NNRTI, DLV, Partially Sensitive: number analyzed (Participants) | 1
  NNRTI, DLV, Partially Sensitive | 0
  NNRTI, DLV, Sensitive: number analyzed (Participants) | 1
  NNRTI, DLV, Sensitive | 0
  NNRTI, EFV, Resistant: number analyzed (Participants) | 1
  NNRTI, EFV, Resistant | 1
  NNRTI, EFV, Partially Sensitive: number analyzed (Participants) | 1
  NNRTI, EFV, Partially Sensitive | 0
  NNRTI, EFV, Sensitive: number analyzed (Participants) | 1
  NNRTI, EFV, Sensitive | 0
  NNRTI, ETR, Resistant: number analyzed (Participants) | 1
  NNRTI, ETR, Resistant | 0
  NNRTI, ETR, Partially Sensitive: number analyzed (Participants) | 1
  NNRTI, ETR, Partially Sensitive | 0
  NNRTI, ETR, Sensitive: number analyzed (Participants) | 1
  NNRTI, ETR, Sensitive | 1
  NNRTI, NVP, Resistant: number analyzed (Participants) | 1
  NNRTI, NVP, Resistant | 1
  NNRTI, NVP, Partially Sensitive: number analyzed (Participants) | 1
  NNRTI, NVP, Partially Sensitive | 0
  NNRTI, NVP, Sensitive: number analyzed (Participants) | 1
  NNRTI, NVP, Sensitive | 0
  NNRTI, RPV, Resistant: number analyzed (Participants) | 1
  NNRTI, RPV, Resistant | 0
  NNRTI, RPV, Partially Sensitive: number analyzed (Participants) | 1
  NNRTI, RPV, Partially Sensitive | 0
  NNRTI, RPV, Sensitive: number analyzed (Participants) | 1
  NNRTI, RPV, Sensitive | 1
  NRTI, 3TC, Resistant: number analyzed (Participants) | 1
  NRTI, 3TC, Resistant | 0
  NRTI, 3TC, Partially Sensitive: number analyzed (Participants) | 1
  NRTI, 3TC, Partially Sensitive | 0
  NRTI, 3TC, Sensitive: number analyzed (Participants) | 1
  NRTI, 3TC, Sensitive | 1
  NRTI, ABC, Resistant: number analyzed (Participants) | 1
  NRTI, ABC, Resistant | 0
  NRTI, ABC, Partially Sensitive: number analyzed (Participants) | 1
  NRTI, ABC, Partially Sensitive | 0
  NRTI, ABC, Sensitive: number analyzed (Participants) | 1
  NRTI, ABC, Sensitive | 1
  NRTI, FTC, Resistant: number analyzed (Participants) | 1
  NRTI, FTC, Resistant | 0
  NRTI, FTC, Partially Sensitive: number analyzed (Participants) | 1
  NRTI, FTC, Partially Sensitive | 0
  NRTI, FTC, Sensitive: number analyzed (Participants) | 1
  NRTI, FTC, Sensitive | 1
  NRTI, TDF, Resistant: number analyzed (Participants) | 1
  NRTI, TDF, Resistant | 0
  NRTI, TDF, Partially Sensitive: number analyzed (Participants) | 1
  NRTI, TDF, Partially Sensitive | 0
  NRTI, TDF, Sensitive: number analyzed (Participants) | 1
  NRTI, TDF, Sensitive | 1
  NRTI, ZDV, Resistant: number analyzed (Participants) | 1
  NRTI, ZDV, Resistant | 0
  NRTI, ZDV, Partially Sensitive: number analyzed (Participants) | 1
  NRTI, ZDV, Partially Sensitive | 0
  NRTI, ZDV, Sensitive: number analyzed (Participants) | 1
  NRTI, ZDV, Sensitive | 1
  NRTI, d4T, Resistant: number analyzed (Participants) | 1
  NRTI, d4T, Resistant | 0
  NRTI, d4T, Partially Sensitive: number analyzed (Participants) | 1
  NRTI, d4T, Partially Sensitive | 0
  NRTI, d4T, Sensitive: number analyzed (Participants) | 1
  NRTI, d4T, Sensitive | 1
  NRTI, ddI, Resistant: number analyzed (Participants) | 1
  NRTI, ddI, Resistant | 0
  NRTI, ddI, Partially Sensitive: number analyzed (Participants) | 1
  NRTI, ddI, Partially Sensitive | 0
  NRTI, ddI, Sensitive: number analyzed (Participants) | 1
  NRTI, ddI, Sensitive | 1
  PI, ATV/r, Resistant: number analyzed (Participants) | 1
  PI, ATV/r, Resistant | 0
  PI, ATV/r, Partially Sensitive: number analyzed (Participants) | 1
  PI, ATV/r, Partially Sensitive | 0
  PI, ATV/r, Sensitive: number analyzed (Participants) | 1
  PI, ATV/r, Sensitive | 1
  PI, DRV/r, Resistant: number analyzed (Participants) | 1
  PI, DRV/r, Resistant | 0
  PI, DRV/r, Partially Sensitive: number analyzed (Participants) | 1
  PI, DRV/r, Partially Sensitive | 0
  PI, DRV/r, Sensitive: number analyzed (Participants) | 1
  PI, DRV/r, Sensitive | 1
  PI, FPV/r, Resistant: number analyzed (Participants) | 1
  PI, FPV/r, Resistant | 0
  PI, FPV/r, Partially Sensitive: number analyzed (Participants) | 1
  PI, FPV/r, Partially Sensitive | 0
  PI, FPV/r, Sensitive: number analyzed (Participants) | 1
  PI, FPV/r, Sensitive | 1
  PI, IDV/r, Resistant: number analyzed (Participants) | 1
  PI, IDV/r, Resistant | 0
  PI, IDV/r, Partially Sensitive: number analyzed (Participants) | 1
  PI, IDV/r, Partially Sensitive | 0
  PI, IDV/r, Sensitive: number analyzed (Participants) | 1
  PI, IDV/r, Sensitive | 1
  PI, LPV/r, Resistant: number analyzed (Participants) | 1
  PI, LPV/r, Resistant | 0
  PI, LPV/r, Partially Sensitive: number analyzed (Participants) | 1
  PI, LPV/r, Partially Sensitive | 0
  PI, LPV/r, Sensitive: number analyzed (Participants) | 1
  PI, LPV/r, Sensitive | 1
  PI, NFV, Resistant: number analyzed (Participants) | 1
  PI, NFV, Resistant | 0
  PI, NFV, Partially Sensitive: number analyzed (Participants) | 1
  PI, NFV, Partially Sensitive | 0
  PI, NFV, Sensitive: number analyzed (Participants) | 1
  PI, NFV, Sensitive | 1
  PI, RTV, Resistant: number analyzed (Participants) | 1
  PI, RTV, Resistant | 0
  PI, RTV, Partially Sensitive: number analyzed (Participants) | 1
  PI, RTV, Partially Sensitive | 0
  PI, RTV, Sensitive: number analyzed (Participants) | 1
  PI, RTV, Sensitive | 1
  PI, SQV/r, Resistant: number analyzed (Participants) | 1
  PI, SQV/r, Resistant | 0
  PI, SQV/r, Partially Sensitive: number analyzed (Participants) | 1
  PI, SQV/r, Partially Sensitive | 0
  PI, SQV/r, Sensitive: number analyzed (Participants) | 1
  PI, SQV/r, Sensitive | 1
  PI, TPV/r, Resistant: number analyzed (Participants) | 1
  PI, TPV/r, Resistant | 0
  PI, TPV/r, Partially Sensitive: number analyzed (Participants) | 1
  PI, TPV/r, Partially Sensitive | 0
  PI, TPV/r, Sensitive: number analyzed (Participants) | 1
  PI, TPV/r, Sensitive | 1

ADVERSE EVENTS:
Time Frame: SAEs and all non-serious AEs were collected from study start until Week 148, thereafter SAEs and only AEs leading to withdrawal were collected until Week 411.
Description: On treatment SAEs and non-serious AEs were reported for the Safety Population for DTG+RPV (Early Switch), CAR (Early Switch) and DTG+RPV (Early+Late Switch). Late Switch Safety Population was used for CAR (Late Switch). Continuation Phase Safety Population was used for DTG+RPV (Continuation Phase) and CAR (Continuation Phase).
Groups:
- DTG + RPV (Early Switch): Participants received DTG 50 mg + RPV 25 mg together once daily at approximately the same time, with a meal, in an open-label fashion up to Week 52 during early switch phase.
- CAR (Early Switch): Participants continued to receive their current antiretroviral regimen (two NRTIs + a third agent). A third agent included either an: INSTI, NNRTI or a PI. CAR was administered according to the approved labeling in an open-label fashion up to Week 52 during early switch phase.
- DTG + RPV (Early + Late Switch): Participants received DTG 50 mg + RPV 25 mg together once daily at approximately the same time, with a meal, in an open-label fashion up to Week 52 during early switch phase. Participants continued to receive DTG 50 mg + RPV 25 mg up to Week 148 during the Late Switch Phase.
- CAR (Late Switch): Participants continued to receive their current antiretroviral regimen (two NRTIs + a third agent). A third agent included either an: INSTI, NNRTI or a PI. CAR was administered according to the approved labeling in an open-label fashion up to Week 52 during early switch phase.
  At Week 52, participants who received CAR during the early switch phase, with HIV-1 RNA <50 c/mL, switched to DTG 50 mg + RPV 25 mg once daily and were followed until Week 148.
- DTG + RPV (Continuation Phase): Participants received DTG 50 mg + RPV 25 mg together, once daily, at approximately the same time, with a meal, in an open-label fashion up to Week 52, during the Early Switch Phase. Participants continued to receive DTG 50 mg + RPV 25 mg up to Week 148 during the Late Switch Phase. Participants who successfully completed 148 weeks of treatment were given the opportunity to continue to receive DTG + RPV once daily in the Continuation Phase (after Week 148).
- CAR (Continuation Phase): Participants continued to receive their CAR (NRTIs + a third agent). A third agent included either an: INSTI, a NNRTI or a PI. CAR was administered according to the approved labeling in an open-label fashion up to Week 52 during the Early Switch Phase. At Week 52, participants with HIV-1 RNA <50 c/mL, switched to DTG 50 mg + RPV 25 mg once daily and were followed-up through the Late Switch Phase, at Week 148 and through the Continuation Phase, after Week 148.
Arm/Group | DTG + RPV (Early Switch) | CAR (Early Switch) | DTG + RPV (Early + Late Switch) | CAR (Late Switch) | DTG + RPV (Continuation Phase) | CAR (Continuation Phase)
All-Cause Mortality (participants affected / at risk) | 0/252 | 1/256 | 1/252 | 0/238 | 0/186 | 0/183
Serious Adverse Events (participants affected / at risk) | 10/252 | 13/256 | 34/252 | 22/238 | 6/186 | 9/183
Other Adverse Events (participants affected / at risk) | 107/252 | 102/256 | 167/252 | 134/238 | 0/186 | 0/183
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DTG + RPV (Early Switch) (N=252) | CAR (Early Switch) (N=256) | DTG + RPV (Early + Late Switch) (N=252) | CAR (Late Switch) (N=238) | DTG + RPV (Continuation Phase) (N=186) | CAR (Continuation Phase) (N=183)
Hepatitis A (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hodgkin's disease mixed cellularity stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Plasmablastic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute hepatitis B (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Arthritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatitis C (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral artery stenosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proctitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Shigella infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Testicular germ cell tumour mixed (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thyroglossal cyst infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thyroid mass (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toxic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wolff-Parkinson-White syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound infection staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Penile contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis obstructive (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DTG + RPV (Early Switch) (N=252) | CAR (Early Switch) (N=256) | DTG + RPV (Early + Late Switch) (N=252) | CAR (Late Switch) (N=238) | DTG + RPV (Continuation Phase) (N=186) | CAR (Continuation Phase) (N=183)
Nasopharyngitis (Infections and infestations) | 27 (33) | 31 (35) | 52 (84) | 39 (55) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 24 (25) | 17 (19) | 37 (43) | 23 (29) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 22 (24) | 17 (18) | 35 (38) | 19 (20) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (9) | 19 (20) | 25 (28) | 18 (19) | 0 (0) | 0 (0)
Syphilis (Infections and infestations) | 8 (10) | 7 (7) | 27 (39) | 20 (24) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 7 (9) | 10 (11) | 26 (32) | 17 (25) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 9 (10) | 6 (6) | 18 (20) | 18 (20) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 (9) | 5 (6) | 18 (19) | 12 (16) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (10) | 4 (5) | 14 (17) | 17 (19) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 4 (4) | 12 (13) | 12 (12) | 13 (16) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 7 (7) | 4 (5) | 16 (19) | 11 (14) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 9 (9) | 10 (10) | 13 (13) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 10 (10) | 2 (2) | 17 (18) | 5 (6) | 0 (0) | 0 (0)
Fatigue (General disorders) | 9 (9) | 3 (3) | 13 (14) | 6 (6) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 9 (9) | 2 (2) | 13 (13) | 3 (3) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.